Replication of Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial (ONTARGET trial)

July 13, 2020

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 <u>Title</u>

Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial (ONTARGET trial)

#### 1.2 <u>Intended aim(s)</u>

The primary objectives of the study were to determine the effectiveness of 80 mg of telmisartan daily, as compared with 10 mg of ramipril daily. If noninferiority was demonstrated, we would test the superiority of telmisartan over ramipril.

#### 1.3 Primary endpoint for replication and RCT finding

Death from cardiovascular causes, myocardial infarction, stroke, or hospitalization for heart failure.

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

The original planned sample size of 7800 patients who were followed for a mean of 4.5 years provided a power of 93% for the superiority hypothesis, if the hazard ratio was 0.87. For noninferiority, the expected power was 89%, for a hazard ratio of 1.00. The non-inferiority margin was 1.13.

#### 1.5 Primary trial estimate targeted for replication

HR = 1.01 (95% CI 0.94–1.09) comparing telmisartan to ramipril (Yusuf et al., 2008, NEJM)

#### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

#### 3. Data Source(s)

United/Optum, MarketScan

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

#### Design Diagram - ONTARGET TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing telmisartan to ramipril. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of telmisartan or the comparator drug (cohort entry date). Follow-up for the outcome, begins the day after drug initiation. Patients are also required to have no prior ACE or ARB use during the 3 months before the cohort entry date, but they are allowed to take other antihypertensive medications during the study, as in the trial.

#### 5.2 Important steps for cohort formation

#### 5.2.1 Eligible cohort entry dates

Market availability of telmisartan in the U.S. started on November 10, 1998, however, the Marketscan and Optum data are available at BWH only from Jan 1, 2003 and Jan 1, 2004, respectively.

- For Marketscan: Jul 1, 2003 -Dec 2018 (end of data availability).
- For Optum: Jan 1, 2004- Dec 2019 (end of data availability).

#### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

| | Optum | | Truven | |
|---|---|---|---|---|
| Less Excluded Patients | Remaining<br>Patients | | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 75,894,642 | | 200,203,908 |
| Did not meet cohort entry criteria | -75,250,227 | 644,415 | -198,892,008 | 1,311,900 |
| Excluded due to insufficient enrollment | -74,705 | 569,710 | -167,142 | 1,144,758 |
| Excluded due to prior use of referent | -295257 | 274,453 | -639288 | 505,470 |

| Excluded due to prior use of exposure | -155,795 | 118,658 | -264,031 | 241,439 |
|---|---|---|---|---|
| Excluded because patient qualified in >1 exposure category | | 118,641 | -25 | 241,414 |
| Excluded based on Age | 0 | 118,641 | 0 | 241,414 |
| Excluded based on Gender | -14 | 118,627 | 0 | 241,414 |
| Excluded based on Inclusion Age >= 55 | -29,428 | 89,199 | -59,190 | 182,224 |
| Excluded based on All inclusion criteria (Coronary artery disease/Peripheral artery disease/Cerebrovascular disease) EXCEPT Age >=55 | -28349 | 60,850 | -51572 | 130,652 |
| Excluded based on Exclusion 2a- Heart failure (CHF) (inpatient/ER) | -2,267 | 58,583 | -4,218 | 126,434 |
| Excluded based on Exclusion 2b- Hemodynamically significant primary valvular or outflow tract obstruction | -950 | 57,633 | -736 | 125,698 |
| Excluded based on Exclusion 2c- Constrictive pericarditis | -1 | 57,632 | -3 | 125,695 |
| Excluded based on Exclusion 2d- Complex congenital heart disease | | 57,386 | -382 | 125,313 |
| Excluded based on Exclusion 2e- Syncopal episodes of unknown etiology <3 months before informed consent | | 56,915 | -1,178 | 124,135 |
| Excluded based on Exclusion 2g- Uncontrolled hypertension on treatment (eg, BP >160/100 mm Hg) | | 56,218 | -1080 | 123,055 |
| Excluded based on Exclusion 2f- Heart transplant recipient | -2 | 56,216 | -2 | 123,053 |
| Excluded based on Exclusion 2g- Stroke due to subarachnoid hemorrhage | -40 | 56,176 | -85 | 122,968 |
| Excluded based on Exclusoin 3a- Significant renal artery disease | -160 | 56,016 | -224 | 122,744 |
| Excluded based on Exclusion 3b- Hepatic dysfunction | -297 | 55,719 | -614 | 122,130 |
| Excluded based on Exclusio 3d- Primary hyperaldosteronism | -1 | 55,718 | -1 | 122,129 |
| Excluded based on Exclusion 3e- Hereditary fructose intolerance | 0 | 55,718 | 0 | 122,129 |
| Excluded based on Exclusion 3f- Other major noncardiac illness expected to reduce life expectancy or interfere with study participation- CCI (180 days) | -222 | 55,496 | -123 | 122,006 |
| Excluded based on ACE or ARB (prior 3 months) | -5,543 | 49,953 | -7,266 | 114,740 |
| Final cohort | | 49,953 | | 114,740 |

## 6. Variables

## 6.1 Exposure-related variables:

## Study drug:

Effectiveness research with Real World Data to support FDA's regulatory decision making

The study exposure of interest is initiation of telmisartan. Initiation will be defined by no use of telmisartan or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents-

- · Initiators of telmisartan will be compared to initiators of
  - o Ramipril (primary)

#### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B). These covariates are based on those used by Patorno et al. (2019).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome of interest (definitions provided in Appendix A):

- <u>Primary outcome</u>: Composite endpoint including death from cardiovascular causes, myocardial infarction, stroke, and hospitalization for heart failure
- Secondary outcomes: Individual components:
  - o Heart failure requiring hospitalization
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)

- Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
- All-cause inpatient mortality/CV mortality:
  - Information on CV mortality through data linkage with the National Death Index (NDI) will only be available for CMS.
  - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of telmisartan and comparator and will continue until the earliest date of the following events:

- · The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (telmisartan
  and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main
  analyses).
- The date of switching from an exposure to a comparator and vice versa, defined as a prescription fill from the other treatment group.

For the intention-to-treat (ITT) analyses, the censoring based on the switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/774/results/55701/result/0
MarketScan- https://bwh-dope.aetion.com/projects/details/775/results/55702/result/0

Date conducted: 06/27/2020

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Complete study flowchart from Section 5.3
- · Report patient characteristics by treatment group
- Report summary parameters of study population
- · Report median follow-up time by treatment group
- · Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/#/projects/details/774/results/31496/result/1
MarketScan- https://bwh-dope.aetion.com/#/projects/details/775/results/31494/result/1

Date conducted: 02/11/2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the

analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 7/16/19 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 7/30/19 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment after PS matching

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/774/results/55703/result/0">https://bwh-dope.aetion.com/projects/details/774/results/55703/result/0</a>
<a href="MarketScan-https://bwh-dope.aetion.com/projects/details/775/results/55704/result/0">https://bwh-dope.aetion.com/projects/details/775/results/55704/result/0</a>

Date conducted: 06/27/2020

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 343 (0.54%) | 211 (0.66%) | 132 (0.41%) |
| Start of an additional exposure | 189 (0.30%) | 95 (0.30%) | 94 (0.29%) |
| End of index exposure | 47,275 (74.16%) | 22,786 (71.49%) | 24,489<br>(76.84%) |
| Specified date reached | 3,666 (5.75%) | 1,949 (6.12%) | 1,717 (5.39%) |
| End of patient enrollment | 10,559 (16.56%) | 5,864 (18.40%) | 4,695 (14.73%) |
| Nursing home + Pharmacy<br>disenrollment | 1,712 (2.69%) | 967 (3.03%) | 745 (2.34%) |

## • Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|--------------|--------------|
| Patient Group Optum Marketscan | | |
| Overall Patient Population | 118 [58-299] | 151 [94-365] |
| Referent | 144 [79-342] | 177 [99-403] |
| Exposure | 118 [58-260] | 128 [91-319] |

## • Report overall risk of the primary outcome.

| | Optum | Marketscan | Pooled |
|---|---|---|---|
| Risk per 1,000 patients (Composite endpoint | | | |
| including death from cardiovascular causes, | | | |
| myocardial infarction, stroke, and hospitalization | | | |
| for heart failure) | 52.3 | 55.2 | 54.3 |

#### 10. Final Power Assessment

#### Date conducted:

Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9.
 All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).

Pooled

| Toolca | | | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | | Number of patients matched | |
| Reference | 31,872 | Reference | 31,872 |
| Exposed | 31,872 | Exposed | 31,872 |
| Risk per 1,000 patients | 54.3 | Risk per 1,000 patients | 54.30 |
| Desired HR from RCT | 0.87 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.13 |
| Number of events expected | 3461.2992 | Number of events expected | 3461.2992 |
| Power | 0.983685756 | Power | 0.949000546 |

Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 10,798 | Reference | 10,798 |
| Exposed | 10,798 | Exposed | 10,798 |
| Risk per 1,000 patients | 52.3 | Risk per 1,000 patients | 52.3 |
| Desired HR from RCT | 0.87 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.13 |
| Number of events expected | 1129.4708 | Number of events expected | 1129.4708 |
| Power | 0.648098168 | Power | 0.537348783 |

## MarketScan

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 21,074 | Reference | 21,074 |
| Exposed | 21,074 | Exposed | 21,074 |
| Risk per 1,000 patients | 55.2 | Risk per 1,000 patients | 55.2 |
| Desired HR from RCT | 0.87 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.13 |
| Number of events expected | 2326.5696 | Number of events expected | 2326.5696 |
| Power | 0.919041969 | Power | 0.838323471 |

Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of
advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of
patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates
of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 7/6/20 |
|-------------------------|------------------|----------------|--------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/5/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

· Register the study on clinicalTrials.gov and upload this document.

#### 13. Comparative Analyses

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### Aetion report name:

#### Date conducted:

#### 13.1 For primary analysis:

• In the PS-matched cohort of telmisartan and ramipril from Section 9, calculate the HR for each outcome for telmisartan versus referent patients using a Cox proportional hazards model.

### 13.2 For sensitivity analyses:

#### 14. Requested Results

#### 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | | After adjust | ment | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

### 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

#### 14.3 Table 3: Censoring events

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

#### 14.4 Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 14.5 <u>Table 5: Results from secondary analyses;</u>

#### 15. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019; in press. (https://www.ahajournals.org/doi/pdf/10.1161/CIRCULATIONAHA.118.039177)

| | T | | | |
|---|---|---|---|---|
| # | ONTARGET trial definitions | Implementation in routine care | References/Rationale | Colorcoding |
| | Trial details- 3- Failed S- No Ni margin specified | - 3 weeks run in | Please see the following Google Drive for further details or any missing information:<br>https://drive.eoogle.com/open?id=1WPG-liferent/IdaReftTcuft-VConbible-eft/ | Ofterla |
| | EXPOSURE vs. COMPARISON | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Pull ICD-10 code lists will be swifiable in the above Google Drive Folder (files above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping: <a href="https://www.nbsr.ors/data/Icd9-Icd-10-cm-and-pc-c-crosswall-general-equivalence-mapping.html">https://www.nbsr.ors/data/Icd9-Icd-10-cm-and-pc-c-crosswall-general-equivalence-mapping.html</a> | Adequate mapping in claims |
| | ONTARGET: Aimed to determine if the combination of ARB(Telmisartan) and the ACB (ramipril) is more effective than namipril alone, and if telmisartan is at least as effective as ramipril | Telmisartan vs Ramipril (Exclude patients who received any ACE-I or ARB in prior) | | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | | Poor mapping or cannot be measured in claims |
| | Death from cardiovascular causes, myocardial infection, stroke, or hospitalization for heart failure. | Measure of 1 days after drug initiation in diagnosis position specified below and impattent care set thing. Gemostife in patient mortality/MidStroke/CVF — Hospital admission for CHE (inpetient only, any position) ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 ME (inpetient only, any position) ICD-9 diagnosis: 410.x excluding 410.x2 Stroke (inpetient only, primary position only) ICD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.xx (excluding 434.x0), 436.x Mortality-See Mortality Sheet. | For MI: +PPV 94% in Medicare claims data (Uyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DM, Accuracy of Medicare claims-based diagnosis of acute myocardial inferaction: estimating positive predictive value on the basis of review of hospital records. American heart Journal 2004;148:99-104.] +PPV 98.4% in commercially-insured population (Wahl) PM, Rodgars X, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacocypidemiology and Drug Safety 2010;19:596-603.] For strolla: PPV of BS % or higher for ischemic stroks PPV of BS % or higher for ischemic stroks PPV of BS % or higher for ischemic stroks * (Andrade SE, Herroid LE, T) is), et al. A systematic review of validated methods for identifying carebrovascular acident for transfert inchemic estack using administrative data. Pharmacocypidemiology and Drug Safety 2012;21 Suppl 1:100-38.] † (Transheell DL, Longstreth WT, Ir. Validating administrative data in trioka research. Stroke; a journal of carebral circulation 1200;3:32-865-70.] † (Bournal of C., Mitchel E, Gléson PS, Versa-Lorenzo C, Castellasgue J, Griffin MR. Validation of LOOG Goods with high positive productive values for incident strokes resulting in hospitalization using Medicald health data. Pharmacocypidemiology and drug safety 1008;17:20-6.] | Can't be measured in claims but not important for the analysis |
| | INCLUSION CRITERIA | | | |
| | | Age 255 years at drug initiation | | |
| 10 | Coronary artery disease Previous myocardial Infraction ( > 2 days post uncomplicated Mi) | Measured from the start of all available data to 2 days prior to drug initiation in any diagnosis position and the impatient or outpetient care setting<br>Acute MI ICD-9 diagnosis: 410.xx<br>Old MI ICD-9 diagnosis: 412.xx | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canagilifodin various other non-gillifodin antidiabetic drugs: population based cohort study." BMU 2018;180:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagilifodin and the Risk of Heart Failure Mospitalization in Routine Clinical Care & First Analysis from the Empagilifodin Comparative Effectiveness and Safety (EMP RISE) Study. "Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 | |
| 1b | Stable angins or unstable angins > 30 days before informed consent and with documented evidence of multivessel coronary artery disease | Measured from the start of all available data to 30 days prior to drug initiation in<br>any disgnosts position and the inpatient or outpetient care setting<br>ACS-Dutable spaning ICP-9 diagnosis: 411.xx<br>Stable analog ICP-9 diagnosis: 413.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagilificatin varius other non-gillificatin antidiabetic drugs: population based cohort study." BMU 2018; 360:ki19 http://dx.doi.org/10.1136/bmj.ki19 Patorno, Elisabetta et al. "Empagilificatin and the Risk of Meart Failure Mospitalization in Routine Clinical Care A Pint Analysis from the Empagilificatin Comparative Effectiveness and Safety (IMP RSE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONAMA.118.039177 | |

| ie. | Multi-vessel PTCA >30 days before informed consent: | Measured from the start of all evallable data to 30 days prior to drug initiation in any procedure position and the care setting indicated below: PICA [Inpatient only] CPT-4: 92973, 92982, 92984, 92995, 92996, 92900 – 92921, 92924 – 92925, 92937, 92935, 92941, 92943, 92944 [Inpatient or outpatient] (CD-9 procedure: 00.66, 36.03, 36.03, 36.03, 36.05, 36.05 Starting [Inpatient only] CPT-4: 92980, 92983, 92928 – 92929, 92933 – 92934 [Inpatient or outpatient] (CD-9 procedure: 36.06, 36.07 Transmospatial revesculerization [Inpatient only] CPT-4: 33140, 33141 [Inpatient only] CPT-4: 33140, 33141 [Inpatient or outpatient] ICD-9 procedure: 36.31-36.34 [Inpatient or outpatient] (CD-9 procedure: 36.31-36.34 [Inpatient or outpa | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canagliflosin warsus other non-gliflosin antidiabetic drugs: population based cohort study." SMJ 2018;360kl;19 http://dx.dol.org/10.1136/bmj.kl;19 Patorno, Elisabetta et al. "Empagliflosin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care. A Pint Analysis from the Empagliflosin Comparative Effectiveness and Safety (GMPRSI) Study." Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONAMA.118.039177 |
|---|---|---|---|
| 1d | Multi-vessel CASG surgery > 4 years before informed consent, or with recurrent angina following surgery | Initiation in any procedure position and the inpatient care setting<br>CANG<br>07-4: 33510 – 33536, 33545, 33572.<br>ICD-9 procedure: 36.1x, 36.2x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagificatin versus other non-gliftodin antidiabetic drugs: population based cohort study." EMJ 2018;360:k119 http://dx.dol.org/10.1136/kmj.k119 Patorno, Elisabetta et al. "Empagificatin and the Risk of Neart Fallure Hospitalization in Routine Clinical Care. A First Analysis from the Empagificatin Comparative Effectiveness and Safety (EMPS) 25-bdy. "Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONANA.118.039177 |
| 2 | Peripheral artery disease | | |
| 2a | Previous limb bypass surgery or Previous limb bypass surgery or angioplasty | Measured from the start of all swellable data prior to and including day of drug initiation in any procedure position and the inpatient or outpetient care setting Previous limb beas as surreary or antipolasty CPT-4: 35556, 35566, 35570, 35572, 35583-35587, 35623, 35595, 35666, 35671 [Cover-estermity endarterectomy, stanting, angionisty, or atherentomy ICD-9 procedure; 38.18, 38.19 [Outpetient only] CPT-4: 35454, 35456, 35459, 35470, 35470, 35473, 35474, 35482, 35483, 35484, 35482, 35493, 35495, 37207, 37208, 37220-327235 [Cover-estremity breas: ICD-9 procedure; 38.23, 39.29 [Outpetient only] CPT-4: 35351, 35354, 35351, 35363, 35583, 35563, 35565, 355563, 35567, 35567, 35571, 35572, 35572, 3557 | |
| 2b | Previous limb or foot amputation | Measured from the start of all evaluable data prior to and including day of drug initiation in any diagnosis/procedure position and the inpetient or outpetient care setting Lower extremity expendiction (ICD-0 diagnosis: VM2.7s (excluding VM9.76, V49.77) ICD-0 procedure: 84.10-84.18 (ICD-0 diagnosis: VM2.7s (excluding VM9.76, V49.77) ICD-0 procedure: 84.10-84.18 (ICD-0 diagnosis: VM2.7s (excluding VM9.76, V49.77) ICD-0 procedure: 84.10-84.18 (ICD-0 diagnosis: VM2.7s ( | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canagificatin various other non-gliffodin antidiabetic drugs: population based cohort study." BMJ 2015;56:k119 http://dx.dol.org/10.1136/kmj.k119 Patorno, Elisabetta et al. "Empagificatin and the Blak of Heart Fallure Hospitalization in Routine Clinical Care. A First Analysis from the Empagificatin Comparative Effectiveness and Safety (0x49-0x3) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| 2e | Intermittent claudication, with anklacarm SP ratio <<0.50 on at least 1 side | Measured from the start of all evaluable data prior to and including day of drug<br>initiation in any diagnosis position and the inputient or outpetient care setting<br>Atheroscience of makes exteries of the extremities with intermittent claudication.<br>ICD-9 diagnosis: 440.21 | |
| 2d | Significant peripheral artery stenosis (>50%) documented by angiography or non-invasive testing Core-broveccular disease | Measured from the start of all evaluable data prior to and including day of drug initiation as at least two claims on as parate days in any diagnosis/procedure position and the inputation or outpetient care setting (unless otherwise specified): Protobard vaccular disease. ICD-9 diagnosis: 440.20 – 440.24, 440.29 – 440.32, 440.3, 440.4, 443.9 | Patorno, Elizabetta et al. "Cardiovaccular outcomes associated with canagliflodin varius other non-gliflodin antidiabetic drugs: population based cohort study." SMJ 2018;350:Kl19 http://dx.dol.org/10.1136/bmj.kl19 Patorno, Elizabetta et al. "Empagliflogin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflodin Comparative Effectiveness and Safety (CMPRSE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONAMA.118.039177 |

| _ | | | |
|---|---|---|---|
| 3a | Previous stroke | Measured from the start of all evallable data prior to and including day of drug initiation in any diagnosis position and the inpatient or outpetient care setting Stroke ICD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.xx (excluding 434.x0), 436.x | Patorno, Elizabetta et al. "Cardiovaccular outcomes associated with canagifficatin versus other non-gifficatin actidishetic drugs population based cohort study." BMJ 2018;390:113 http://dx.doi.org/10.1136/pml.113 Patorno, Elizabetta et al. "Empagifficatin and the Risk of Heart Fallure Hospitalization in Routins-Clinical Care. A First Analysis from the Empagifficatin Comparative Effectiveness and Safety (EMPSIS Study." Circulation. 2019 Apr 8. doi: 10.1161/CRCULATIONAMA.118.039177 |
| 3b | Transient ischemic attacks >7 days and <1 year before informed consent | Measured S65 days prior to drug initiation to 7 days prior to drug initiation in any<br>diagnosis position and the inpatient or outpatient care setting<br>TIA ICD-9 diagnosis: 425.xx | |
| 4 | Diabetus mellitus | | |
| 3e | Diabetes mellitus High-risk diabetics with evidence of endorgen demage | Measured at the start of all evaluable data prior to and including day of drug inhibition in any diagnosis position and the lispatient or outpetient care setting Diabetic retinopathy ICD-9 diagnosis: 362.0s. Diabetic swith other ophthalmic manifestations ICD-9 diagnosis: 250.5x (without maniford 952.0-362.07), 366.41, 365.44 Diabetic necknosthy ICD-9 diagnosis: 250.4x, 353.81 Diabetic necknosthy ICD-9 diagnosis: 250.6x, 357.2x, 337.1 Diabetic host NCD-9 diagnosis: 707.1x | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canagiffodin wrass other non-glificolin antidiabetic drugs: population based cohort study." EMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagiffodin and the Risk of Heart Fallure Hospitalization in Routine-Clinical Care: A First Analysis from the Empagiffodin Comparative Effectiveness and Safety (EMPRESE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| | | Exclusion criteria | |
| 1 | Medication use | | |
| 1a | Inability to discontinue ACE inhibitors or ARB | N/A | |
| 1b | Known hypersensitivity or intolerance to ACE inhibitors or ARB (patient intolerant of ACE inhibitor can be enrolled in<br>TRANSCEND) | N/A | |
| 2 | Cardiovacular disease (HF) | | |
| 2a | Symptomatic congestive heart fallure | Measured 180 days prior to and incuding day of drug initiation in any diagnosis position and the lapstantin femapraper cyrono crass setting—theart failure diserrois resulting to be calculated in ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.01, 402.91, 404.01, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93, 404.13, 404.93, 404.13, 404.93, 405.01, 105.02, 105 | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canagiffodin versus other non-gliffodin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagiffodin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagiffodin Comparative Effectiveness and Safety (IMP 1923) Study." Circulation. 2019 Apr 8. doi: 10.1161/GROUATOMAMALIS.09177 |
| 25 | Hiemodynamically significant primary valvular or outflow tract obstruction | Measure d 180 days prior to and incuding day of drug initiation in any diagnosis position and the inpatient or outpatient care setting Vintricular sectial defect (ICD-0 diagnosis: 745.4x Historitoshic Cardiamonoshik (CD-0 diagnosis: 425.1x Stantificant valvolar heart disease ICD-0 diagnosis: 394.x, 395.x, 397.x, 398.9x, V42.2, V43.3 ICD-0 procedure: 33.1x, 35.5x CD-14: 33660-33663, 33400-33403, 33405, 33420-33430, 33460, 33463-33468, 33475, 33496, 02577, 02587, 02597, 02627 | |
| 25 | Hiemodynamically significant primary velvular or outflow tract obstruction Constrictive pericarditis | position and the inputient or outpetient care setting Verticular securi didect (ICD-0 diagnosis: 745.4x Ilavostrophic Cardiomonathy (ICD-0 diagnosis: 425.1x Sizelficant valvoiar heart disease ICD-0 diagnosis: 394.x, 395.x, 396.x, 397.x, 398.9x, V42.2, V43.3 ICD-0 procedure: 35.1x, 35.2x OT+1: 33660-33605, 33400-334403, 33405, 33420-33430, 33460, 33463-33468, | |

| | | Measured 90 days prior to and incuding day of drug initiation in any diagnosis | |
|---|---|---|---|
| | | position and the Inpatient or outpatient care setting<br>Syncope and collapse ICD-9 diagnosis: 780.2 | |
| 2e | Syncopal aplaces of unknown attology <3 months before informed consent | Syncope and conlegate (CD-9 diagnosis: 780.2 | |
| 1 | | | |
| 39 | Planned cardiac surgery or PTCA-G months of informed consent | N/A | |
| | Processing Contract State State Contract Contrac | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpatient care setting | |
| 246 | Uncontrolled hypertension on treatment (eg. BP >160/100 mm Hg) | Mailgnant Hypertansion ICD-9 diagnosis: 401.0, 402.0, 402.00, 402.01, 403.0, | |
| | | 403.00, 403.01, 404.0, 404.00, 404.01, 404.02, 404.03, 405.0, 405.01, 405.09 | |
| | | Measured 180 days prior to and incuding day of drug initiation in any | |
| 1 | | diagnosis/procedure position and the inpetient or outpetient care setting | |
| 25 | Heart transplant recipient | Heart transplantation | |
| - | | ICD-9 diagnosis: V42.1<br>ICD-9 procedure: 37.51 | |
| 1 | | The special state of the state | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpetient care setting | |
| 2g | Stroke due to suberechnoid hemorrhage | Subarachnold hemorrhage (SAH) ICD-9 diagnosis: 430.xx | |
| Ц_ | | | |
| 3 | Other conditions | | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| 3a | Significant renal enterly disease | position and the inpatient or outpatient care setting | |
| Ь— | | Renovascular hypertension ICD-9 diagnosis: 405.01, 405.11, 405.91, 440.1 | |
| l l | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| I | apatic dynfunction | position and the inpatient or outpatient care setting<br>Hepatitis ICD-9 diagnosis: 070.0, 070.1, 070.20, 070.21, 070.30, 070.31, 070.41, | |
| 3b | | 070.51 | |
| | | Chronic liver disease and cirrhosis ICD-9 diagnosis: 571.x, 572.x, 573.x | |
| l | | | |
| <u>9e</u> | Uncorrected volume or sodium depletion | N/A | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpatient care setting | |
| 34 | Primary hyperaldosteronism | Hyperaldosteronism ICD-9 diagnosis: 255.10 | |
| l | | | |
| ${f \Box}$ | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | Hamaditan Sandan Intelement | position and the inpatient or outpatient care setting | |
| * | Hereditary fructose Intolerance | Hereditary Fructose Intolerance ICD-9 diagnosis: 271.2 | |
| Ь | | | |
| ı | | | Gagne, Josh J et. al. ""A combined comorbidity score predicted mortality in elderly |
| l l | | | patients better than existing scores." J Clin Epidemiol. 2011 Jul;64(7):749-59. doi: |
| l | Other major noncardiac illness expected to reduce life expectancy or interfere with study participation | Measured 180 days prior to and including day of drug initiation- | 10.1016/j.jclinepi.2010.10.004. |
| 38 | | CC1≥10 | Sun, Jenny W et. al. ""Validation of the Combined Comorbidity Index of Charlson and |
| ı | | | Elixhauser to Predict 30-Day Mortality Across ICD-9 and ICD-10." Med Care. 2018 |
| l l | | | Sep;56(9):812. doi: 10.1097/MLR.000000000000954. |
| 9g | Simultaneously taking another experimental drug | N/A | |
| 3h | Significent disability precluding regular follow-up visits | N/A | |
| 31 | Unable or unwilling to provide written informed consent | N/A | |
| 31 | | | |

| Trial ID | Neg4 |
|---|---|
| Trial Name (with web links) | ONTARGET |
| Trial Name (with pdf links) | <u>ONTARGET</u> |
| <u>NCT</u> | NCT00153101 |
| Trial category | Negative trial |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | Antihypertensives (ARBs+aliskiren) |
| RCT Category | 3- Failed S- No NI margin specified |
| Brand Name | Micardis |
| Generic Name | telmisartan + ramipril |
| <u>Sponsor</u> | Boehringer Ingelheim |
| <u>Year</u> | 2008 |
| Measurable endpoint | Primary composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fa |
| Weasurable enuponic | Stroke and Hospitalization for Congestive Heart Failure |
| <u>Exposure</u> | Telmisartan |
| <u>Comparator</u> | Ramipril |
| Population | Patients aged 55 years or older with established atherosclerotic vascular disease or with diabetes |
| | with end-organ damage |
| <u>Trial finding</u> | HR = 1.01 (95% CI 0.94–1.09) |
| Notes | |
| No. of Patients | 31546 |
| Non-inferiority margin | Not provided |
| Assay Sens. Outcome | Angioedema |
| Assay Sens. Endpoint (from trial) | Angioedema |
| Finding for potential Assay Sens. Outcome from | |
| <u>trial-</u> | HR, 0.40; P = .01 |
| <u>Power</u> | |
| Blinding | Double-blinded |
| Statistical Method | Non-inferiority margin was 1.13 |

## Mortality-Dependent on data source. All-cause mortality / inpatient mortality Identified using the vital status file-Medicare Identified using the discharge status codes-Optum-20 = EXPIRED 21 = EXPIRED TO BE DEFINED AT STATE LEVEL 22 = EXPIRED TO BE DEFINED AT STATE LEVEL 23 = EXPIRED TO BE DEFINED AT STATE LEVEL 24 = EXPIRED TO BE DEFINED AT STATE LEVEL 25 = EXPIRED TO BE DEFINED AT STATE LEVEL 26 = EXPIRED TO BE DEFINED AT STATE LEVEL 27 = EXPIRED TO BE DEFINED AT STATE LEVEL 28 = EXPIRED TO BE DEFINED AT STATE LEVEL 29 = EXPIRED TO BE DEFINED AT STATE LEVEL 40 = EXPIRED AT HOME (HOSPICE) 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE) 42 = EXPIRED - PLACE UNKNOWN (HOSPICE) Truven- 20 - Died 22 - Died 23 - Died 24 - Died 25 - Died 26 - Died 27 - Died 28 - Died 29 - Died 40 - Other died status or Expired at home (Hospice claims only) (depends on year) 41 - Other died status or Expired in medical facility (Hospice claims only) (depends on year) 42 - Other died status or Expired - place unknown (Hospice claims only) (depends on year) 21 - Died or Disch./Transf. to court/law enforcement (depends on year)

## Appendix B







Table 1: Telmisartan vs Ramipril

| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Орг | tum | | Tru | | | POO | LED | |
| Variable | Ramipril (Any dose) | Telmisartan (Any dose) | St. Diff. | Ramipril (Any dose) | Telmisartan (Any | St. Diff. | Ramipril (Any dose) | Telmisartan (Any | |
| Number of patients | 37,963 | 11,955 | | 92,821 | 21,871 | | 130,784 | 33,826 | |
| Age | | | | | | | | | |
| mean (sd) | 68.65 (9.21) | 69.57 (9.24) | -0.10 | 68.25 (9.67) | 68.60 (9.78) | -0.04 | 68.37 (9.54) | 68.94 (9.59) | -0.06 |
| median [IQR] | 68.00 [61.00, 75.00] | 69.00 [62.00, 76.00] | -0.11 | 66.00 [60.00, 76.00] | 67.00 [60.00, 76.00] | -0.10 | 66.58 (9.54) | 67.71 (9.59) | -0.12 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| 55 - 64; n (%) | 14,313 (37.7%) | 3,963 (33.1%) | 0.10 | 42,090 (45.3%) | 9,615 (44.0%) | 0.03 | 56,403 (43.1%) | 13,578 (40.1%) | 0.06 |
| 65 - 74; n (%) | 13,132 (34.6%) | 4,251 (35.6%) | -0.02 | 24,764 (26.7%) | 5,807 (26.6%) | 0.00 | 37,896 (29.0%) | 10,058 (29.7%) | -0.02 |
| ≻=75; n (%) | 10,518 (27.7%) | 3,741 (31.3%) | -0.08 | 25,967 (28.0%) | 6,449 (29.5%) | -0.03 | 36,485 (27.9%) | 10,190 (30.1%) | -0.05 |
| Gender | | | | | | | | | |
| Males; n (%) | 23,547 (62.0%) | 5,225 (43.7%) | 0.37 | 57,804 (62.3%) | 9,926 (45.4%) | 0.34 | 81,351 (62.2%) | 15,151 (44.8%) | 0.35 |
| Females; n (%) | 14,416 (38.0%) | 6,730 (56.3%) | -0.37 | 35,017 (37.7%) | 11,945 (54.6%) | -0.34 | 49,433 (37.8%) | 18,675 (55.2%) | -0.35 |
| Region | | | | | | | | | |
| Northeast; n (%) | 6,036 (15.9%) | 1,167 (9.8%) | 0.18 | 20,614 (22.2%) | 3,034 (13.9%) | 0.22 | 26,650 (20.4%) | 4,201 (12.4%) | 0.22 |
| South; n (%) | 20,157 (53.1%) | 7,419 (62.1%) | -0.18 | 25,327 (27.3%) | 5,130 (23.5%) | 0.09 | 45,484 (34.8%) | 12,549 (37.1%) | -0.05 |
| Midwest; n (%) | 5,635 (14.8%) | 1,385 (11.6%) | 0.09 | 36,314 (39.1%) | 10,403 (47.6%) | -0.17 | 41,949 (32.1%) | 11,788 (34.8%) | -0.06 |
| West; n (%) | 6,135 (16.2%) | 1,984 (16.6%) | -0.01 | 9,966 (10.7%) | 3,170 (14.5%) | -0.11 | 16,101 (12.3%) | 5,154 (15.2%) | -0.08 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 600 (0.6%) | 134 (0.6%) | 0.00 | 600 (0.5%) | 134 (0.4%) | 0.01 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 19,508 (51.4%) | 3,708 (31.0%) | 0.42 | 45,103 (48.6%) | 6,024 (27.5%) | 0.45 | 64,611 (49.4%) | 9,732 (28.8%) | 0.43 |
| Acute MI; n (%) | 4,164 (11.0%) | 217 (1.8%) | 0.38 | 10,774 (11.6%) | 344 (1.6%) | 0.41 | 14938 (11.4%) | 561 (1.7%) | 0.40 |
| ACS/unstable angina; n (%) | 3,085 (8.1%) | 327 (2.7%) | 0.24 | 7,863 (8.5%) | 666 (3.0%) | 0.24 | 10948 (8.4%) | 993 (2.9%) | 0.24 |
| Old MI; n (%) | 3,612 (9.5%) | 516 (4.3%) | 0.21 | 3,971 (4.3%) | 354 (1.6%) | 0.16 | 7583 (5.8%) | 870 (2.6%) | 0.16 |
| Stable angina; n (%) | 3,884 (10.2%) | 824 (6.9%) | 0.12 | 7,781 (8.4%) | 1,206 (5.5%) | 0.11 | 11,665 (8.9%) | 2,030 (6.0%) | 0.11 |
| Coronary atherosclerosis and other forms<br>of chronic ischemic heart disease; n (%) | 18,048 (47.5%) | 3,234 (27.1%) | 0.43 | 40,383 (43.5%) | 5,175 (23.7%) | 0.43 | 58,431 (44.7%) | 8,409 (24.9%) | 0.42 |
| Other atherosclerosis with ICD10; n (%) | 1,228 (3.2%) | 218 (1.8%) | 0.09 | 2,275 (2.5%) | 358 (1.6%) | 0.06 | 3503 (2.7%) | 576 (1.7%) | 0.07 |
| Previous cardiac procedure (CABG or PTCA | 3,749 (9.9%) | 141 (1.2%) | 0.39 | 8,424 (9.1%) | 293 (1.3%) | 0.36 | 12173 (9.3%) | 434 (1.3%) | 0.36 |
| or Stent); n (%) | 5,7 15 (5.576) | 212(2.27) | 0.55 | 5,121(5.276) | 255 (2.576) | 0.50 | 22273 (3.376) | 131 (2.374) | 0.50 |
| History of CABG or PTCA; n (%) | 5,500 (14.5%) | 791 (6.6%) | 0.26 | 5,538 (6.0%) | 526 (2.4%) | 0.18 | 11,038 (8.4%) | 1,317 (3.9%) | 0.19 |
| Any stroke; n (%) | 6,534 (17.2%) | 1,771 (14.8%) | 0.07 | 15,361 (16.5%) | 3,048 (13.9%) | 0.07 | 21,895 (16.7%) | 4,819 (14.2%) | 0.07 |
| Ischemic stroke (w and w/o mention of | 6,483 (17.1%) | 1,758 (14.7%) | 0.07 | 15,281 (16.5%) | 3,024 (13.8%) | 0.08 | 21,764 (16.6%) | 4,782 (14.1%) | 0.07 |
| cerebral infarction); n (%) | | | | | | | | | |
| Hemorrhagic stroke; n (%) | 155 (0.4%) | 39 (0.3%) | 0.02 | 302 (0.3%) | 60 (0.3%) | 0.00 | 457 (0.3%) | 99 (0.3%) | 0.00 |
| TIA; n (%) | 1,799 (4.7%) | 502 (4.2%) | 0.02 | 4,340 (4.7%) | 854 (3.9%) | 0.04 | 6139 (4.7%) | 1356 (4.0%) | 0.03 |
| Other cerebrovascular disease; n (%) | 1,361 (3.6%) | 366 (3.1%) | 0.03 | 2,392 (2.6%) | 467 (2.1%) | 0.03 | 3753 (2.9%) | 833 (2.5%) | 0.02 |
| Late effects of cerebrovascular disease; n | 1,141 (3.0%) | 280 (2.3%) | 0.04 | 1,693 (1.8%) | 296 (1.4%) | 0.03 | 2834 (2.2%) | 576 (1.7%) | 0.04 |
| (%) | | | | | | | | | |
| Cerebrovascular procedure; n (%) | 183 (0.5%) | 36 (0.3%) | 0.03 | 460 (0.5%) | 87 (0.4%) | 0.01 | 643 (0.5%) | 123 (0.4%) | 0.01 |
| Heart failure (CHF); n (%) | 4,149 (10.9%) | 901 (7.5%) | 0.12 | 6,644 (7.2%) | 1,019 (4.7%) | 0.11 | 10,793 (8.3%) | 1,920 (5.7%) | 0.10 |
| Peripheral Vascular Disease (PVD) or PVD | 4,262 (11.2%) | 1,255 (10.5%) | 0.02 | 7,315 (7.9%) | 1,563 (7.1%) | 0.03 | 11,577 (8.9%) | 2,818 (8.3%) | 0.02 |
| Surgery; n (%) | | | | | | | | | |
| Atrial fibrillation; n (%) | 3,981 (10.5%) | 938 (7.8%) | 0.09 | 8,576 (9.2%) | 1,430 (6.5%) | 0.10 | 12,557 (9.6%) | 2,368 (7.0%) | 0.09 |
| Other cardiac dysrhythmia; n (%) | 5,611 (14.8%) | 1,339 (11.2%) | 0.11 | 10,682 (11.5%) | 1,720 (7.9%) | 0.12 | 16,293 (12.5%) | 3,059 (9.0%) | 0.11 |

Table 1: Telmisartan vs Ramipril

| Cardiac conduction disorders; n (%) Other CVD; n (%) Diabetes-related complications | 1,740 (4.6%)<br>7,644 (20.1%) | 360 (3.0%)<br>1,732 (14.5%) | 0.08<br>0.15 | 2,943 (3.2%)<br>16,519 (17.8%) | 394 (1.8%)<br>2,560 (11.7%) | 0.09<br>0.17 | 4683 (3.6%) | 754 (2.2%) | 0.08 |
|---|---|---|---|---|---|---|---|---|---|
| Diabetes-related complications | 7,644 (20.1%) | 1,732 (14.5%) | 0.15 | 16 519 (17 8%) | 2 ECD (44 70/) | 0.17 | OR ACT (AC CO) | 4 000 (40 TO/) | |
| | | | | 10,515 (17.670) | 2,560 (11.7%) | 0.17 | 24,163 (18.5%) | 4,292 (12.7%) | 0.16 |
| Diabetic retinopathy; n (%) | 2,266 (6.0%) | 735 (6.1%) | 0.00 | 3,866 (4.2%) | 835 (3.8%) | 0.02 | 6,132 (4.7%) | 1,570 (4.6%) | 0.00 |
| Diabetes with other ophthalmic manifestations; n (%) | 128 (0.3%) | 60 (0.5%) | -0.03 | 2,595 (2.8%) | 586 (2.7%) | 0.01 | 2,723 (2.1%) | 0,646 (1.9%) | 0.01 |
| Retinal detachment, vitreous hemorrhage, vitrectomy; n (%) | 214 (0.6%) | 63 (0.5%) | 0.01 | 344 (0.4%) | 79 (0.4%) | 0.00 | 558 (0.4%) | 142 (0.4%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 309 (0.8%) | 93 (0.8%) | 0.00 | 832 (0.9%) | 178 (0.8%) | 0.01 | 1141 (0.9%) | 271 (0.8%) | 0.01 |
| Occurrence of Diabetic Neuropathy; n (%) | 4,676 (12.3%) | 1,528 (12.8%) | -0.02 | 6,411 (6.9%) | 1,417 (6.5%) | 0.02 | 11,087 (8.5%) | 2,945 (8.7%) | -0.01 |
| Occurrence of diabetic nephropathy with ICD10; n (%) | 2,627 (6.9%) | 1,065 (8.9%) | -0.07 | 2,726 (2.9%) | 745 (3.4%) | -0.03 | 5,353 (4.1%) | 1,810 (5.4%) | -0.06 |
| Hypoglycemia; n (%) | 760 (2.0%) | 159 (1.3%) | 0.05 | 1,607 (1.7%) | 309 (1.4%) | 0.02 | 2,367 (1.8%) | 0,468 (1.4%) | 0.03 |
| Hyperglycemia; n (%) | 1,254 (3.3%) | 430 (3.6%) | -0.02 | 1,298 (1.4%) | 312 (1.4%) | 0.00 | 2,552 (2.0%) | 0,742 (2.2%) | -0.01 |
| Disorders of fluid electrolyte and acid-base | 2,764 (7.3%) | 873 (7.3%) | 0.00 | 4,269 (4.6%) | 866 (4.0%) | 0.03 | 7,033 (5.4%) | 1,739 (5.1%) | 0.01 |
| balance; n (%) | | | | | | | | | |
| Diabetic ketoacidosis; n (%) | 152 (0.4%) | 22 (0.2%) | 0.04 | 269 (0.3%) | 27 (0.1%) | 0.04 | 421 (0.3%) | 49 (0.1%) | 0.04 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 107 (0.3%) | 25 (0.2%) | 0.02 | 145 (0.2%) | 25 (0.1%) | 0.03 | 252 (0.2%) | 50 (0.1%) | 0.03 |
| Diabetes with peripheral circulatory disorders with ICD-10; n (%) | 1,596 (4.2%) | 482 (4.0%) | 0.01 | 2,032 (2.2%) | 364 (1.7%) | 0.04 | 3,628 (2.8%) | 0,846 (2.5%) | 0.02 |
| Diabetic Foot; n (%) | 1,161 (3.1%) | 319 (2.7%) | 0.02 | 2,589 (2.8%) | 586 (2.7%) | 0.01 | 3750 (2.9%) | 905 (2.7%) | 0.01 |
| Gangrene; n (%) | 121 (0.3%) | 22 (0.2%) | 0.02 | 243 (0.3%) | 24 (0.1%) | 0.04 | 364 (0.3%) | 46 (0.1%) | 0.04 |
| Lower extremity amputation; n (%) | 239 (0.6%) | 66 (0.6%) | 0.00 | 350 (0.4%) | 45 (0.2%) | 0.04 | 589 (0.5%) | 111 (0.3%) | 0.03 |
| Osteomyelitis; n (%) | 307 (0.8%) | 62 (0.5%) | 0.04 | 612 (0.7%) | 91 (0.4%) | 0.04 | 919 (0.7%) | 153 (0.5%) | 0.03 |
| Skin infections; n (%) | 2,117 (5.6%) | 635 (5.3%) | 0.01 | 5,025 (5.4%) | 1,101 (5.0%) | 0.02 | 7,142 (5.5%) | 1,736 (5.1%) | 0.02 |
| Erectile dysfunction; n (%) | 1,035 (2.7%) | 317 (2.7%) | 0.00 | 1,359 (1.5%) | 275 (1.3%) | 0.02 | 2,394 (1.8%) | 0,592 (1.8%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 969 (2.6%) | 316 (2.6%) | 0.00 | 1,763 (1.9%) | 342 (1.6%) | 0.02 | 2,732 (2.1%) | 0,658 (1.9%) | 0.01 |
| (79) Diabetes mellitus without mention of complications; n (%) | 16,496 (43.5%) | 5,002 (41.8%) | 0.03 | 34,936 (37.6%) | 7,565 (34.6%) | 0.06 | 51,432 (39.3%) | 12,567 (37.2%) | 0.04 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 27,935 (73.6%) | 10,512 (87.9%) | -0.37 | 48,516 (52.3%) | 15,315 (70.0%) | -0.37 | 76,451 (58.5%) | 25,827 (76.4%) | -0.39 |
| Hyperlipidemia ; n (%) | 25,720 (67.8%) | 7,595 (63.5%) | 0.09 | 37,915 (40.8%) | 8,384 (38.3%) | 0.05 | 63,635 (48.7%) | 15,979 (47.2%) | 0.03 |
| Edema; n (%) | 2,181 (5.7%) | 1,016 (8.5%) | -0.11 | 3,441 (3.7%) | 1,012 (4.6%) | -0.05 | 5,622 (4.3%) | 2,028 (6.0%) | -0.08 |
| Renal Dysfunction (non-diabetic) ; n (%) | 5,308 (14.0%) | 2,309 (19.3%) | -0.14 | 7,474 (8.1%) | 2,213 (10.1%) | -0.07 | 12,782 (9.8%) | 4,522 (13.4%) | -0.11 |
| Occurrence of acute renal disease ; n (%) | 862 (2.3%) | 295 (2.5%) | -0.01 | 1,360 (1.5%) | 303 (1.4%) | 0.01 | 2222 (1.7%) | 598 (1.8%) | -0.01 |
| Occurrence of chronic renal insufficiency;<br>n (%) | 3,832 (10.1%) | 1,818 (15.2%) | -0.15 | 4,683 (5.0%) | 1,543 (7.1%) | -0.09 | 8,515 (6.5%) | 3,361 (9.9%) | -0.12 |
| Chronic kidney disease ; n (%) | 3,530 (9.3%) | 1,739 (14.5%) | -0.16 | 4,116 (4.4%) | 1,430 (6.5%) | -0.09 | 7,646 (5.8%) | 3,169 (9.4%) | -0.14 |
| CKD Stage 3-4; n (%) | 2,087 (5.5%) | 1,181 (9.9%) | -0.17 | 2,245 (2.4%) | 893 (4.1%) | -0.10 | 4,332 (3.3%) | 2,074 (6.1%) | -0.13 |
| Occurrence of hypertensive nephropathy;<br>n (%) | 1,681 (4.4%) | 912 (7.6%) | -0.14 | 1,616 (1.7%) | 592 (2.7%) | -0.07 | 3297 (2.5%) | 1504 (4.4%) | -0.10 |
| Occurrence of miscellaneous renal insufficiency; n (%) | 1,850 (4.9%) | 712 (6.0%) | -0.05 | 3,018 (3.3%) | 754 (3.4%) | -0.01 | 4,868 (3.7%) | 1,466 (4.3%) | -0.03 |
| Glaucoma or cataracts ; n (%) | 6,825 (18.0%) | 2,530 (21.2%) | -0.08 | 14,801 (15.9%) | 3,941 (18.0%) | -0.06 | 21,626 (16.5%) | 6,471 (19.1%) | -0.07 |
| Cellulitis or abscess of toe; n (%) | 460 (1.2%) | 136 (1.1%) | 0.01 | 792 (0.9%) | 145 (0.7%) | 0.02 | 1252 (1.0%) | 281 (0.8%) | 0.02 |

Table 1: Telmisartan vs Ramipril

| Bladder stones; n (%) Kidney stones; n (%) Urinary tract infections (UTIs); n (%) Dipstick urinalysis; n (%) Non-dipstick urinalysis; n (%) Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Falls; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hyperthyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) SleepDisorder; n (%) Dementia; n (%) | 58 (0.2%) 728 (1.9%) 3,325 (8.8%) 12,280 (32.3%) 7,839 (20.6%) 1,152 (3.0%) 572 (1.5%) 773 (2.0%) 633 (1.7%) 5,538 (14.6%) 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 16 (0.1%) 250 (2.1%) 1,215 (10.2%) 4,415 (36.9%) 2,658 (22.2%) 335 (2.8%) 146 (1.2%) 231 (1.9%) 298 (2.5%) 2,189 (18.3%) 4,673 (39.1%) 2,886 (24.1%) 426 (3.6%) 386 (3.2%) 1,053 (8.8%) 103 (0.9%) | 0.03<br>-0.01<br>-0.05<br>-0.10<br>-0.04<br>0.01<br>0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09<br>-0.01<br>-0.02 | 121 (0.1%) 1,685 (1.8%) 5,653 (6.1%) 21,781 (23.5%) 11,042 (11.9%) 3,048 (3.3%) 1,723 (1.9%) 2,146 (2.3%) 776 (0.8%) 10,078 (10.9%) 27,287 (29.4%) 15,687 (16.9%) 3,257 (3.5%) | 22 (0.1%)<br>358 (1.6%)<br>1,384 (6.3%)<br>5,317 (24.3%)<br>2,434 (11.1%)<br>705 (3.2%)<br>321 (1.5%)<br>442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%)<br>4,425 (20.2%) | 0.00<br>0.02<br>-0.01<br>-0.02<br>0.03<br>0.01<br>0.03<br>0.02<br>0.01<br>-0.07<br>-0.07 | 179 (0.1%) 2,413 (1.8%) 8,978 (6.9%) 34,061 (26.0%) 18,881 (14.4%) 4,200 (3.2%) 2295 (1.8%) 2919 (2.2%) 1,409 (1.1%) 15,616 (11.9%) 40,452 (30.9%) | 38 (0.1%)<br>0,608 (1.8%)<br>2,599 (7.7%)<br>9,732 (28.8%)<br>5,092 (15.1%)<br>1,040 (3.1%)<br>467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%)<br>11,786 (34.8%) | 0.00<br>0.00<br>-0.03<br>-0.06<br>-0.02<br>0.01<br>0.03<br>0.01<br>-0.03<br>-0.09<br>-0.08 |
|---|---|---|---|---|---|---|---|---|---|
| Urinary tract infections (UTIs); n (%) Dipstick urinalysis; n (%) Non-dipstick urinalysis; n (%) Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Practures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypethyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) SleepDisorder; n (%) Dementia; n (%) | 3,325 (8.8%) 12,280 (32.3%) 7,839 (20.6%) 1,152 (3.0%) 572 (1.5%) 773 (2.0%) 633 (1.7%) 5,538 (14.6%) 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 1,215 (10.2%) 4,415 (36.9%) 2,658 (22.2%) 335 (2.8%) 146 (1.2%) 231 (1.9%) 298 (2.5%) 2,189 (18.3%) 4,673 (39.1%) 2,886 (24.1%) 426 (3.6%) 386 (3.2%) 1,053 (8.8%) | -0.05<br>-0.10<br>-0.04<br>0.01<br>0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09 | 5,653 (6.1%)<br>21,781 (23.5%)<br>11,042 (11.9%)<br>3,048 (3.3%)<br>1,723 (1.9%)<br>2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%) | 1,384 (6.3%) 5,317 (24.3%) 2,434 (11.1%) 705 (3.2%) 321 (1.5%) 442 (2.0%) 162 (0.7%) 2,895 (13.2%) 7,113 (32.5%) | -0.01<br>-0.02<br>0.03<br>0.01<br>0.03<br>0.02<br>0.01<br>-0.07 | 8,978 (6.9%)<br>34,061 (26.0%)<br>18,881 (14.4%)<br>4,200 (3.2%)<br>2295 (1.8%)<br>2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 2,599 (7.7%)<br>9,732 (28.8%)<br>5,092 (15.1%)<br>1,040 (3.1%)<br>467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | -0.03<br>-0.06<br>-0.02<br>0.01<br>0.03<br>0.01<br>-0.03<br>-0.09 |
| Dipstick urinalysis; n (%) Non-dipstick urinalysis; n (%) Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypethyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) SleepDisorder; n (%) Dementia; n (%) | 12,280 (32.3%) 7,839 (20.6%) 1,152 (3.0%) 572 (1.5%) 773 (2.0%) 633 (1.7%) 5,538 (14.6%) 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 4,415 (36.9%) 2,658 (22.2%) 335 (2.8%) 146 (1.2%) 231 (1.9%) 298 (2.5%) 2,189 (18.3%) 4,673 (39.1%) 2,886 (24.1%) 426 (3.6%) 386 (3.2%) 1,053 (8.8%) | -0.10<br>-0.04<br>0.01<br>0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09 | 21,781 (23.5%)<br>11,042 (11.9%)<br>3,048 (3.3%)<br>1,723 (1.9%)<br>2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 5,317 (24.3%)<br>2,434 (11.1%)<br>705 (3.2%)<br>321 (1.5%)<br>442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | -0.02<br>0.03<br>0.01<br>0.03<br>0.02<br>0.01<br>-0.07 | 34,061 (26.0%)<br>18,881 (14.4%)<br>4,200 (3.2%)<br>2295 (1.8%)<br>2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 9,732 (28.8%)<br>5,092 (15.1%)<br>1,040 (3.1%)<br>467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | -0.06<br>-0.02<br>0.01<br>0.03<br>0.01<br>-0.03<br>-0.09 |
| Non-dipstick urinalysis; n (%) Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) SleepDisorder; n (%) Dementia; n (%) | 7,839 (20.6%) 1,152 (3.0%) 572 (1.5%) 773 (2.0%) 633 (1.7%) 5,538 (14.6%) 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 2,658 (22.2%)<br>335 (2.8%)<br>146 (1.2%)<br>231 (1.9%)<br>298 (2.5%)<br>2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.04<br>0.01<br>0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09 | 11,042 (11.9%)<br>3,048 (3.3%)<br>1,723 (1.9%)<br>2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 2,434 (11.1%)<br>705 (3.2%)<br>321 (1.5%)<br>442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | 0.03<br>0.01<br>0.03<br>0.02<br>0.01<br>-0.07 | 18,881 (14.4%)<br>4,200 (3.2%)<br>2295 (1.8%)<br>2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 5,092 (15.1%)<br>1,040 (3.1%)<br>467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | -0.02<br>0.01<br>0.03<br>0.01<br>-0.03<br>-0.09 |
| Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 1,152 (3.0%) 572 (1.5%) 773 (2.0%) 633 (1.7%) 5,538 (14.6%) 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 335 (2.8%)<br>146 (1.2%)<br>231 (1.9%)<br>298 (2.5%)<br>2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | 0.01<br>0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09 | 3,048 (3.3%)<br>1,723 (1.9%)<br>2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 705 (3.2%)<br>321 (1.5%)<br>442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | 0.01<br>0.03<br>0.02<br>0.01<br>-0.07<br>-0.07 | 4,200 (3.2%)<br>2295 (1.8%)<br>2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 1,040 (3.1%)<br>467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | 0.01<br>0.03<br>0.01<br>-0.03<br>-0.09 |
| Urine function test; n (%) Cytology; n (%) Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 572 (1.5%)<br>773 (2.0%)<br>633 (1.7%)<br>5,538 (14.6%)<br>13,165 (34.7%)<br>7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 146 (1.2%)<br>231 (1.9%)<br>298 (2.5%)<br>2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | 0.03<br>0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09 | 1,723 (1.9%)<br>2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 321 (1.5%)<br>442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | 0.03<br>0.02<br>0.01<br>-0.07<br>-0.07 | 2295 (1.8%)<br>2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 467 (1.4%)<br>673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | 0.03<br>0.01<br>-0.03<br>-0.09 |
| Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 572 (1.5%)<br>773 (2.0%)<br>633 (1.7%)<br>5,538 (14.6%)<br>13,165 (34.7%)<br>7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 231 (1.9%)<br>298 (2.5%)<br>2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | 0.01<br>-0.06<br>-0.10<br>-0.09<br>-0.09<br>-0.01 | 2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 442 (2.0%)<br>162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | 0.02<br>0.01<br>-0.07<br>-0.07 | 2919 (2.2%)<br>1,409 (1.1%)<br>15,616 (11.9%) | 673 (2.0%)<br>0,460 (1.4%)<br>5,084 (15.0%) | 0.01<br>-0.03<br>-0.09 |
| Cystos; n (%) Other Covariates Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 633 (1.7%)<br>5,538 (14.6%)<br>13,165 (34.7%)<br>7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 298 (2.5%)<br>2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.06<br>-0.10<br>-0.09<br>-0.09<br>-0.01 | 2,146 (2.3%)<br>776 (0.8%)<br>10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 162 (0.7%)<br>2,895 (13.2%)<br>7,113 (32.5%) | 0.01<br>-0.07<br>-0.07 | 1,409 (1.1%)<br>15,616 (11.9%) | 0,460 (1.4%)<br>5,084 (15.0%) | -0.03<br>-0.09 |
| Liver disease; n (%) Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 5,538 (14.6%)<br>13,165 (34.7%)<br>7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.10<br>-0.09<br>-0.09<br>-0.01 | 10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 2,895 (13.2%)<br>7,113 (32.5%) | -0.07<br>-0.07 | 15,616 (11.9%) | 5,084 (15.0%) | -0.09 |
| Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 5,538 (14.6%)<br>13,165 (34.7%)<br>7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 2,189 (18.3%)<br>4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.10<br>-0.09<br>-0.09<br>-0.01 | 10,078 (10.9%)<br>27,287 (29.4%)<br>15,687 (16.9%) | 2,895 (13.2%)<br>7,113 (32.5%) | -0.07<br>-0.07 | 15,616 (11.9%) | 5,084 (15.0%) | -0.09 |
| Other arthritis, arthropathies and musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 13,165 (34.7%) 7,713 (20.3%) 1,320 (3.5%) 1,059 (2.8%) 2,577 (6.8%) 264 (0.7%) 5,075 (13.4%) | 4,673 (39.1%)<br>2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.09<br>-0.09<br>-0.01 | 27,287 (29.4%)<br>15,687 (16.9%) | 7,113 (32.5%) | -0.07 | | | |
| musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures, n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 7,713 (20.3%)<br>1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 2,886 (24.1%)<br>426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.09<br>-0.01 | 15,687 (16.9%) | | | 40,452 (30.9%) | 11,786 (34.8%) | -0.08 |
| musculoskeletal pain; n (%) Dorsopathies; n (%) Fractures, n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.01 | 15,687 (16.9%) | 4,425 (20.2%) | _0.00 | | | |
| Dorsopathies; n (%) Fractures; n (%) Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 1,320 (3.5%)<br>1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 426 (3.6%)<br>386 (3.2%)<br>1,053 (8.8%) | -0.01 | | 4,425 (20.2%) | _n ne | | | |
| Falls; n (%) Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | 1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 386 (3.2%)<br>1,053 (8.8%) | | 3.257 (3.5%) | | -0.00 | 23,400 (17.9%) | 7,311 (21.6%) | -0.09 |
| Osteoporosis; n (%) Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 1,059 (2.8%)<br>2,577 (6.8%)<br>264 (0.7%)<br>5,075 (13.4%) | 1,053 (8.8%) | -0.02 | -, () | 735 (3.4%) | 0.01 | 4,577 (3.5%) | 1,161 (3.4%) | 0.01 |
| Hyperthyroidism; n (%) Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 264 (0.7%)<br>5,075 (13.4%) | | | 567 (0.6%) | 136 (0.6%) | 0.00 | 1626 (1.2%) | 522 (1.5%) | -0.03 |
| Hypothyroidism; n (%) Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 5,075 (13.4%) | 103 (0.9%) | -0.07 | 5,906 (6.4%) | 1,733 (7.9%) | -0.06 | 8,483 (6.5%) | 2,786 (8.2%) | -0.07 |
| Other disorders of thyroid gland; n (%) Depression; n (%) Anxiety; n (%) SleepDisorder; n (%) Dementia; n (%) | | | -0.02 | 373 (0.4%) | 103 (0.5%) | -0.01 | 637 (0.5%) | 206 (0.6%) | -0.01 |
| Depression; n (%)<br>Anxiety; n (%)<br>SleepDisorder; n (%)<br>Dementia; n (%) | 1 121 /2 00/ | 1,932 (16.2%) | -0.08 | 6,835 (7.4%) | 1,915 (8.8%) | -0.05 | 11,910 (9.1%) | 3,847 (11.4%) | -0.08 |
| Anxiety, n (%) SleepDisorder; n (%) Dementia; n (%) | 1,131 (3.0%) | 520 (4.3%) | -0.07 | 2,105 (2.3%) | 640 (2.9%) | -0.04 | 3,236 (2.5%) | 1,160 (3.4%) | -0.05 |
| SleepDisorder; n (%)<br>Dementia; n (%) | 2,849 (7.5%) | 890 (7.4%) | 0.00 | 4,424 (4.8%) | 1,054 (4.8%) | 0.00 | 7,273 (5.6%) | 1,944 (5.7%) | 0.00 |
| Dementia; n (%) | 2,267 (6.0%) | 896 (7.5%) | -0.06 | 2,793 (3.0%) | 703 (3.2%) | -0.01 | 5,060 (3.9%) | 1,599 (4.7%) | -0.04 |
| Dementia; n (%) | 2,613 (6.9%) | 902 (7.5%) | -0.02 | 5,740 (6.2%) | 1,789 (8.2%) | -0.08 | 8,353 (6.4%) | 2,691 (8.0%) | -0.06 |
| | 1,718 (4.5%) | 466 (3.9%) | 0.03 | 3,033 (3.3%) | 548 (2.5%) | 0.05 | 4751 (3.6%) | 1014 (3.0%) | 0.03 |
| Delirium; n (%) | 579 (1.5%) | 134 (1.1%) | 0.04 | 1,192 (1.3%) | 168 (0.8%) | 0.05 | 1771 (1.4%) | 302 (0.9%) | 0.05 |
| Psychosis; n (%) | 472 (1.2%) | 95 (0.8%) | 0.04 | 853 (0.9%) | 124 (0.6%) | 0.03 | 1325 (1.0%) | 219 (0.6%) | 0.04 |
| Obesity; n (%) | 3,470 (9.1%) | 1,501 (12.6%) | -0.11 | 3,759 (4.0%) | 1,033 (4.7%) | -0.03 | 7,229 (5.5%) | 2,534 (7.5%) | -0.08 |
| Overweight; n (%) | 1,069 (2.8%) | 505 (4.2%) | -0.08 | 606 (0.7%) | 173 (0.8%) | -0.01 | 1,675 (1.3%) | 0,678 (2.0%) | -0.05 |
| Smoking; n (%) | 4,937 (13.0%) | 1,069 (8.9%) | 0.13 | 4,821 (5.2%) | 661 (3.0%) | 0.11 | 9,758 (7.5%) | 1,730 (5.1%) | 0.10 |
| Alcohol abuse or dependence; n (%) | 427 (1.1%) | 73 (0.6%) | 0.05 | 524 (0.6%) | 80 (0.4%) | 0.03 | 951 (0.7%) | 153 (0.5%) | 0.03 |
| Drug abuse or dependence; n (%) | 361 (1.0%) | 142 (1.2%) | -0.02 | 340 (0.4%) | 75 (0.3%) | 0.02 | 701 (0.5%) | 217 (0.6%) | -0.01 |
| COPD; n (%) | 4,437 (11.7%) | 1,308 (10.9%) | 0.03 | 8,552 (9.2%) | 1,752 (8.0%) | 0.04 | 12,989 (9.9%) | 3,060 (9.0%) | 0.03 |
| Asthma; n (%) | 1,741 (4.6%) | 784 (6.6%) | -0.09 | 3,318 (3.6%) | 1,135 (5.2%) | -0.08 | 5,059 (3.9%) | 1,919 (5.7%) | -0.08 |
| Obstructive sleep apnea; n (%) | 1,805 (4.8%) | 895 (7.5%) | -0.11 | 3,711 (4.0%) | 1,272 (5.8%) | -0.08 | 5,516 (4.2%) | 2,167 (6.4%) | -0.10 |
| Pneumonia; n (%) | 1,189 (3.1%) | 296 (2.5%) | 0.04 | 3,095 (3.3%) | 497 (2.3%) | 0.06 | 4,284 (3.3%) | 0,793 (2.3%) | 0.06 |
| Imaging, n (%) | 166 (0.4%) | 24 (0.2%) | 0.04 | 14,801 (15.9%) | 17 (0.1%) | 0.61 | 291 (0.2%) | 41 (0.1%) | 0.03 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 37,963 (100.0%) | 303 (2.5%) | 8.83 | 92,821 (100.0%) | 508 (2.3%) | 9.22 | 130,784 (100.0%) | 0,811 (2.4%) | 9.02 |
| Use of ARBs; n (%) | 325 (0.9%) | 11,955 (100.0%) | -14.84 | 833 (0.9%) | 21,871 (100.0%) | -14.84 | 1,158 (0.9%) | 33,826 (100.0%) | -14.84 |
| Use of Loop Diuretics - ; n (%) | 5,252 (13.8%) | 1,577 (13.2%) | 0.02 | 14,397 (15.5%) | 3,030 (13.9%) | 0.05 | 19,649 (15.0%) | 4,607 (13.6%) | 0.04 |
| Use of other diuretics-; n (%) | 1,157 (3.0%) | 294 (2.5%) | 0.03 | 2,865 (3.1%) | 556 (2.5%) | 0.04 | 4,022 (3.1%) | 0,850 (2.5%) | 0.04 |
| Use of nitrates-; n (%) | 5,526 (14.6%) | 846 (7.1%) | 0.24 | 16,635 (17.9%) | 1,960 (9.0%) | 0.26 | 22,161 (16.9%) | 2,806 (8.3%) | 0.26 |
| Use of other hypertension drugs; n (%) | 1,939 (5.1%) | 1,098 (9.2%) | -0.16 | 4,883 (5.3%) | 1,796 (8.2%) | -0.12 | 6,822 (5.2%) | 2,894 (8.6%) | -0.13 |
| Use of digoxin-; n (%) | 1,234 (3.3%) | 208 (1.7%) | 0.10 | 4,285 (4.6%) | 574 (2.6%) | 0.11 | 5519 (4.2%) | 782 (2.3%) | 0.11 |
| Use of Anti-arrhythmics; n (%) | 1,082 (2.9%) | 242 (2.0%) | 0.06 | 3,365 (3.6%) | 490 (2.2%) | 0.08 | 4447 (3.4%) | 732 (2.2%) | 0.07 |
| Use of COPD/asthma meds-; n (%) | 4,953 (13.0%) | 1,961 (16.4%) | -0.10 | 14,331 (15.4%) | 3,907 (17.9%) | -0.07 | 19,284 (14.7%) | 5,868 (17.3%) | -0.07 |
| Use of statins; n (%) | 24,481 (64.5%) | 6,411 (53.6%) | 0.22 | 61,328 (66.1%) | 11,663 (53.3%) | 0.26 | 85,809 (65.6%) | 18,074 (53.4%) | 0.25 |
| Use of other lipid-lowering drugs; n (%) | | 1,293 (10.8%) | 0.06 | 14,291 (15.4%) | 2,905 (13.3%) | 0.06 | | | |

Table 1: Telmisartan vs Ramipril

| Use of oral anticoagulants (Dabigatran, | 3,071 (8.1%) | 750 (6.3%) | 0.07 | 8,984 (9.7%) | 1,533 (7.0%) | 0.10 | 12,055 (9.2%) | 2,283 (6.7%) | 0.09 |
|---|---|---|---|---|---|---|---|---|---|
| Rivaroxaban, Apixaban, Warfarin); n (%) | | | | | | | | | |
| Use of heparin and other low-molecular | 251 (0.7%) | 60 (0.5%) | 0.03 | 45 (0.0%) | 4 (0.0%) | #DIV/0! | 296 (0.2%) | 64 (0.2%) | 0.00 |
| weight heparins; n (%) | | () | | | | | () | | |
| Use of NSAIDs; n (%) | 4,320 (11.4%) | 1,727 (14.4%) | -0.09 | 10,853 (11.7%) | 3,115 (14.2%) | -0.07 | 15,173 (11.6%) | 4,842 (14.3%) | -0.08 |
| Use of oral corticosteroids; n (%) | 5,292 (13.9%) | 2,068 (17.3%) | -0.09 | 14,014 (15.1%) | 3,758 (17.2%) | -0.06 | 19,306 (14.8%) | 5,826 (17.2%) | -0.07 |
| Use of bisphosphonate (); n (%) | 1,419 (3.7%) | 570 (4.8%) | -0.05 | 4,290 (4.6%) | 1,266 (5.8%) | -0.05 | 5709 (4.4%) | 1836 (5.4%) | -0.05 |
| Use of opioids-; n (%) | 9,421 (24.8%) | 3,054 (25.5%) | -0.02 | 24,882 (26.8%) | 6,229 (28.5%) | -0.04 | 34,303 (26.2%) | 9,283 (27.4%) | -0.03 |
| Use of antidepressants; n (%) | 7,526 (19.8%) | 2,613 (21.9%) | -0.05 | 19,409 (20.9%) | 4,795 (21.9%) | -0.02 | 26,935 (20.6%) | 7,408 (21.9%) | -0.03 |
| Use of antipsychotics; n (%) | 699 (1.8%) | 186 (1.6%) | 0.02 | 1,810 (1.9%) | 386 (1.8%) | 0.01 | 2,509 (1.9%) | 0,572 (1.7%) | 0.02 |
| Use of anticonvulsants; n (%) | 4,282 (11.3%) | 1,487 (12.4%) | -0.03 | 9,523 (10.3%) | 2,404 (11.0%) | -0.02 | 13,805 (10.6%) | 3,891 (11.5%) | -0.03 |
| Use of lithium-; n (%) | 74 (0.2%) | 9 (0.1%) | 0.03 | 159 (0.2%) | 30 (0.1%) | 0.03 | 233 (0.2%) | 39 (0.1%) | 0.03 |
| Use of Benzos- ; n (%) | 3,780 (10.0%) | 1,435 (12.0%) | -0.06 | 12,311 (13.3%) | 3,365 (15.4%) | -0.06 | 16,091 (12.3%) | 4,800 (14.2%) | -0.06 |
| Use of anxiolytics/hypnotics-; n (%) | 2,506 (6.6%) | 858 (7.2%) | -0.02 | 7,377 (7.9%) | 2,006 (9.2%) | -0.05 | 9,883 (7.6%) | 2,864 (8.5%) | -0.03 |
| Use of dementia meds-; n (%) | 1,026 (2.7%) | 322 (2.7%) | 0.00 | 2,537 (2.7%) | 592 (2.7%) | 0.00 | 3563 (2.7%) | 914 (2.7%) | 0.00 |
| Use of antiparkinsonian meds-; n (%) | 769 (2.0%) | 254 (2.1%) | -0.01 | 2,048 (2.2%) | 575 (2.6%) | -0.03 | 2,817 (2.2%) | 0,829 (2.5%) | -0.02 |
| Entresto (sacubitril/valsartan); n (%) | 22 (0.1%) | 3 (0.0%) | 0.04 | 17 (0.0%) | 1 (0.0%) | #DIV/0! | 39 (0.0%) | 4 (0.0%) | #DIV/0! |
| Labs | | | | | | | 0 | 0 | |
| Lab values- HbA1c (%); n (%) | 6,272 (16.5%) | 2,302 (19.3%) | -0.07 | 1,279 (1.4%) | 286 (1.3%) | 0.01 | 7,551 (5.8%) | 2,588 (7.7%) | -0.08 |
| Lab values-HbA1c (%) (within 3 months) ; n<br>(%) | 4,439 (11.7%) | 1,572 (13.1%) | -0.04 | 917 (1.0%) | 198 (0.9%) | 0.01 | 5,356 (4.1%) | 1,770 (5.2%) | -0.05 |
| Lab values-HbA1c (%) (within 6 months); n | 6,272 (16.5%) | 2,302 (19.3%) | -0.07 | 1,279 (1.4%) | 286 (1.3%) | 0.01 | 7,551 (5.8%) | 2,588 (7.7%) | -0.08 |
| (%) | | | | | | | | | |
| Lab values-BNP; n (%) | 242 (0.6%) | 82 (0.7%) | -0.01 | 30 (0.0%) | 6 (0.0%) | #DIV/0! | 272 (0.2%) | 88 (0.3%) | -0.02 |
| Lab values-BNP (within 3 months); n (%) | 173 (0.5%) | 55 (0.5%) | 0.00 | 21 (0.0%) | 3 (0.0%) | #DIV/0! | 194 (0.1%) | 58 (0.2%) | -0.03 |
| Lab values-BNP (within 6 months); n (%) | 242 (0.6%) | 82 (0.7%) | -0.01 | 30 (0.0%) | 6 (0.0%) | #DIV/0! | 272 (0.2%) | 88 (0.3%) | -0.02 |
| Lab values-BUN (mg/dl); n (%) | 9,218 (24.3%) | 3,511 (29.4%) | -0.12 | 1,435 (1.5%) | 341 (1.6%) | -0.01 | 10,653 (8.1%) | 3,852 (11.4%) | -0.11 |
| Lab values-BUN (mg/dl) (within 3 months); | 6,592 (17.4%) | 2,507 (21.0%) | -0.09 | 1,028 (1.1%) | 238 (1.1%) | 0.00 | 7,620 (5.8%) | 2,745 (8.1%) | -0.09 |
| n (%) | | | | | | | | | |
| Lab values-BUN (mg/dl) (within 6 months); | 9,218 (24.3%) | 3,511 (29.4%) | -0.12 | 1,435 (1.5%) | 341 (1.6%) | -0.01 | 10,653 (8.1%) | 3,852 (11.4%) | -0.11 |
| n (%) | | | | | | | | | |
| Lab values- Creatinine (mg/dl); n (%) | 9,536 (25.1%) | 3,630 (30.4%) | -0.12 | 1,550 (1.7%) | 372 (1.7%) | 0.00 | 11,086 (8.5%) | 4,002 (11.8%) | -0.11 |
| Lab values- Creatinine (mg/dl) (within 3 | 6,818 (18.0%) | 2,584 (21.6%) | -0.09 | 1,127 (1.2%) | 260 (1.2%) | 0.00 | 7,945 (6.1%) | 2,844 (8.4%) | -0.09 |
| months); n (%) | | | | | | | | | |
| Lab values-Creatinine (mg/dl) (within 6 | 9,536 (25.1%) | 3,630 (30.4%) | -0.12 | 1,550 (1.7%) | 372 (1.7%) | 0.00 | 11,086 (8.5%) | 4,002 (11.8%) | -0.11 |
| months); n (%) | | | | | | | | | |
| Lab values- HDL level (mg/dl); n (%) | 7,182 (18.9%) | 2,656 (22.2%) | -0.08 | 1,289 (1.4%) | 290 (1.3%) | 0.01 | 8,471 (6.5%) | 2,946 (8.7%) | -0.08 |
| Lab values- HDL level (mg/dl) (within 3<br>months); n (%) | 4,912 (12.9%) | 1,760 (14.7%) | -0.05 | 893 (1.0%) | 184 (0.8%) | 0.02 | 5,805 (4.4%) | 1,944 (5.7%) | -0.06 |
| Lab values- HDL level (mg/dl) (within 6<br>months); n (%) | 7,182 (18.9%) | 2,656 (22.2%) | -0.08 | 1,289 (1.4%) | 290 (1.3%) | 0.01 | 8,471 (6.5%) | 2,946 (8.7%) | -0.08 |
| Lab values-LDL level (mg/dl); n (%) | 8,000 (21.1%) | 2,859 (23.9%) | -0.07 | 1,313 (1.4%) | 299 (1.4%) | 0.00 | 9,313 (7.1%) | 3,158 (9.3%) | -0.08 |
| Lab values-LDL level (mg/dl) (within 3<br>months) ; n (%) | 5,499 (14.5%) | 1,895 (15.9%) | -0.04 | 910 (1.0%) | 190 (0.9%) | 0.01 | 6,409 (4.9%) | 2,085 (6.2%) | -0.06 |
| Lab values-LDL level (mg/dl) (within 6<br>months) ; n (%) | 8,000 (21.1%) | 2,859 (23.9%) | -0.07 | 1,313 (1.4%) | 299 (1.4%) | 0.00 | 9,313 (7.1%) | 3,158 (9.3%) | -0.08 |
| Lab values- NT-proBNP; n (%) | 38 (0.1%) | 22 (0.2%) | -0.03 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 41 (0.0%) | 22 (0.1%) | -0.04 |
| Lab values- NT-proBNP (within 3 months); | 24 (0.1%) | 12 (0.1%) | 0.00 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 27 (0.0%) | 12 (0.0%) | #DIV/0! |
| n (%) | | | | | | | , , | . , | |

# Table 1: Telmisartan vs Ramipril

| Lab values-NT-proBNP (within 6 months);<br>n (%) | 38 (0.1%) | 22 (0.2%) | -0.03 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | 41 (0.0%) | 22 (0.1%) | -0.04 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values-Total cholesterol (mg/dl); n (%) | 8,031 (21.2%) | 2,864 (24.0%) | -0.07 | 1,323 (1.4%) | 299 (1.4%) | 0.00 | 9,354 (7.2%) | 3,163 (9.4%) | -0.08 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 5,524 (14.6%) | 1,899 (15.9%) | -0.04 | 919 (1.0%) | 188 (0.9%) | 0.01 | 6,443 (4.9%) | 2,087 (6.2%) | -0.06 |
| Lab values-Total cholesterol (mg/dl)<br>(within 6 months); n (%) | 8,031 (21.2%) | 2,864 (24.0%) | -0.07 | 1,323 (1.4%) | 299 (1.4%) | 0.00 | 9,354 (7.2%) | 3,163 (9.4%) | -0.08 |
| Lab values-Triglyceride level (mg/dl); n (%) | 7,813 (20.6%) | 2,828 (23.7%) | -0.07 | 1,314 (1.4%) | 293 (1.3%) | 0.01 | 9,127 (7.0%) | 3,121 (9.2%) | -0.08 |
| Lab values-Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 5,376 (14.2%) | 1,878 (15.7%) | -0.04 | 912 (1.0%) | 186 (0.9%) | 0.01 | 6,288 (4.8%) | 2,064 (6.1%) | -0.06 |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 7,813 (20.6%) | 2,828 (23.7%) | -0.07 | 1,314 (1.4%) | 293 (1.3%) | 0.01 | 9,127 (7.0%) | 3,121 (9.2%) | -0.08 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 5,992 | 2,235 | | 1,237 | 276 | | 0 | 0 | |
| mean (sd) | 7.19 (1.66) | 6.93 (1.58) | 0.16 | 7.59 (1.79) | 7.24 (1.63) | 0.20 | 7.47 (1.75) | 7.13 (1.61) | 0.20 |
| median [IQR] | 6.70 [6.00, 7.85] | 6.50 [5.90, 7.55] | 0.12 | 7.10 [6.30, 8.30] | 6.75 [6.10, 8.00] | 0.20 | 6.98 (1.75) | 6.66 (1.61) | 0.19 |
| Missing; n (%) | 31,971 (84.2%) | 9,720 (81.3%) | 0.08 | 91,584 (98.7%) | 21,595 (98.7%) | 0.00 | 123,555 (94.5%) | 31,315 (92.6%) | 0.08 |
| Lab result number- BNP mean | 242 | 82 | | 30 | 6 | | 0 | 0 | - 1 |
| mean (sd) | 231.84 (419.63) | 184.35 (414.42) | 0.11 | 8,444.38 (45,622.79) | 40.33 (28.20) | 0.26 | 6060.51 (38435.82) | 91.23 (247.41) | 0.22 |
| median [IQR] | 105.35 [39.08,<br>225.15] | 69.65 [30.48, 152.00] | 0.09 | 74.10 [23.00,<br>177.00] | 42.00 [18.00, 66.00] | 0.00 | 83.17 (38435.82) | 51.77 (247.41) | 0.00 |
| Missing; n (%) | 37,721 (99.4%) | 11,873 (99.3%) | 0.01 | 92,791 (100.0%) | 21,865 (100.0%) | #DIV/0! | 130,512 (99.8%) | 33,738 (99.7%) | 0.02 |
| Lab result number- BUN (mg/dl) mean | 9,218 | 3,511 | | 1,435 | 341 | | 0 | 0 | - 1 |
| mean (sd) | -18.62 (3,471.95) | -503.49 (19,685.58) | 0.03 | 1,284.61 (16,530.91) | 634.14 (8,037.23) | 0.05 | 906.32 (14051.61) | 232.07 (13368.79) | 0.05 |
| median [IQR] | 17.00 [13.00, 21.00] | 17.00 [13.50, 22.00] | 0.00 | 16.67 [13.00, 21.00] | 16.50 [14.00, 21.62] | 0.00 | 16.77 (14051.61) | 16.68 (13368.79) | 0.00 |
| Missing; n (%) | 28,745 (75.7%) | 8,444 (70.6%) | 0.12 | 91,386 (98.5%) | 21,530 (98.4%) | 0.01 | 120,131 (91.9%) | 29,974 (88.6%) | 0.11 |
| Lab result number- Creatinine (mg/dl) | 8,971 | 3,488 | | 1,514 | 364 | | 0 | 0 | - 1 |
| mean (only 0.1 to 15 included) | | | | | | | | | - 1 |
| mean (sd) | 1.04 (0.43) | 1.08 (0.55) | -0.08 | 1.00 (0.39) | 1.04 (0.46) | -0.09 | 1.01 (0.40) | 1.05 (0.49) | -0.09 |
| median [IQR] | 0.97 [0.82, 1.16] | 0.97 [0.80, 1.20] | 0.00 | 0.94 [0.79, 1.10] | 0.94 [0.78, 1.15] | 0.00 | 0.95 (0.40) | 0.95 (0.49) | 0.00 |
| Missing; n (%) | 28,992 (76.4%) | 8,467 (70.8%) | 0.13 | 91,307 (98.4%) | 21,507 (98.3%) | 0.01 | 120,299 (92.0%) | 29,974 (88.6%) | 0.12 |
| Lab result number- HDL level (mg/dl) mean | 7,182 | 2,656 | | 1,283 | 289 | | 0 | 0 | ı |
| (only =<5000 included) | | | | | | | | | - 1 |
| mean (sd) | 47.33 (17.84) | 50.53 (17.48) | -0.18 | 46.98 (15.84) | 48.11 (17.13) | -0.07 | 47.08 (16.45) | 48.97 (17.25) | -0.11 |
| median [IQR] | 46.00 [38.00, 57.00] | 49.00 [40.00, 59.62] | -0.17 | 45.00 [37.50, 54.67] | 46.00 [37.00, 57.00] | -0.06 | 45.29 (16.45) | 47.06 (17.25) | -0.11 |
| Missing; n (%) | 30,781 (81.1%) | 9,299 (77.8%) | 0.08 | 91,538 (98.6%) | 21,582 (98.7%) | -0.01 | 122,319 (93.5%) | 30,881 (91.3%) | 0.08 |
| Lab result number-LDL level (mg/dl) mean (only =<5000 included) | 7,845 | 2,824 | | 1,270 | 293 | | 0 | 0 | |
| mean (sd) | -3,429.61 (57,169.13) | -1,780.42 (40,246.04) | -0.03 | 90.45 (42.42) | 94.53 (47.17) | -0.09 | -931.33 (30800.83) | -568.13 (23925.88) | -0.01 |
| median [IQR] | 85.00 [61.50, 112.00] | 90.00 [67.00, 116.00] | 0.00 | 88.00 [65.00,<br>113.00] | 89.00 [65.00,<br>121.00] | -0.02 | 87.13 (30800.83) | 89.35 (23925.88) | 0.00 |
| Missing; n (%) | 30,118 (79.3%) | 9,131 (76.4%) | 0.07 | 91,551 (98.6%) | 21,578 (98.7%) | -0.01 | 121,669 (93.0%) | 30,709 (90.8%) | 0.08 |

# Table 1: Telmisartan vs Ramipril

| Lab result number-Total cholesterol | 8,026 | 2,862 | | 1,317 | 297 | | 0 | 0 | - 1 |
|---|---|---|---|---|---|---|---|---|---|
| (mg/dl) mean (only =<5000 included) | | | | | | | | | - 1 |
| mean (sd) | 163.98 (62.21) | 170.82 (54.20) | -0.12 | 172.04 (54.21) | 182.87 (58.76) | -0.19 | 169.70 (56.65) | 178.61 (57.19) | -0.16 |
| median [IQR] | 165.00 [137.00,<br>198.00] | 171.00 [143.38,<br>201.00] | -0.10 | 168.00 [141.17,<br>199.75] | 177.75 [151.00,<br>206.25] | -0.17 | 167.13 (56.65) | 175.36 (57.19) | -0.14 |
| Missing; n (%) | 29,937 (78.9%) | 9,093 (76.1%) | 0.07 | 91,504 (98.6%) | 21,574 (98.6%) | 0.00 | 121,441 (92.9%) | 30,667 (90.7%) | 0.08 |
| Lab result number-Triglyceride level | 7,812 | 2,828 | | 1,308 | 292 | | 0 | 0 | - 1 |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | - 1 |
| mean (sd) | 145.34 (119.44) | 141.55 (95.58) | 0.04 | 162.46 (135.71) | 192.41 (285.64) | -0.13 | 157.49 (131.20) | 174.43 (236.61) | -0.09 |
| median [IQR] | 122.00 [84.00,<br>177.00] | 121.00 [87.00,<br>172.00] | 0.01 | 136.00 [92.00,<br>190.50] | 145.00 [102.00,<br>211.75] | -0.04 | 131.94 (131.20) | 136.52 (236.61) | -0.02 |
| Missing; n (%) | 30,151 (79.4%) | 9,127 (76.3%) | 0.07 | 91,513 (98.6%) | 21,579 (98.7%) | -0.01 | 121,664 (93.0%) | 30,706 (90.8%) | 0.08 |
| Lab result number- Hemoglobin mean<br>(only >0 included) | 6,569 | 2,671 | | 990 | 254 | | 0 | 0 | |
| mean (sd) | -1,026.52 (29,854.92) | 13.30 (1.68) | -0.05 | 11,174.87<br>(318,011.67) | 1,071.92 (11,916.90) | 0.04 | 7633.14<br>(268392.99) | 697.78 (9582.42) | 0.04 |
| median [IQR] | 13.80 [12.70, 14.90] | 13.30 [12.20, 14.40] | 0.00 | 13.90 [12.70, 14.90] | 13.40 [12.30, 14.22] | 0.00 | 13.87 (268392.99) | 13.36 (9582.42) | 0.00 |
| Missing; n (%) | 31,394 (82.7%) | 9,284 (77.7%) | 0.13 | 91,831 (98.9%) | 21,617 (98.8%) | 0.01 | 123,225 (94.2%) | 30,901 (91.4%) | 0.11 |
| Lab result number- Serum sodium mean<br>(only > 90 and < 190 included) | 8,774 | 3,449 | | 1,297 | 309 | | 0 | 0 | |
| mean (sd) | 140.07 (2.63) | 140.28 (2.88) | -0.08 | 139.68 (2.44) | 139.60 (2.37) | 0.03 | 139.79 (2.50) | 139.84 (2.56) | -0.02 |
| median [IQR] | 140.00 [139.00,<br>142.00] | 140.50 [139.00,<br>142.00] | -0.18 | 140.00 [138.00,<br>141.00] | 140.00 [138.00,<br>141.00] | 0.00 | 140.00 (2.50) | 140.18 (2.56) | -0.07 |
| Missing; n (%) | 29,189 (76.9%) | 8,506 (71.2%) | 0.13 | 91,524 (98.6%) | 21,562 (98.6%) | 0.00 | 120,713 (92.3%) | 30,068 (88.9%) | 0.12 |
| Lab result number- Albumin mean (only >0 and <=10 included) | 8,299 | 3,240 | | 1,218 | 293 | | 0 | 0 | |
| mean (sd) | 4.22 (0.34) | 4.21 (0.35) | 0.03 | 4.18 (0.66) | 4.12 (0.69) | 0.09 | 4.19 (0.59) | 4.15 (0.59) | 0.07 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.25 [4.06, 4.50] | 4.20 [4.00, 4.40] | 0.07 | 4.24 (0.59) | 4.20 (0.59) | 0.07 |
| Missing; n (%) | 29,664 (78.1%) | 8,715 (72.9%) | 0.12 | 91,603 (98.7%) | 21,578 (98.7%) | 0.00 | 121,267 (92.7%) | 30,293 (89.6%) | 0.11 |
| Lab result number- Glucose (fasting or | 8,610 | 3,424 | | 1,294 | 309 | | 0 | 0 | |
| random) mean (only 10-1000 included) | | | | | | | | | - 1 |
| mean (sd) | 128.64 (56.57) | 121.53 (51.47) | 0.13 | 143.08 (62.07) | 137.82 (59.51) | 0.09 | 138.89 (60.53) | 132.06 (56.80) | 0.12 |
| median [IQR] | 109.00 [94.00, | 105.00 [92.54, | 0.07 | 125.00 [102.00, | 120.00 [100.00, | 0.08 | 120.36 (60.53) | 114.70 (56.80) | 0.10 |
| Missing; n (%) | 143.00]<br>29,353 (77.3%) | 133.00]<br>8,531 (71.4%) | 0.14 | 164.25]<br>91,527 (98.6%) | 157.50]<br>21,562 (98.6%) | 0.00 | 120,880 (92.4%) | 30,093 (89.0%) | 0.12 |
| iviissing, n (%)<br>Lab result number- Potassium mean (only | 29,353 (77.3%)<br>8.888 | 8,531 (/1.4%)<br>3.490 | 0.14 | 1,383 | 21,562 (98.6%) | 0.00 | 120,880 (92.4%) | 30,093 (89.0%) | 0.12 |
| 1-7 included) | 0,000 | 3,430 | | 1,303 | 334 | | U | J | |
| mean (sd) | 4.44 (0.42) | 4.39 (0.44) | 0.12 | 4.41 (0.41) | 4.33 (0.43) | 0.19 | 4.42 (0.41) | 4.35 (0.43) | 0.17 |
| median [IQR] | 4.40 [4.20, 4.70] | 4.40 [4.10, 4.70] | 0.00 | 4.40 [4.18, 4.70] | 4.30 [4.10, 4.60] | 0.24 | 4.40 (0.41) | 4.34 (0.43) | 0.14 |
| Missing, n (%) | 29,075 (76.6%) | 8,465 (70.8%) | 0.13 | 91,438 (98.5%) | 21,537 (98.5%) | 0.00 | 120,513 (92.1%) | 30,002 (88.7%) | 0.12 |
| Comorbidity Scores | | _, , , | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.43 (1.94) | 2.49 (1.89) | -0.03 | 1.71 (1.64) | 1.71 (1.52) | 0.00 | 1.92 (1.73) | 1.99 (1.66) | -0.04 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 1.29 (1.73) | 1.35 (1.66) | -0.04 |
| Frailty Score (mean): Empirical Version 365 | | | | | | | | | |
| days, | | | | | | | | | |
| mean (sd) | 0.18 (0.06) | 0.17 (0.06) | 0.17 | 0.16 (0.05) | 0.16 (0.05) | 0.00 | 0.17 (0.05) | 0.16 (0.05) | 0.20 |
| median [IQR] | 0.16 [0.14, 0.20] | 0.16 [0.14, 0.20] | 0.00 | 0.15 [0.13, 0.18] | 0.15 [0.13, 0.18] | 0.00 | 0.15 (0.05) | 0.15 (0.05) | 0.00 |

Table 1: Telmisartan vs Ramipril

| Healthcare Utilization | 1 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization; n (%) | 8,075 (21.3%) | 1,130 (9.5%) | 0.33 | 24,371 (26.3%) | 2,561 (11.7%) | 0.38 | 32,446 (24.8%) | 3,691 (10.9%) | 0.37 |
| Any hospitalization during prior 31-180 | 3,508 (9.2%) | 900 (7.5%) | 0.06 | 11,208 (12.1%) | 1,988 (9.1%) | 0.10 | 14,716 (11.3%) | 2,888 (8.5%) | 0.09 |
| days; n (%) | 3,300 (3.2%) | 500 (7.5%) | 0.00 | 11,200 (12.1%) | 1,500 (5.1%) | 0.10 | 14,710 (11.570) | 2,000 (0.5%) | 0.03 |
| Endocrinologist Visit; n (%) | 3,025 (8.0%) | 835 (7.0%) | 0.04 | 6,470 (7.0%) | 1,263 (5.8%) | 0.05 | 9,495 (7.3%) | 2,098 (6.2%) | 0.04 |
| Endocrinologist Visit (30 days prior); n (%) | 1,441 (3.8%) | 300 (2.5%) | 0.07 | 3,063 (3.3%) | 475 (2.2%) | 0.07 | 4,504 (3.4%) | 0,775 (2.3%) | 0.07 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 2,445 (6.4%) | 722 (6.0%) | 0.02 | 5,250 (5.7%) | 1,105 (5.1%) | 0.03 | 7,695 (5.9%) | 1,827 (5.4%) | 0.02 |
| Internal medicine/family medicine visits; n<br>(%) | 28,199 (74.3%) | 9,198 (76.9%) | -0.06 | 68,739 (74.1%) | 17,095 (78.2%) | -0.10 | 96,938 (74.1%) | 26,293 (77.7%) | -0.08 |
| Internal medicine/family medicine visits<br>(30 days prior); n (%) | 18,818 (49.6%) | 5,859 (49.0%) | 0.01 | 43,764 (47.1%) | 10,543 (48.2%) | -0.02 | 62,582 (47.9%) | 16,402 (48.5%) | -0.01 |
| Internal medicine/family medicine visits<br>(31 to 180 days prior); n (%) | 23,757 (62.6%) | 8,113 (67.9%) | -0.11 | 59,359 (63.9%) | 15,346 (70.2%) | -0.13 | 83,116 (63.6%) | 23,459 (69.4%) | -0.12 |
| Cardiologist visit; n (%) | 19,758 (52.0%) | 4,641 (38.8%) | 0.27 | 38,839 (41.8%) | 7,118 (32.5%) | 0.19 | 58,597 (44.8%) | 11,759 (34.8%) | 0.21 |
| Number of Cardiologist visits (30 days | 12,595 (33.2%) | 1,986 (16.6%) | 0.39 | 23,165 (25.0%) | 3,090 (14.1%) | 0.28 | 35,760 (27.3%) | 5,076 (15.0%) | 0.30 |
| prior); n (%) | 12,333 (33.270) | 1,500 (10.070) | 0.33 | 23,203 (23.070) | 3,030 (14.170) | 0.20 | 33,100 (21.370) | 3,070 (13.070) | 0.30 |
| Number of Cardiologist visits (31 to 180 | 12,948 (34.1%) | 3,810 (31.9%) | 0.05 | 27,848 (30.0%) | 5,830 (26.7%) | 0.07 | 40,796 (31.2%) | 9,640 (28.5%) | 0.06 |
| days prior); n (%) | , (, | -, (, | | | -,, | | ,, | -,, | |
| Electrocardiogram ; n (%) | 18,432 (48.6%) | 4,720 (39.5%) | 0.18 | 44,610 (48.1%) | 8,382 (38.3%) | 0.20 | 63,042 (48.2%) | 13,102 (38.7%) | 0.19 |
| Use of glucose test strips; n (%) | 983 (2.6%) | 304 (2.5%) | 0.01 | 1,782 (1.9%) | 359 (1.6%) | 0.02 | 2,765 (2.1%) | 0,663 (2.0%) | 0.01 |
| Dialysis; n (%) | 97 (0.3%) | 38 (0.3%) | 0.00 | 270 (0.3%) | 46 (0.2%) | 0.02 | 367 (0.3%) | 84 (0.2%) | 0.02 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 8.27 (4.55) | 8.49 (4.96) | -0.05 | 8.96 (4.84) | 8.80 (5.02) | 0.03 | 8.76 (4.76) | 8.69 (5.00) | 0.01 |
| median [IQR] | 7.00 [5.00, 11.00] | 8.00 [5.00, 11.00] | -0.21 | 8.00 [5.00, 12.00] | 8.00 [5.00, 11.00] | 0.00 | 7.71 (4.76) | 8.00 (5.00) | -0.06 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.25 (0.54) | 0.11 (0.38) | 0.30 | 0.30 (0.55) | 0.13 (0.39) | 0.36 | 0.29 (0.55) | 0.12 (0.39) | 0.36 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.55) | 0.00 (0.39) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 1.43 (4.41) | 0.63 (3.03) | 0.21 | 1.68 (4.87) | 0.69 (3.02) | 0.24 | 1.61 (4.74) | 0.67 (3.02) | 0.24 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (4.74) | 0.00 (3.02) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.49 (1.17) | 0.45 (1.17) | 0.03 | 0.38 (2.09) | 0.12 (0.99) | 0.16 | 0.41 (1.87) | 0.24 (1.06) | 0.11 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.87) | 0.00 (1.06) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 4.96 (4.38) | 5.57 (4.52) | -0.14 | 5.13 (4.53) | 5.68 (4.71) | -0.12 | 5.08 (4.49) | 5.64 (4.64) | -0.12 |
| median [IQR] | 4.00 [2.00, 7.00] | 5.00 [2.00, 8.00] | -0.22 | 4.00 [2.00, 7.00] | 5.00 [2.00, 8.00] | -0.22 | 4.00 (4.49) | 5.00 (4.64) | -0.22 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.40 (2.14) | 0.33 (1.90) | 0.03 | 0.35 (2.02) | 0.27 (1.73) | 0.04 | 0.39 (1.81) | 0.33 (1.56) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.81) | 0.00 (1.56) | 0.00 |
| Number of internal medicine/family<br>medicine visits | | | | | | | | | |
| mean (sd) | 7.74 (13.04) | 8.18 (12.63) | -0.03 | 6.03 (10.20) | 6.47 (9.97) | -0.04 | 6.53 (11.10) | 7.07 (10.98) | -0.05 |
| median [IQR] | 4.00 [0.00, 9.00] | 4.00 [1.00, 10.00] | 0.00 | 3.00 [0.00, 8.00] | 4.00 [1.00, 8.00] | -0.10 | 3.29 (11.10) | 4.00 (10.98) | -0.06 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 4.20 (7.38) | 2.14 (4.66) | 0.33 | 2.55 (5.30) | 1.74 (4.19) | 0.17 | 3.03 (5.98) | 1.88 (4.36) | 0.22 |

Table 1: Telmisartan vs Ramipril

| median [IQR] | 1.00 [0.00, 6.00] | 0.00 [0.00, 2.00] | 0.16 | 0.00 [0.00, 3.00] | 0.00 [0.00, 2.00] | 0.00 | 0.29 (5.98) | 0.00 (4.36) | 0.06 |
|---|---|---|---|---|---|---|---|---|---|
| Number electrocardiograms received | 1.00 [0.00, 6.00] | 0.00 [0.00, 2.00] | 0.16 | 0.00 [0.00, 5.00] | 0.00 [0.00, 2.00] | 0.00 | 0.23 (5.36) | 0.00 (4.36) | 0.06 |
| mean (sd) | 1.24 (2.26) | 0.79 (1.46) | 0.24 | 0.93 (1.50) | 0.66 (1.17) | 0.20 | 1.02 (1.75) | 0.71 (1.28) | 0.20 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.75) | 0.00 (1.28) | 0.00 |
| Number of HbA1c tests ordered | 5.55 [5.55, 2.55] | | | | [,] | | | () | |
| mean (sd) | 0.59 (0.86) | 0.63 (0.85) | -0.05 | 0.33 (0.69) | 0.31 (0.66) | 0.03 | 0.41 (0.74) | 0.42 (0.73) | -0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.74) | 0.00 (0.73) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.32 (2.23) | 0.30 (1.23) | 0.01 | 0.19 (1.31) | 0.18 (0.73) | 0.01 | 0.23 (1.63) | 0.22 (0.94) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.63) | 0.00 (0.94) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.83 (1.02) | 0.82 (0.96) | 0.01 | 0.49 (0.98) | 0.46 (0.91) | 0.03 | 0.59 (0.99) | 0.59 (0.93) | 0.00 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.29 (0.99) | 0.35 (0.93) | -0.06 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.07 (0.41) | 0.08 (0.45) | -0.02 | 0.05 (0.32) | 0.06 (0.34) | -0.03 | 0.06 (0.35) | 0.07 (0.38) | -0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.35) | 0.00 (0.38) | 0.00 |
| Number of BUN tests ordered | 0.05 (0.44) | 0.05 (0.54) | 0.00 | 0.04/0.70\ | 0.04/0.75\ | 0.00 | 0.04 (0.35) | 0.05 (0.40) | 0.00 |
| mean (sd)<br>median [IQR] | 0.05 (0.41)<br>0.00 [0.00, 0.00] | 0.06 (0.51)<br>0.00 [0.00, 0.00] | -0.02<br>0.00 | 0.04 (0.32)<br>0.00 [0.00, 0.00] | 0.04 (0.36)<br>0.00 [0.00, 0.00] | 0.00 | 0.04 (0.35)<br>0.00 (0.35) | 0.05 (0.42)<br>0.00 (0.42) | -0.03<br>0.00 |
| Number of tests for microal burninuria | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.55) | 0.00 (0.42) | 0.00 |
| mean (sd) | 0.37 (0.91) | 0.40 (0.94) | -0.03 | 0.19 (0.64) | 0.17 (0.61) | 0.03 | 0.24 (0.73) | 0.25 (0.74) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.73) | 0.00 (0.74) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at | | | | | | | | | |
| the 3rd digit level | | | | | | | | | |
| mean (sd) | 4.10 (6.83) | 5.20 (7.87) | -0.15 | 1.74 (4.15) | 1.33 (3.39) | 0.11 | 2.43 (5.08) | 2.70 (5.41) | -0.05 |
| median [IQR] | 0.00 [0.00, 6.00] | 2.00 [0.00, 8.00] | -0.27 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (5.08) | 0.71 (5.41) | -0.14 |
| For PS | | | | | | | | | |
| Hemorrhagic stroke+Other | 1,573 (4.1%) | 420 (3.5%) | 0.03 | 2,937 (3.2%) | 576 (2.6%) | 0.04 | 4510 (3.4%) | 996 (2.9%) | 0.03 |
| cerebrovascular disease+Cerebrovascular<br>procedure (for PS); n (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for PS); n (%) | 2,017 (5.3%) | 671 (5.6%) | -0.01 | 3,713 (4.0%) | 866 (4.0%) | 0.00 | 5,730 (4.4%) | 1,537 (4.5%) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n<br>(%) | 1,339 (3.5%) | 433 (3.6%) | -0.01 | 2,756 (3.0%) | 607 (2.8%) | 0.01 | 4,095 (3.1%) | 1,040 (3.1%) | 0.00 |
| Occurrence of chronic renal insufficiency<br>w/o CKD (for PS); n (%) | 1,645 (4.3%) | 672 (5.6%) | -0.06 | 1,963 (2.1%) | 584 (2.7%) | -0.04 | 3,608 (2.8%) | 1,256 (3.7%) | -0.05 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 779 (2.1%) | 344 (2.9%) | -0.05 | 669 (0.7%) | 241 (1.1%) | -0.04 | 1448 (1.1%) | 585 (1.7%) | -0.05 |
| Chronic kidney disease Stage 3-6 (for PS); n<br>(%) | 2,242 (5.9%) | 1,272 (10.6%) | -0.17 | 2,667 (2.9%) | 1,012 (4.6%) | -0.09 | 4,909 (3.8%) | 2,284 (6.8%) | -0.13 |
| Bladder stones+Kidney stones (for PS); n<br>(%) | 758 (2.0%) | 257 (2.1%) | -0.01 | 1,741 (1.9%) | 369 (1.7%) | 0.02 | 2,499 (1.9%) | 0,626 (1.9%) | 0.00 |
| Diabetes with peripheral circulatory<br>disorders+Gangrene+Osteomyelitis(for PS)<br>with ICD10; n (%) | 1,851 (4.9%) | 532 (4.5%) | 0.02 | 2,580 (2.8%) | 460 (2.1%) | 0.05 | 4,431 (3.4%) | 0,992 (2.9%) | 0.03 |
| Alcohol abuse or dependence+Drug abuse or dependence (for PS); n (%) | 750 (2.0%) | 210 (1.8%) | 0.01 | 820 (0.9%) | 149 (0.7%) | 0.02 | 1570 (1.2%) | 359 (1.1%) | 0.01 |

Table 1: Telmisartan vs Ramipril

| Diabetes with other ophthalmic<br>manifestations+Retinal detachment,<br>vitreous hemorrhage, vitrectomy+Retinal<br>laser coagulation therapy (for PS); n (%) | 584 (1.5%) | 197 (1.6%) | -0.01 | 3,380 (3.6%) | 755 (3.5%) | 0.01 | 3,964 (3.0%) | 0,952 (2.8%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS); n (%) | 9,446 (24.9%) | 2,138 (17.9%) | 0.17 | 19,987 (21.5%) | 3,130 (14.3%) | 0.19 | 29,433 (22.5%) | 5,268 (15.6%) | 0.18 |
| Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA (for PS) ; n (%) | 7,667 (20.2%) | 847 (7.1%) | 0.39 | 11,938 (12.9%) | 721 (3.3%) | 0.36 | 19,605 (15.0%) | 1,568 (4.6%) | 0.36 |
| Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 5,896 (15.5%) | 2,314 (19.4%) | -0.10 | 8,543 (9.2%) | 2,435 (11.1%) | -0.06 | 14,439 (11.0%) | 4,749 (14.0%) | -0.09 |
| Delirium + Psychosis (for PS); n (%) | 945 (2.5%) | 209 (1.7%) | 0.06 | 1,834 (2.0%) | 273 (1.2%) | 0.06 | 2779 (2.1%) | 482 (1.4%) | 0.05 |
| Any use of Meglitinides (for PS); n (%) | 315 (0.8%) | 72 (0.6%) | 0.02 | 1,137 (1.2%) | 239 (1.1%) | 0.01 | 1452 (1.1%) | 311 (0.9%) | 0.02 |
| Any use of AGIs (for PS); n (%) | 64 (0.2%) | 17 (0.1%) | 0.03 | 216 (0.2%) | 41 (0.2%) | 0.00 | 29,433 (22.5%) | 5,268 (15.6%) | 0.18 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 2,258 (5.9%) | 1,280 (10.7%) | -0.17 | 2,756 (3.0%) | 1,015 (4.6%) | -0.08 | 5,014 (3.8%) | 2,295 (6.8%) | -0.13 |
| Use of thiazide; n (%) | 3,399 (9.0%) | 1,398 (11.7%) | -0.09 | 8,655 (9.3%) | 2,289 (10.5%) | -0.04 | 69,385 (53.1%) | 13,491 (39.9%) | 0.27 |
| Use of beta blockers; n (%) | 19,309 (50.9%) | 4,780 (40.0%) | 0.22 | 50,076 (53.9%) | 8,711 (39.8%) | 0.29 | 25,567 (19.5%) | 10,073 (29.8%) | -0.24 |
| Use of calcium channel blockers; n (%) | 7,144 (18.8%) | 3,694 (30.9%) | -0.28 | 18,423 (19.8%) | 6,379 (29.2%) | -0.22 | 43,200 (33.0%) | 10,354 (30.6%) | 0.05 |
| All antidiabetic medications except<br>Insulin; n (%) | 12,807 (33.7%) | 3,883 (32.5%) | 0.03 | 30,393 (32.7%) | 6,471 (29.6%) | 0.07 | 12,054 (9.2%) | 3,687 (10.9%) | -0.06 |
| DM Medications - Insulin ; n (%) | 4,891 (12.9%) | 1,386 (11.6%) | 0.04 | 11,894 (12.8%) | 2,323 (10.6%) | 0.07 | 16,785 (12.8%) | 3,709 (11.0%) | 0.06 |
| Use of Low Intensity Statins; n (%) | 11,986 (31.6%) | 3,096 (25.9%) | 0.13 | 31,153 (33.6%) | 5,929 (27.1%) | 0.14 | 43139 (33.0%) | 9,025 (26.7%) | 0.14 |
| Use of High Intensity Statins; n (%) | 12,278 (32.3%) | 3,103 (26.0%) | 0.14 | 28,435 (30.6%) | 4,919 (22.5%) | 0.18 | 40713 (31.1%) | 8,022 (23.7%) | 0.17 |
| Malignant hypertension; n (%) | 1,131 (3.0%) | 320 (2.7%) | 0.02 | 28,309 (30.5%) | 8,199 (37.5%) | -0.15 | 29440 (22.5%) | 8,519 (25.2%) | -0.06 |
| Cardiovascular stress test; n (%) | 110 (0.3%) | 38 (0.3%) | 0.00 | 292 (0.3%) | 80 (0.4%) | -0.02 | 0,402 (0.3%) | 118 (0.3%) | 0.00 |
| Echocardiogram; n (%) | 9,024 (23.8%) | 1,883 (15.8%) | 0.20 | 26,426 (28.5%) | 3,831 (17.5%) | 0.26 | 35,450 (27.1%) | 5714 (16.9%) | 0.25 |
| Number of BNP tests | 0.05 (0.00) | 0.05 (0.00) | | 0.00 (0.00) | 0.00 (0.00) | | ( ) | 0.00 (0.04) | |
| mean (sd) | 0.06 (0.32) | 0.06 (0.29) | 0.00 | 0.03 (0.22) | 0.02 (0.20) | 0.05 | 0.04 (0.25) | 0.03 (0.24) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.25) | 0.00 (0.24) | 0.00 |
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK)<br>mean (sd) | 0.42 (1.56) | 0.29 (1.07) | 0.10 | 0.23 (1.03) | 0.17 (0.93) | 0.06 | 0.29 (1.21) | 0.21 (0.98) | 0.07 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.21) | 0.00 (0.98) | 0.00 |
| Number of Ambulatory Blood pressure<br>monitoring tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (2.22) | 0.00 (0.50) | |
| mean (sd) | 0.00 (0.06) | 0.00 (0.06) | 0.00 | 0.00 (0.06) | 0.00 (0.07) | 0.00 | 0.00 (0.06) | 0.00 (0.07) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.06) | 0.00 (0.07) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | |
| during baseline | | | | | | | | | - 1 |
| mean (sd) | 75.24 (73.17) | 86.41 (73.17) | -0.15 | 86.01 (74.38) | 90.27 (72.25) | -0.06 | 82.88 (74.03) | 88.91 (72.58) | -0.08 |
| median [IQR] | 58.00 [1.00, 159.00] | 83.00 [1.00, 167.00] | -0.34 | 82.00 [1.00, 168.00] | 87.00 [1.00, 169.00] | -0.07 | 75.03 (74.03) | 85.59 (72.58) | -0.14 |
| N of days in database anytime prior | | | | | | | | | - 1 |
| mean (sd) | 1,454.93 (1,091.34) | 1,700.65 (1,241.25) | -0.21 | 1,460.72 (1,093.13) | 1,710.55 (1,132.92) | -0.22 | 1459.04 (1092.61) | 1707.05 (1172.35) | -0.22 |
| median [IQR] | 1,164.00 [623.00,<br>1,976.00] | 1,383.00 [753.00,<br>2,317.00] | -0.19 | 1,140.00 [622.00,<br>2,024.00] | 1,484.00 [789.00,<br>2,428.00] | -0.31 | 1146.97 (1092.61) | 1448.30 (1172.35) | -0.27 |

Table 1: Telmisartan vs Ramipril

| Mean Copay for per prescription cost | 1 | | | | | | | | - 1 |
|---|---|---|---|---|---|---|---|---|---|
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 32.53 (40.29) | 30.00 (37.37) | 0.07 | 23.24 (25.91) | 23.56 (26.11) | -0.01 | 25.94 (30.78) | 25.84 (30.57) | 0.00 |
| median [IQR] | 23.33 [10.13, 40.52] | 21.04 [8.60, 37.65] | 0.06 | 17.35 [6.24, 32.14] | 17.74 [6.69, 32.48] | -0.01 | 19.09 (30.78) | 18.91 (30.57) | 0.01 |
| Missing; n (%) | 3,106 (8.2%) | 738 (6.2%) | 0.08 | 5,692 (6.1%) | 1,063 (4.9%) | 0.05 | 8,798 (6.7%) | 1801 (5.3%) | 0.06 |
| Colonos; n (%) | 1,792 (4.7%) | 563 (4.7%) | 0.00 | 5,008 (5.4%) | 1,161 (5.3%) | 0.00 | 6,800 (5.2%) | 1724 (5.1%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 1,914 (5.0%) | 611 (5.1%) | 0.00 | 3,485 (3.8%) | 800 (3.7%) | 0.01 | 5,399 (4.1%) | 1411 (4.2%) | -0.01 |
| Flu vaccine; n (%) | 5,787 (15.2%) | 1,904 (15.9%) | -0.02 | 8,869 (9.6%) | 2,177 (10.0%) | -0.01 | 14,656 (11.2%) | 4081 (12.1%) | -0.03 |
| Mammogram; n (%) | 2,932 (7.7%) | 1,576 (13.2%) | -0.18 | 6,866 (7.4%) | 2,526 (11.5%) | -0.14 | 9,798 (7.5%) | 4102 (12.1%) | -0.16 |
| Pap smear; n (%) | 1,133 (3.0%) | 519 (4.3%) | -0.07 | 2,971 (3.2%) | 1,074 (4.9%) | -0.09 | 4,104 (3.1%) | 1593 (4.7%) | -0.08 |
| Pneumonia vaccine; n (%) | 3,129 (8.2%) | 1,237 (10.3%) | -0.07 | 3,097 (3.3%) | 695 (3.2%) | 0.01 | 6,226 (4.8%) | 1932 (5.7%) | -0.04 |
| PSA test or Prostate exam for DRE; n (%) | 6,733 (17.7%) | 1,741 (14.6%) | 0.08 | 10,296 (11.1%) | 1,977 (9.0%) | 0.07 | 17,029 (13.0%) | 3718 (11.0%) | 0.06 |
| Bone mineral density; n (%) | 1,041 (2.7%) | 547 (4.6%) | -0.10 | 1,784 (1.9%) | 684 (3.1%) | -0.08 | 2,825 (2.2%) | 1231 (3.6%) | -0.08 |
| Use of Sympatomimetic agents; n (%) | 472 (1.2%) | 150 (1.3%) | -0.01 | 1,832 (2.0%) | 444 (2.0%) | 0.00 | 2,304 (1.8%) | 594 (1.8%) | 0.00 |
| Use of CNS stimulants; n (%) | 164 (0.4%) | 77 (0.6%) | -0.03 | 596 (0.6%) | 188 (0.9%) | -0.03 | 0,760 (0.6%) | 265 (0.8%) | -0.02 |
| Use of estrogens, progestins, androgens; n<br>(%) | 1,423 (3.7%) | 612 (5.1%) | -0.07 | 4,658 (5.0%) | 1,612 (7.4%) | -0.10 | 6,081 (4.6%) | 2224 (6.6%) | -0.09 |
| Use of Angiogenesis inhibitors; n (%) | 15 (0.0%) | 5 (0.0%) | #DIV/0! | 60 (0.1%) | 12 (0.1%) | 0.00 | 0,075 (0.1%) | 17 (0.1%) | 0.00 |
| | | | 0.00 | | | -0.02 | | | 0.00 |
| Use of Oral Immunosuppressants; n (%) | 70 (0.2%) | 25 (0.2%) | 0.00 | 215 (0.2%) | 56 (0.3%) | 0.02 | 0,285 (0.2%) | 81 (0.2%) | 0.00 |
| Cardiomegaly, LVH, and other cardiopathy<br>due to hypertension; n (%) | 4,467 (11.8%) | 1,343 (11.2%) | 0.02 | 7,841 (8.4%) | 1,788 (8.2%) | 0.01 | 12,308 (9.4%) | 3131 (9.3%) | 0.00 |
| Ultrasound; n (%) | 7,429 (19.6%) | 2,288 (19.1%) | 0.01 | 21,445 (23.1%) | 4,601 (21.0%) | 0.05 | 28,874 (22.1%) | 6889 (20.4%) | 0.04 |
| Symptomatic hypotension; n (%) | 1,117 (2.9%) | 209 (1.7%) | 0.08 | 1,677 (1.8%) | 248 (1.1%) | 0.06 | 2,794 (2.1%) | 457 (1.4%) | 0.05 |
| Syncopal episodes; n (%) | 678 (1.8%) | 270 (2.3%) | -0.04 | 1,252 (1.3%) | 330 (1.5%) | -0.02 | 1,930 (1.5%) | 600 (1.8%) | -0.02 |
| N of Generic name drugs only | | | | | | | | | |
| mean (sd) | 9.94 (11.91) | 11.40 (12.37) | -0.12 | 8.09 (8.46) | 8.54 (8.60) | -0.05 | 8.63 (9.59) | 9.55 (10.09) | -0.09 |
| median [IQR] | 6.00 [2.00, 14.00] | 8.00 [3.00, 16.00] | -0.16 | 6.00 [2.00, 11.00] | 6.00 [2.00, 12.00] | 0.00 | 6.00 (9.59) | 6.71 (10.09) | -0.07 |
| N of Brand name drugs only | | | | | | | | | |
| mean (sd) | 4.71 (6.39) | 4.59 (6.18) | 0.02 | 5.95 (6.84) | 5.70 (6.42) | 0.04 | 5.59 (6.71) | 5.31 (6.34) | 0.04 |
| median [IQR] | 2.00 [0.00, 7.00] | 2.00 [0.00, 6.00] | 0.00 | 4.00 [1.00, 8.00] | 4.00 [1.00, 8.00] | 0.00 | 3.42 (6.71) | 3.29 (6.34) | 0.02 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications (180-1 days before | | | | | | | | | |
| index) | | | | | | | | | |
| mean (sd) | 0.96 (1.12) | 1.13 (1.24) | -0.14 | 1.05 (1.17) | 1.11 (1.22) | -0.05 | 1.02 (1.16) | 1.12 (1.23) | -0.08 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 (1.16) | 1.00 (1.23) | 0.00 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications on CED | | | | | | | | | |
| mean (sd) | 1.41 (0.72) | 1.25 (0.60) | 0.24 | 1.44 (0.75) | 1.26 (0.59) | 0.27 | 1.43 (0.74) | 1.26 (0.59) | 0.25 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 2.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.74) | 1.00 (0.59) | 0.00 |
| Hypertensive retinopathy; n (%) | 271 (0.7%) | 122 (1.0%) | -0.03 | 405 (0.4%) | 118 (0.5%) | -0.01 | 0,676 (0.5%) | 240 (0.7%) | -0.03 |
| Commercial vs Medicare Advantage-<br>Business Type Code - CORRECT ONE -<br>TRUVEN | | | | | | | | | |
| Commercial; n (%) | 18,308 (48.2%) | 5,129 (42.9%) | 0.11 | 51,603 (55.6%) | 12,453 (56.9%) | -0.03 | 69,911 (53.5%) | 17582 (52.0%) | 0.00 |
| Medicare Advantage; n (%) | 19,655 (51.8%) | 6,826 (57.1%) | -0.11 | 41,218 (44.4%) | 9,418 (43.1%) | 0.03 | 60,873 (46.5%) | 16244 (48.0%) | 0.00 |
| Commercial vs Medicare Advantage- | ,, | -,, | | | -,, | | -,,, | | |
| Business Type Code | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 18,308 (48.2%) | 5,129 (42.9%) | 0.11 | - | - | #VALUE! | 18,308 (48.2%) | 5,129 (42.9%) | 0.11 |

Table 1: Telmisartan vs Ramipril

| MCR = MEDICARE; n (%) | 19,655 (51.8%) | 6,826 (57.1%) | -0.11 | - | - | #VALUE! | 19,655 (51.8%) | 6,826 (57.1%) | -0.11 |
|---|---|---|---|---|---|---|---|---|---|
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data | | | | | | | | | |
| Туре | | | | | | | | | - 1 |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 36,614 (39.4%) | 8,586 (39.3%) | 0.00 | 36,614 (39.4%) | 8,586 (39.3%) | 0.00 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 4,604 (5.0%) | 832 (3.8%) | 0.06 | 4,604 (5.0%) | 832 (3.8%) | 0.06 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 47,043 (50.7%) | 11,770 (53.8%) | -0.06 | 47,043 (50.7%) | 11,770 (53.8%) | -0.06 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 4,560 (4.9%) | 683 (3.1%) | 0.09 | 4,560 (4.9%) | 683 (3.1%) | 0.09 |
| Metropolitan Statistical Area - Urban (any | | | | | | | | | |
| MSA) vs Rural (non-MSA) | | | | | | | | | - 1 |
| Urban; n (%) | - | - | #VALUE! | 64,126 (69.1%) | 16,537 (75.6%) | -0.15 | 64,126 (69.1%) | 16,537 (75.6%) | -0.15 |
| Rural; n (%) | - | - | #VALUE! | 844 (0.9%) | 203 (0.9%) | 0.00 | 844 (0.9%) | 203 (0.9%) | 0.00 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 27,851 (30.0%) | 5,131 (23.5%) | 0.15 | 27,851 (30.0%) | 5,131 (23.5%) | 0.15 |

Table 1: Telmisartan vs Ramipril

| | | | F | PS-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | tum | | Truv | en | | POO | LED | |
| Variable | Ramipril (Any dose) | Telmisartan (Any | St. Diff. | Ramipril (Any dose) | Telmisartan (Any | St. Diff. | Ramipril (Any dose) | Telmisartan (Any | St. Diff. |
| Number of patients | 10,798 | 10,798 | | 21,074 | 21,074 | | 31,872 | 31,872 | |
| Age | | | | | | | | | |
| mean (sd) | 69.53 (9.48) | 69.41 (9.22) | 0.01 | 68.68 (9.90) | 68.55 (9.76) | 0.01 | 68.97 (9.76) | 68.84 (9.58) | 0.01 |
| median [IQR] | 69.00 [62.00, 76.00] | 69.00 [62.00, 76.00] | 0.00 | 67.00 [60.00, | 67.00 [60.00, | 0.00 | 67.68 (9.76) | 67.68 (9.58) | 0.00 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| 55 - 64; n (%) | 3,668 (34.0%) | 3,655 (33.8%) | 0.00 | 9,212 (43.7%) | 9,304 (44.1%) | -0.01 | 12,880 (40.4%) | 12,959 (40.7%) | -0.01 |
| 65 - 74; n (%) | 3,738 (34.6%) | 3,815 (35.3%) | -0.01 | 5,632 (26.7%) | 5,604 (26.6%) | 0.00 | 9,370 (29.4%) | 9,419 (29.6%) | 0.00 |
| >=75; n (%) | 3,392 (31.4%) | 3,328 (30.8%) | 0.01 | 6,230 (29.6%) | 6,166 (29.3%) | 0.01 | 9,622 (30.2%) | 9,494 (29.8%) | 0.01 |
| Gender | | | | | | | | | |
| Males; n (%) | 4,912 (45.5%) | 4,984 (46.2%) | -0.01 | 9,692 (46.0%) | 9,823 (46.6%) | -0.01 | 14,604 (45.8%) | 14,807 (46.5%) | -0.01 |
| Females; n (%) | 5,886 (54.5%) | 5,814 (53.8%) | 0.01 | 11,382 (54.0%) | 11,251 (53.4%) | 0.01 | 17,268 (54.2%) | 17,065 (53.5%) | 0.01 |
| Region | | | | | | | | | |
| Northeast; n (%) | 1,185 (11.0%) | 1,125 (10.4%) | 0.02 | 2,950 (14.0%) | 3,023 (14.3%) | -0.01 | 4,135 (13.0%) | 4,148 (13.0%) | 0.00 |
| South; n (%) | 6,441 (59.6%) | 6,556 (60.7%) | -0.02 | 5,131 (24.3%) | 5,035 (23.9%) | 0.01 | 11,572 (36.3%) | 11,591 (36.4%) | 0.00 |
| Midwest; n (%) | 1,350 (12.5%) | 1,308 (12.1%) | 0.01 | 9,833 (46.7%) | 9,916 (47.1%) | -0.01 | 11,183 (35.1%) | 11,224 (35.2%) | 0.00 |
| West; n (%) | 1,822 (16.9%) | 1,809 (16.8%) | 0.00 | 3,021 (14.3%) | 2,968 (14.1%) | 0.01 | 4,843 (15.2%) | 4,777 (15.0%) | 0.01 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 139 (0.7%) | 132 (0.6%) | 0.01 | 139 (0.4%) | 132 (0.4%) | 0.00 |
| CV Covariates | | | | | | | | | |
| lschemic heart disease; n (%) | 3,469 (32.1%) | 3,519 (32.6%) | -0.01 | 5,902 (28.0%) | 5,947 (28.2%) | 0.00 | 9,371 (29.4%) | 9,466 (29.7%) | -0.01 |
| Acute MI; n (%) | 190 (1.8%) | 209 (1.9%) | -0.01 | 340 (1.6%) | 344 (1.6%) | 0.00 | 530 (1.7%) | 553 (1.7%) | 0.00 |
| ACS/unstable angina; n (%) | 282 (2.6%) | 314 (2.9%) | -0.02 | 627 (3.0%) | 655 (3.1%) | -0.01 | 909 (2.9%) | 969 (3.0%) | -0.01 |
| Old MI; n (%) | 494 (4.6%) | 504 (4.7%) | 0.00 | 349 (1.7%) | 354 (1.7%) | 0.00 | 843 (2.6%) | 858 (2.7%) | -0.01 |
| Stable angina; n (%) | 721 (6.7%) | 768 (7.1%) | -0.02 | 1,166 (5.5%) | 1,174 (5.6%) | 0.00 | 1,887 (5.9%) | 1,942 (6.1%) | -0.01 |
| Coronary atherosclerosis and other forms<br>of chronic ischemic heart disease; n (%) | 3,081 (28.5%) | 3,093 (28.6%) | 0.00 | 5,064 (24.0%) | 5,133 (24.4%) | -0.01 | 8,145 (25.6%) | 8,226 (25.8%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 231 (2.1%) | 208 (1.9%) | 0.01 | 336 (1.6%) | 354 (1.7%) | -0.01 | 567 (1.8%) | 562 (1.8%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent); n (%) | 161 (1.5%) | 141 (1.3%) | 0.02 | 329 (1.6%) | 293 (1.4%) | 0.02 | 490 (1.5%) | 434 (1.4%) | 0.01 |
| History of CABG or PTCA; n (%) | 756 (7.0%) | 771 (7.1%) | 0.00 | 479 (2.3%) | 525 (2.5%) | -0.01 | 1,235 (3.9%) | 1,296 (4.1%) | -0.01 |
| Any stroke; n (%) | 1,668 (15.4%) | 1,634 (15.1%) | 0.01 | 3,038 (14.4%) | 2,955 (14.0%) | 0.01 | 4,706 (14.8%) | 4,589 (14.4%) | 0.01 |
| Ischemic stroke (w and w/o mention of<br>cerebral infarction); n (%) | 1,649 (15.3%) | 1,622 (15.0%) | 0.01 | 3,018 (14.3%) | 2,932 (13.9%) | 0.01 | 4,667 (14.6%) | 4,554 (14.3%) | 0.01 |
| Hemorrhagic stroke; n (%) | 43 (0.4%) | 37 (0.3%) | 0.02 | 66 (0.3%) | 58 (0.3%) | 0.00 | 109 (0.3%) | 95 (0.3%) | 0.00 |
| TIA; n (%) | 464 (4.3%) | 475 (4.4%) | 0.00 | 847 (4.0%) | 833 (4.0%) | 0.00 | 1311 (4.1%) | 1308 (4.1%) | 0.00 |
| Other cerebrovascular disease; n (%) | 365 (3.4%) | 338 (3.1%) | 0.02 | 508 (2.4%) | 456 (2.2%) | 0.01 | 873 (2.7%) | 794 (2.5%) | 0.01 |
| Late effects of cerebrovascular disease; n<br>(%) | 285 (2.6%) | 263 (2.4%) | 0.01 | 296 (1.4%) | 293 (1.4%) | 0.00 | 581 (1.8%) | 556 (1.7%) | 0.01 |
| Cerebrovascular procedure; n (%) | 40 (0.4%) | 35 (0.3%) | 0.02 | 71 (0.3%) | 86 (0.4%) | -0.02 | 111 (0.3%) | 121 (0.4%) | -0.02 |
| Heart failure (CHF); n (%) | 857 (7.9%) | 830 (7.7%) | 0.01 | 1,058 (5.0%) | 1,005 (4.8%) | 0.01 | 1,915 (6.0%) | 1,835 (5.8%) | 0.01 |
| Peripheral Vascular Disease (PVD) or PVD<br>Surgery ; n (%) | 1,149 (10.6%) | 1,123 (10.4%) | 0.01 | 1,564 (7.4%) | 1,518 (7.2%) | 0.01 | 2,713 (8.5%) | 2,641 (8.3%) | 0.01 |
| Atrial fibrillation; n (%) | 871 (8.1%) | 864 (8.0%) | 0.00 | 1,409 (6.7%) | 1,390 (6.6%) | 0.00 | 2,280 (7.2%) | 2,254 (7.1%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 1,232 (11.4%) | 1,199 (11.1%) | 0.01 | 1,617 (7.7%) | 1,665 (7.9%) | -0.01 | 2,849 (8.9%) | 2,864 (9.0%) | 0.00 |

Table 1: Telmisartan vs Ramipril

| Cardiac conduction disorders; n (%) | 307 (2.8%) | 322 (3.0%) | -0.01 | 399 (1.9%) | 386 (1.8%) | 0.01 | 706 (2.2%) | 708 (2.2%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Other CVD; n (%) | 1,543 (14.3%) | 1,568 (14.5%) | -0.01 | 2,604 (12.4%) | 2,508 (11.9%) | 0.02 | 4,147 (13.0%) | 4,076 (12.8%) | 0.01 |
| Diabetes-related complications | 1,545 (14.570) | 1,500 (14.570) | 0.01 | 2,001(12.170) | 2,500 (11.570) | 0.02 | 4,147 (13.070) | 4,070 (12.0%) | 0.01 |
| Diabetic retinopathy; n (%) | 675 (6.3%) | 673 (6.2%) | 0.00 | 791 (3.8%) | 819 (3.9%) | -0.01 | 1,466 (4.6%) | 1,492 (4.7%) | 0.00 |
| Diabetes with other ophthalmic | 45 (0.4%) | 51 (0.5%) | -0.01 | 603 (2.9%) | 578 (2.7%) | 0.01 | 0,648 (2.0%) | 0,629 (2.0%) | 0.00 |
| manifestations; n (%) | | | | | | | | | |
| Retinal detachment, vitreous hemorrhage,<br>vitrectomy; n (%) | 69 (0.6%) | 56 (0.5%) | 0.01 | 74 (0.4%) | 79 (0.4%) | 0.00 | 143 (0.4%) | 135 (0.4%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 79 (0.7%) | 87 (0.8%) | -0.01 | 176 (0.8%) | 176 (0.8%) | 0.00 | 255 (0.8%) | 263 (0.8%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n (%) | 1,350 (12.5%) | 1,373 (12.7%) | -0.01 | 1,384 (6.6%) | 1,389 (6.6%) | 0.00 | 2,734 (8.6%) | 2,762 (8.7%) | 0.00 |
| Occurrence of diabetic nephropathy with ICD10; n (%) | 945 (8.8%) | 926 (8.6%) | 0.01 | 682 (3.2%) | 717 (3.4%) | -0.01 | 1,627 (5.1%) | 1,643 (5.2%) | 0.00 |
| Hypoglycemia; n (%) | 169 (1.6%) | 154 (1.4%) | 0.02 | 331 (1.6%) | 305 (1.4%) | 0.02 | 0,500 (1.6%) | 0,459 (1.4%) | 0.02 |
| Hyperglycemia; n (%) | 363 (3.4%) | 377 (3.5%) | -0.01 | 290 (1.4%) | 297 (1.4%) | 0.00 | 0,653 (2.0%) | 0,674 (2.1%) | -0.01 |
| Disorders of fluid electrolyte and acid-base | 746 (6.9%) | 737 (6.8%) | 0.00 | 846 (4.0%) | 831 (3.9%) | 0.01 | 1,592 (5.0%) | 1,568 (4.9%) | 0.00 |
| balance; n (%) | | | | | | | | | |
| Diabetic ketoacidosis; n (%) | 29 (0.3%) | 21 (0.2%) | 0.02 | 34 (0.2%) | 27 (0.1%) | 0.03 | 63 (0.2%) | 48 (0.2%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic<br>syndrome (HONK); n (%) | 25 (0.2%) | 23 (0.2%) | 0.00 | 27 (0.1%) | 23 (0.1%) | 0.00 | 52 (0.2%) | 46 (0.1%) | 0.03 |
| Diabetes with peripheral circulatory disorders with ICD-10; n (%) | 428 (4.0%) | 434 (4.0%) | 0.00 | 354 (1.7%) | 358 (1.7%) | 0.00 | 0,782 (2.5%) | 0,792 (2.5%) | 0.00 |
| Diabetic Foot; n (%) | 323 (3.0%) | 301 (2.8%) | 0.01 | 577 (2.7%) | 566 (2.7%) | 0.00 | 900 (2.8%) | 867 (2.7%) | 0.01 |
| Gangrene; n (%) | 24 (0.2%) | 22 (0.2%) | 0.00 | 23 (0.1%) | 24 (0.1%) | 0.00 | 47 (0.1%) | 46 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 65 (0.6%) | 61 (0.6%) | 0.00 | 48 (0.2%) | 44 (0.2%) | 0.00 | 113 (0.4%) | 105 (0.3%) | 0.02 |
| Osteomyelitis; n (%) | 76 (0.7%) | 61 (0.6%) | 0.01 | 104 (0.5%) | 85 (0.4%) | 0.01 | 180 (0.6%) | 146 (0.5%) | 0.01 |
| Skin infections; n (%) | 622 (5.8%) | 581 (5.4%) | 0.02 | 1,087 (5.2%) | 1,066 (5.1%) | 0.00 | 1,709 (5.4%) | 1,647 (5.2%) | 0.01 |
| Erectile dysfunction; n (%) | 279 (2.6%) | 290 (2.7%) | -0.01 | 243 (1.2%) | 271 (1.3%) | -0.01 | 0,522 (1.6%) | 0,561 (1.8%) | -0.02 |
| Diabetes with unspecified complication; n (%) | 291 (2.7%) | 286 (2.6%) | 0.01 | 351 (1.7%) | 339 (1.6%) | 0.01 | 0,642 (2.0%) | 0,625 (2.0%) | 0.00 |
| Diabetes mellitus without mention of complications; n (%) | 4,622 (42.8%) | 4,599 (42.6%) | 0.00 | 7,440 (35.3%) | 7,412 (35.2%) | 0.00 | 12,062 (37.8%) | 12,011 (37.7%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 9,425 (87.3%) | 9,377 (86.8%) | 0.01 | 14,509 (68.8%) | 14,543 (69.0%) | 0.00 | 23,934 (75.1%) | 23,920 (75.1%) | 0.00 |
| Hyperlipidemia ; n (%) | 6,924 (64.1%) | 6,904 (63.9%) | 0.00 | 8,046 (38.2%) | 8,175 (38.8%) | -0.01 | 14,970 (47.0%) | 15,079 (47.3%) | -0.01 |
| Edema; n (%) | 829 (7.7%) | 826 (7.6%) | 0.00 | 968 (4.6%) | 944 (4.5%) | 0.00 | 1,797 (5.6%) | 1,770 (5.6%) | 0.00 |
| Renal Dysfunction (non-diabetic); n (%) | 1,958 (18.1%) | 1,937 (17.9%) | 0.01 | 2,085 (9.9%) | 2,082 (9.9%) | 0.00 | 4,043 (12.7%) | 4,019 (12.6%) | 0.00 |
| Occurrence of acute renal disease; n (%) | 250 (2.3%) | 243 (2.3%) | 0.00 | 280 (1.3%) | 281 (1.3%) | 0.00 | 530 (1.7%) | 524 (1.6%) | 0.01 |
| Occurrence of chronic renal insufficiency;<br>n (%) | 1,567 (14.5%) | 1,508 (14.0%) | 0.01 | 1,458 (6.9%) | 1,446 (6.9%) | 0.00 | 3,025 (9.5%) | 2,954 (9.3%) | 0.01 |
| Chronic kidney disease ; n (%) | 1,480 (13.7%) | 1,433 (13.3%) | 0.01 | 1,339 (6.4%) | 1,336 (6.3%) | 0.00 | 2,819 (8.8%) | 2,769 (8.7%) | 0.00 |
| CKD Stage 3-4; n (%) | 989 (9.2%) | 933 (8.6%) | 0.02 | 789 (3.7%) | 830 (3.9%) | -0.01 | 1,778 (5.6%) | 1,763 (5.5%) | 0.00 |
| Occurrence of hypertensive nephropathy;<br>n (%) | 722 (6.7%) | 730 (6.8%) | 0.00 | 572 (2.7%) | 539 (2.6%) | 0.01 | 1294 (4.1%) | 1269 (4.0%) | 0.01 |
| Occurrence of miscellaneous renal | 604 (5.6%) | 603 (5.6%) | 0.00 | 728 (3.5%) | 718 (3.4%) | 0.01 | 1,332 (4.2%) | 1,321 (4.1%) | 0.01 |
| insufficiency; n (%) | . , | | | | . , | | | | l |
| Glaucoma or cataracts ; n (%) | 2,158 (20.0%) | 2,251 (20.8%) | -0.02 | 3,746 (17.8%) | 3,780 (17.9%) | 0.00 | 5,904 (18.5%) | 6,031 (18.9%) | -0.01 |
| Cellulitis or abscess of toe; n (%) | 143 (1.3%) | 120 (1.1%) | 0.02 | 155 (0.7%) | 143 (0.7%) | 0.00 | 298 (0.9%) | 263 (0.8%) | 0.01 |
| Foot ulcer; n (%) | 328 (3.0%) | 311 (2.9%) | 0.01 | 591 (2.8%) | 576 (2.7%) | 0.01 | 919 (2.9%) | 887 (2.8%) | 0.01 |

Table 1: Telmisartan vs Ramipril

| Bladder stones; n (%) | 20 (0.2%) | 12 (0.1%) | 0.03 | 29 (0.1%) | 21 (0.1%) | 0.00 | 49 (0.2%) | 33 (0.1%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Kidney stones; n (%) | 225 (2.1%) | 219 (2.0%) | 0.01 | 335 (1.6%) | 349 (1.7%) | -0.01 | 0,560 (1.8%) | 0,568 (1.8%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | 1,097 (10.2%) | 1,071 (9.9%) | 0.01 | 1,349 (6.4%) | 1,322 (6.3%) | 0.00 | 2,446 (7.7%) | 2,393 (7.5%) | 0.01 |
| Dipstick urinalysis; n (%) | 3,856 (35.7%) | 3,902 (36.1%) | -0.01 | 5,162 (24.5%) | 5,125 (24.3%) | 0.00 | 9,018 (28.3%) | 9,027 (28.3%) | 0.00 |
| Non-dipstick urinalysis; n (%) | 2,413 (22.3%) | 2,359 (21.8%) | 0.01 | 2,434 (11.5%) | 2,386 (11.3%) | 0.01 | 4,847 (15.2%) | 4,745 (14.9%) | 0.01 |
| Urine function test; n (%) | 344 (3.2%) | 298 (2.8%) | 0.02 | 617 (2.9%) | 688 (3.3%) | -0.02 | 0,961 (3.0%) | 0,986 (3.1%) | -0.01 |
| Cytology; n (%) | 163 (1.5%) | 128 (1.2%) | 0.03 | 357 (1.7%) | 308 (1.5%) | 0.02 | 520 (1.6%) | 436 (1.4%) | 0.02 |
| Cystos; n (%) | 226 (2.1%) | 204 (1.9%) | 0.01 | 471 (2.2%) | 428 (2.0%) | 0.01 | 697 (2.2%) | 632 (2.0%) | 0.01 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 230 (2.1%) | 249 (2.3%) | -0.01 | 150 (0.7%) | 160 (0.8%) | -0.01 | 0,380 (1.2%) | 0,409 (1.3%) | -0.01 |
| Osteoarthritis; n (%) | 1,871 (17.3%) | 1,879 (17.4%) | 0.00 | 2,725 (12.9%) | 2,734 (13.0%) | 0.00 | 4,596 (14.4%) | 4,613 (14.5%) | 0.00 |
| Other arthritis, arthropathies and | 4,118 (38.1%) | 4,111 (38.1%) | 0.00 | 6,818 (32.4%) | 6,762 (32.1%) | 0.01 | 10,936 (34.3%) | 10,873 (34.1%) | 0.00 |
| musculoskeletal pain; n (%) | | | | | | | | | |
| Dorsopathies; n (%) | 2,521 (23.3%) | 2,520 (23.3%) | 0.00 | 4,212 (20.0%) | 4,191 (19.9%) | 0.00 | 6,733 (21.1%) | 6,711 (21.1%) | 0.00 |
| Fractures; n (%) | 386 (3.6%) | 394 (3.6%) | 0.00 | 718 (3.4%) | 703 (3.3%) | 0.01 | 1,104 (3.5%) | 1,097 (3.4%) | 0.01 |
| Falls; n (%) | 325 (3.0%) | 328 (3.0%) | 0.00 | 126 (0.6%) | 133 (0.6%) | 0.00 | 451 (1.4%) | 461 (1.4%) | 0.00 |
| Osteoporosis; n (%) | 935 (8.7%) | 937 (8.7%) | 0.00 | 1,657 (7.9%) | 1,641 (7.8%) | 0.00 | 2,592 (8.1%) | 2,578 (8.1%) | 0.00 |
| Hyperthyroidism; n (%) | 88 (0.8%) | 93 (0.9%) | -0.01 | 96 (0.5%) | 96 (0.5%) | 0.00 | 184 (0.6%) | 189 (0.6%) | 0.00 |
| Hypothyroidism; n (%) | 1,759 (16.3%) | 1,686 (15.6%) | 0.02 | 1,896 (9.0%) | 1,814 (8.6%) | 0.01 | 3,655 (11.5%) | 3,500 (11.0%) | 0.02 |
| Other disorders of thyroid gland; n (%) | 396 (3.7%) | 460 (4.3%) | -0.03 | 554 (2.6%) | 606 (2.9%) | -0.02 | 0,950 (3.0%) | 1,066 (3.3%) | -0.02 |
| Depression; n (%) | 835 (7.7%) | 813 (7.5%) | 0.01 | 1,017 (4.8%) | 1,012 (4.8%) | 0.00 | 1,852 (5.8%) | 1,825 (5.7%) | 0.00 |
| Anxiety; n (%) | 747 (6.9%) | 774 (7.2%) | -0.01 | 664 (3.2%) | 674 (3.2%) | 0.00 | 1,411 (4.4%) | 1,448 (4.5%) | 0.00 |
| SleepDisorder; n (%) | 825 (7.6%) | 818 (7.6%) | 0.00 | 1,721 (8.2%) | 1,678 (8.0%) | 0.01 | 2,546 (8.0%) | 2,496 (7.8%) | 0.01 |
| Dementia; n (%) | 440 (4.1%) | 435 (4.0%) | 0.01 | 558 (2.6%) | 535 (2.5%) | 0.01 | 998 (3.1%) | 970 (3.0%) | 0.01 |
| Delirium; n (%) | 130 (1.2%) | 118 (1.1%) | 0.01 | 156 (0.7%) | 162 (0.8%) | -0.01 | 286 (0.9%) | 280 (0.9%) | 0.00 |
| Psychosis; n (%) | 94 (0.9%) | 89 (0.8%) | 0.01 | 116 (0.6%) | 121 (0.6%) | 0.00 | 210 (0.7%) | 210 (0.7%) | 0.00 |
| Obesity; n (%) | 1,239 (11.5%) | 1,229 (11.4%) | 0.00 | 948 (4.5%) | 978 (4.6%) | 0.00 | 2,187 (6.9%) | 2,207 (6.9%) | 0.00 |
| Overweight; n (%) | 405 (3.8%) | 401 (3.7%) | 0.01 | 175 (0.8%) | 160 (0.8%) | 0.00 | 0,580 (1.8%) | 0,561 (1.8%) | 0.00 |
| Smoking; n (%) | 928 (8.6%) | 974 (9.0%) | -0.01 | 660 (3.1%) | 655 (3.1%) | 0.00 | 1,588 (5.0%) | 1,629 (5.1%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 78 (0.7%) | 67 (0.6%) | 0.01 | 71 (0.3%) | 79 (0.4%) | -0.02 | 149 (0.5%) | 146 (0.5%) | 0.00 |
| Drug abuse or dependence; n (%) | 113 (1.0%) | 118 (1.1%) | -0.01 | 78 (0.4%) | 73 (0.3%) | 0.02 | 191 (0.6%) | 191 (0.6%) | 0.00 |
| COPD; n (%) | 1,134 (10.5%) | 1,166 (10.8%) | -0.01 | 1,702 (8.1%) | 1,683 (8.0%) | 0.00 | 2,836 (8.9%) | 2,849 (8.9%) | 0.00 |
| Asthma; n (%) | 622 (5.8%) | 628 (5.8%) | 0.00 | 1,026 (4.9%) | 1,026 (4.9%) | 0.00 | 1,648 (5.2%) | 1,654 (5.2%) | 0.00 |
| Obstructive sleep apnea; n (%) | 731 (6.8%) | 720 (6.7%) | 0.00 | 1,187 (5.6%) | 1,193 (5.7%) | 0.00 | 1,918 (6.0%) | 1,913 (6.0%) | 0.00 |
| Pneumonia; n (%) | 277 (2.6%) | 269 (2.5%) | 0.01 | 465 (2.2%) | 479 (2.3%) | -0.01 | 0,742 (2.3%) | 0,748 (2.3%) | 0.00 |
| Imaging; n (%) | 18 (0.2%) | 24 (0.2%) | 0.00 | 11 (0.1%) | 17 (0.1%) | 0.00 | 29 (0.1%) | 41 (0.1%) | 0.00 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 10,798 (100.0%) | 268 (2.5%) | 8.83 | 21,074 (100.0%) | 471 (2.2%) | 9.43 | 31,872 (100.0%) | 0,739 (2.3%) | 9.22 |
| Use of ARBs; n (%) | 132 (1.2%) | 10,798 (100.0%) | -12.83 | 268 (1.3%) | 21,074 (100.0%) | -12.32 | 0.400 (1.3%) | 31,872 (100.0%) | -12.32 |
| Use of Loop Diuretics - ; n (%) | 1,441 (13.3%) | 1,399 (13.0%) | 0.01 | 2,988 (14.2%) | 2,905 (13.8%) | 0.01 | 4,429 (13.9%) | 4,304 (13.5%) | 0.01 |
| Use of other diuretics-; n (%) | 246 (2.3%) | 249 (2.3%) | 0.00 | 544 (2.6%) | 525 (2.5%) | 0.01 | 0,790 (2.5%) | 0,774 (2.4%) | 0.01 |
| Use of nitrates-; n (%) | 790 (7.3%) | 805 (7.5%) | -0.01 | 1,974 (9.4%) | 1,929 (9.2%) | 0.01 | 2,764 (8.7%) | 2,734 (8.6%) | 0.00 |
| Use of other hypertension drugs; n (%) | 854 (7.9%) | 872 (8.1%) | -0.01 | 1,577 (7.5%) | 1,602 (7.6%) | 0.00 | 2,431 (7.6%) | 2,474 (7.8%) | -0.01 |
| Use of digoxin-; n (%) | 185 (1.7%) | 200 (1.9%) | -0.02 | 591 (2.8%) | 563 (2.7%) | 0.01 | 776 (2.4%) | 763 (2.4%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 213 (2.0%) | 218 (2.0%) | 0.00 | 489 (2.3%) | 476 (2.3%) | 0.00 | 702 (2.2%) | 694 (2.2%) | 0.00 |
| Use of COPD/asthma meds-; n (%) | 1,650 (15.3%) | 1,668 (15.4%) | 0.00 | 3,684 (17.5%) | 3,673 (17.4%) | 0.00 | 5,334 (16.7%) | 5,341 (16.8%) | 0.00 |
| Use of statins; n (%) | 5,936 (55.0%) | 5,891 (54.6%) | 0.01 | 11,370 (54.0%) | 11,431 (54.2%) | 0.00 | 17,306 (54.3%) | 17,322 (54.3%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 1,241 (11.5%) | 1,192 (11.0%) | 0.02 | 2,807 (13.3%) | 2,838 (13.5%) | -0.01 | 4,048 (12.7%) | 4,030 (12.6%) | 0.00 |
| | -, (-1.570) | -, () | 2.02 | _, | 2,000 (20.070) | | ., | ., | 5.50 |

Table 1: Telmisartan vs Ramipril

| Use of oral anticoagulants (Dabigatran, | 699 (6.5%) | 702 (6.5%) | 0.00 | 1,505 (7.1%) | 1,492 (7.1%) | 0.00 | 2,204 (6.9%) | 2,194 (6.9%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Rivaroxaban, Apixaban, Warfarin); n (%) | | | | | | | | | |
| Use of heparin and other low-molecular | 51 (0.5%) | 56 (0.5%) | 0.00 | 14 (0.1%) | 4 (0.0%) | 0.04 | 65 (0.2%) | 60 (0.2%) | 0.00 |
| weight heparins; n (%) | () | | | | () | | | | |
| Use of NSAIDs; n (%) | 1,536 (14.2%) | 1,493 (13.8%) | 0.01 | 2,962 (14.1%) | 2,956 (14.0%) | 0.00 | 4,498 (14.1%) | 4,449 (14.0%) | 0.00 |
| Use of oral corticosteroids; n (%) | 1,734 (16.1%) | 1,771 (16.4%) | -0.01 | 3,556 (16.9%) | 3,564 (16.9%) | 0.00 | 5,290 (16.6%) | 5,335 (16.7%) | 0.00 |
| Use of bisphosphonate (); n (%) | 527 (4.9%) | 517 (4.8%) | 0.00 | 1,204 (5.7%) | 1,200 (5.7%) | 0.00 | 1731 (5.4%) | 1717 (5.4%) | 0.00 |
| Use of opioids-; n (%) | 2,755 (25.5%) | 2,771 (25.7%) | 0.00 | 5,922 (28.1%) | 5,931 (28.1%) | 0.00 | 8,677 (27.2%) | 8,702 (27.3%) | 0.00 |
| Use of antidepressants; n (%) | 2,370 (21.9%) | 2,331 (21.6%) | 0.01 | 4,632 (22.0%) | 4,623 (21.9%) | 0.00 | 7,002 (22.0%) | 6,954 (21.8%) | 0.00 |
| Use of antipsychotics; n (%) | 190 (1.8%) | 171 (1.6%) | 0.02 | 386 (1.8%) | 370 (1.8%) | 0.00 | 0,576 (1.8%) | 0,541 (1.7%) | 0.01 |
| Use of anticonvulsants; n (%) | 1,307 (12.1%) | 1,295 (12.0%) | 0.00 | 2,347 (11.1%) | 2,324 (11.0%) | 0.00 | 3,654 (11.5%) | 3,619 (11.4%) | 0.00 |
| Use of lithium-; n (%) | 15 (0.1%) | 9 (0.1%) | 0.00 | 35 (0.2%) | 30 (0.1%) | 0.03 | 50 (0.2%) | 39 (0.1%) | 0.03 |
| Use of Benzos- ; n (%) | 1,248 (11.6%) | 1,225 (11.3%) | 0.01 | 3,252 (15.4%) | 3,189 (15.1%) | 0.01 | 4,500 (14.1%) | 4,414 (13.8%) | 0.01 |
| Use of anxiolytics/hypnotics-; n (%) | 766 (7.1%) | 751 (7.0%) | 0.00 | 1,917 (9.1%) | 1,897 (9.0%) | 0.00 | 2,683 (8.4%) | 2,648 (8.3%) | 0.00 |
| Use of dementia meds- ; n (%) | 294 (2.7%) | 286 (2.6%) | 0.01 | 588 (2.8%) | 576 (2.7%) | 0.01 | 882 (2.8%) | 862 (2.7%) | 0.01 |
| Use of antiparkinsonian meds-; n (%) | 235 (2.2%) | 228 (2.1%) | 0.01 | 519 (2.5%) | 551 (2.6%) | -0.01 | 0,754 (2.4%) | 0,779 (2.4%) | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 4 (0.0%) | 3 (0.0%) | #DIV/0! | 2 (0.0%) | 1 (0.0%) | #DIV/0! | 6 (0.0%) | 4 (0.0%) | #DIV/0! |
| Labs | | | | | | | | | |
| Lab values- HbA1c (%); n (%) | 2,027 (18.8%) | 2,001 (18.5%) | 0.01 | 303 (1.4%) | 280 (1.3%) | 0.01 | 2,330 (7.3%) | 2,281 (7.2%) | 0.00 |
| Lab values- HbA1c (%) (within 3 months) ; n<br>(%) | 1,421 (13.2%) | 1,374 (12.7%) | 0.01 | 204 (1.0%) | 194 (0.9%) | 0.01 | 1,625 (5.1%) | 1,568 (4.9%) | 0.01 |
| Lab values- HbA1c (%) (within 6 months); n | 2,027 (18.8%) | 2,001 (18.5%) | 0.01 | 303 (1.4%) | 280 (1.3%) | 0.01 | 2,330 (7.3%) | 2,281 (7.2%) | 0.00 |
| (%) | | | | | | | | | |
| Lab values- BNP; n (%) | 72 (0.7%) | 71 (0.7%) | 0.00 | 8 (0.0%) | 6 (0.0%) | #DIV/0! | 80 (0.3%) | 77 (0.2%) | 0.02 |
| Lab values- BNP (within 3 months); n (%) | 49 (0.5%) | 47 (0.4%) | 0.01 | 5 (0.0%) | 3 (0.0%) | #DIV/0! | 54 (0.2%) | 50 (0.2%) | 0.00 |
| Lab values-BNP (within 6 months); n (%) | 72 (0.7%) | 71 (0.7%) | 0.00 | 8 (0.0%) | 6 (0.0%) | #DIV/0! | 80 (0.3%) | 77 (0.2%) | 0.02 |
| Lab values- BUN (mg/dl); n (%) | 2,965 (27.5%) | 3,034 (28.1%) | -0.01 | 349 (1.7%) | 335 (1.6%) | 0.01 | 3,314 (10.4%) | 3,369 (10.6%) | -0.01 |
| Lab values-BUN (mg/dl) (within 3 months);<br>n (%) | 2,060 (19.1%) | 2,165 (20.1%) | -0.03 | 240 (1.1%) | 234 (1.1%) | 0.00 | 2,300 (7.2%) | 2,399 (7.5%) | -0.01 |
| Lab values-BUN (mg/dl) (within 6 months);<br>n (%) | 2,965 (27.5%) | 3,034 (28.1%) | -0.01 | 349 (1.7%) | 335 (1.6%) | 0.01 | 3,314 (10.4%) | 3,369 (10.6%) | -0.01 |
| Lab values- Creatinine (mg/dl) ; n (%) | 3,074 (28.5%) | 3,133 (29.0%) | -0.01 | 377 (1.8%) | 366 (1.7%) | 0.01 | 3,451 (10.8%) | 3,499 (11.0%) | -0.01 |
| Lab values- Creatinine (mg/dl) (within 3 | 2,137 (19.8%) | 2,224 (20.6%) | -0.02 | 263 (1.2%) | 256 (1.2%) | 0.00 | 2,400 (7.5%) | 2,480 (7.8%) | -0.01 |
| months); n (%) | -, (, | -,, | | | | | _, (, | -,(, | |
| Lab values- Creatinine (mg/dl) (within 6<br>months) ; n (%) | 3,074 (28.5%) | 3,133 (29.0%) | -0.01 | 377 (1.8%) | 366 (1.7%) | 0.01 | 3,451 (10.8%) | 3,499 (11.0%) | -0.01 |
| Lab values- HDL level (mg/dl); n (%) | 2,339 (21.7%) | 2,294 (21.2%) | 0.01 | 308 (1.5%) | 284 (1.3%) | 0.02 | 2,647 (8.3%) | 2,578 (8.1%) | 0.01 |
| Lab values-HDL level (mg/dl) (within 3<br>months); n (%) | 1,559 (14.4%) | 1,529 (14.2%) | 0.01 | 202 (1.0%) | 181 (0.9%) | 0.01 | 1,761 (5.5%) | 1,710 (5.4%) | 0.00 |
| Lab values-HDL level (mg/dl) (within 6<br>months); n (%) | 2,339 (21.7%) | 2,294 (21.2%) | 0.01 | 308 (1.5%) | 284 (1.3%) | 0.02 | 2,647 (8.3%) | 2,578 (8.1%) | 0.01 |
| Lab values-LDL level (mg/dl) ; n (%) | 2,527 (23.4%) | 2,492 (23.1%) | 0.01 | 312 (1.5%) | 293 (1.4%) | 0.01 | 2,839 (8.9%) | 2,785 (8.7%) | 0.01 |
| Lab values-LDL level (mg/dl) (within 3 | 1,695 (15.7%) | 1,662 (15.4%) | 0.01 | 203 (1.0%) | 187 (0.9%) | 0.01 | 1,898 (6.0%) | 1,849 (5.8%) | 0.01 |
| months); n (%) | _, | _, | | | (0.574) | | -, (0.0.0) | -1- 1- (3.574) | |
| Lab values-LDL level (mg/dl) (within 6 | 2,527 (23.4%) | 2,492 (23.1%) | 0.01 | 312 (1.5%) | 293 (1.4%) | 0.01 | 2,839 (8.9%) | 2,785 (8.7%) | 0.01 |
| months); n (%) | _, | _, ,, | | () | | | _,, | -1 () | |
| Lab values- NT-proBNP; n (%) | 13 (0.1%) | 17 (0.2%) | -0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13 (0.0%) | 17 (0.1%) | -0.04 |
| Lab values- NT-proBNP (within 3 months); | 9 (0.1%) | 8 (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 9 (0.0%) | 8 (0.0%) | #DIV/0! |
| n (%) | | | | | | • | | | • |

Table 1: Telmisartan vs Ramipril

| Lab values-NT-proBNP (within 6 months);<br>n (%) | 13 (0.1%) | 17 (0.2%) | -0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 13 (0.0%) | 17 (0.1%) | -0.04 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values-Total cholesterol (mg/dl); n (%) | 2,519 (23.3%) | 2,497 (23.1%) | 0.00 | 314 (1.5%) | 293 (1.4%) | 0.01 | 2,833 (8.9%) | 2,790 (8.8%) | 0.00 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 1,690 (15.7%) | 1,665 (15.4%) | 0.01 | 207 (1.0%) | 185 (0.9%) | 0.01 | 1,897 (6.0%) | 1,850 (5.8%) | 0.01 |
| Lab values-Total cholesterol (mg/dl)<br>(within 6 months); n (%) | 2,519 (23.3%) | 2,497 (23.1%) | 0.00 | 314 (1.5%) | 293 (1.4%) | 0.01 | 2,833 (8.9%) | 2,790 (8.8%) | 0.00 |
| Lab values-Triglyceride level (mg/dl); n (%) | 2,479 (23.0%) | 2,463 (22.8%) | 0.00 | 314 (1.5%) | 287 (1.4%) | 0.01 | 2,793 (8.8%) | 2,750 (8.6%) | 0.01 |
| Lab values-Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 1,659 (15.4%) | 1,644 (15.2%) | 0.01 | 206 (1.0%) | 183 (0.9%) | 0.01 | 1,865 (5.9%) | 1,827 (5.7%) | 0.01 |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 2,479 (23.0%) | 2,463 (22.8%) | 0.00 | 314 (1.5%) | 287 (1.4%) | 0.01 | 2,793 (8.8%) | 2,750 (8.6%) | 0.01 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 1,968 | 1,935 | | 296 | 270 | | 0 | 0 | |
| mean (sd) | 7.11 (1.65) | 6.98 (1.59) | 0.08 | 7.50 (1.79) | 7.24 (1.62) | 0.15 | 7.37 (1.74) | 7.15 (1.61) | 0.13 |
| median [IQR] | 6.62 [6.00, 7.70] | 6.50 [5.90, 7.60] | 0.07 | 7.10 [6.30, 8.10] | 6.75 [6.10, 8.00] | 0.21 | 6.94 (1.74) | 6.67 (1.61) | 0.16 |
| Missing; n (%) | 8,830 (81.8%) | 8,863 (82.1%) | -0.01 | 20,778 (98.6%) | 20,804 (98.7%) | -0.01 | 29,608 (92.9%) | 29,667 (93.1%) | -0.01 |
| Lab result number- BNP mean | 72 | 71 | | 8 | 6 | | 0 | 0 | |
| mean (sd) | 192.43 (286.24) | 181.05 (419.77) | 0.03 | 55.18 (41.00) | 40.33 (28.20) | 0.42 | 101.68 (169.91) | 88.00 (245.40) | 0.06 |
| median [IQR] | 98.05 [27.50,<br>201.60] | 69.40 [29.50,<br>152.00] | 80.0 | 57.95 [20.50,<br>80.30] | 42.00 [18.00,<br>66.00] | 0.45 | 71.54 (169.91) | 51.28 (245.40) | 0.10 |
| Missing; n (%) | 10,726 (99.3%) | 10,727 (99.3%) | 0.00 | 21,066 (100.0%) | 21,068 (100.0%) | #DIV/0! | 31,792 (99.7%) | 31,795 (99.8%) | -0.02 |
| Lab result number- BUN (mg/dl) mean | 2,965 | 3,034 | | 349 | 335 | | 0 | 0 | |
| mean (sd) | 17.98 (8.45) | -585.70 (21,175.88) | 0.04 | 360.96 (6,422.54) | 645.23 (8,108.67) | -0.04 | 244.76 (5222.51) | 228.20 (13978.25) | 0.00 |
| median [IQR] | 17.00 [13.33, 21.00] | 17.00 [13.33, 22.00] | 0.00 | 16.00 [13.00,<br>21.00] | 16.50 [14.00,<br>21.75] | 0.00 | 16.34 (5222.51) | 16.67 (13978.25) | 0.00 |
| Missing; n (%) | 7,833 (72.5%) | 7,764 (71.9%) | 0.01 | 20,725 (98.3%) | 20,739 (98.4%) | -0.01 | 28,558 (89.6%) | 28,503 (89.4%) | 0.01 |
| Lab result number- Creatinine (mg/dl) | 2,957 | 3,004 | | 371 | 358 | | 3,328 | 3,362 | |
| mean (only 0.1 to 15 included) | | | | | | | | | |
| mean (sd) | 1.04 (0.53) | 1.08 (0.55) | -0.07 | 0.96 (0.36) | 1.04 (0.46) | -0.19 | 0.99 (0.43) | 1.05 (0.49) | -0.13 |
| median [IQR] | 0.94 [0.80, 1.15] | 0.97 [0.80, 1.19] | -0.06 | 0.90 [0.74, 1.07] | 0.95 [0.78, 1.16] | -0.12 | 0.91 (0.43) | 0.96 (0.49) | -0.11 |
| Missing; n (%) | 7,841 (72.6%) | 7,794 (72.2%) | 0.01 | 20,703 (98.2%) | 20,716 (98.3%) | -0.01 | 28,544 (89.6%) | 28,510 (89.5%) | 0.00 |
| Lab result number- HDL level (mg/dl) mean | 2,339 | 2,294 | | 307 | 283 | | 2,646 | 2,577 | |
| (only =<5000 included) | | | | | | | | | |
| mean (sd) | 50.19 (17.83) | 50.14 (17.34) | 0.00 | 49.24 (16.21) | 48.06 (17.06) | 0.07 | 49.56 (16.78) | 48.76 (17.16) | 0.05 |
| median [IQR] | 49.00 [40.00, 60.00] | 49.00 [40.00, 59.00] | 0.00 | 49.00 [39.50,<br>57.00] | 46.00 [37.00,<br>57.00] | 0.18 | 49.00 (16.78) | 47.02 (17.16) | 0.12 |
| Missing; n (%) | 8,459 (78.3%) | 8,504 (78.8%) | -0.01 | 20,767 (98.5%) | 20,791 (98.7%) | -0.02 | 29,226 (91.7%) | 29,295 (91.9%) | -0.01 |
| Lab result number-LDL level (mg/dl) mean<br>(only =<5000 included) | 2,481 | 2,458 | | 303 | 288 | | 2,784 | 2,746 | |
| mean (sd) | -2,429.55<br>(47,296.88) | -2,059.43<br>(43,132.62) | -0.01 | 97.05 (47.66) | 93.76 (46.96) | 0.07 | -758.94 (27529.19) | -635.72 (25105.38) | 0.00 |
| median [IQR] | 87.50 [65.00,<br>113.00] | 89.00 [67.00,<br>115.00] | 0.00 | 92.00 [69.00,<br>122.00] | 89.00 [65.00,<br>119.75] | 0.06 | 90.48 (27529.19) | 89.00 (25105.38) | 0.00 |
| Missing; n (%) | 8,317 (77.0%) | 8,340 (77.2%) | 0.00 | 20,771 (98.6%) | 20,786 (98.6%) | 0.00 | 29,088 (91.3%) | 29,126 (91.4%) | 0.00 |

Table 1: Telmisartan vs Ramipril

| | Lab result number-Total cholesterol | 2,518 | 2,495 | | 313 | 291 | | 2,831 | 2,786 | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| | (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| Missing n (%) 201.00 200.50 201.00 200.50 20.00 20.50 | mean (sd) | 169.81 (55.72) | 170.21 (54.89) | -0.01 | 179.74 (59.11) | 181.98 (58.55) | -0.04 | 176.38 (57.98) | 177.99 (57.34) | -0.03 |
| Massing n % Lab result number - Frigivorride level (mg/df) mean (only ~5000 included) 143.65 §9.39 142.29 §8.50 0.01 157.67 (107.86) 191.88 (28.25) -0.16 152.92 (105.07) 175.08 (241.03) -0.12 143.65 (93.93) 142.29 (95.50) 0.01 133.00 (90.00) 144.05 (102.00) -0.05 122.27 (105.07) 136.71 (241.03) -0.01 | median [IQR] | 169.00 [142.00, | 171.00 [143.00, | -0.04 | 174.00 [146.00, | 177.00 [151.00, | -0.05 | 172.31 (57.98) | 174.97 (57.34) | -0.05 |
| Lab result number - Triglycenide level (mg/gll) mane (not) v=5000 included) 143.56 [99.39] 142.29 [96.50] 0.01 157.67 [107.86] 191.88 [288.25] 0.01 129.27 [105.07] 136.7 [124.103] 0.01 120.00 120.25] 120.00 [10.00 120.20] 120.20 [10.00] 120.20 [1 | | 201.00] | 200.50] | | 210.00] | 205.00] | | | | |
| fing/dil mean (only =5000 included) mean (rad) m | Missing; n (%) | 8,280 (76.7%) | 8,303 (76.9%) | 0.00 | 20,761 (98.5%) | 20,783 (98.6%) | -0.01 | 29,041 (91.1%) | 29,086 (91.3%) | -0.01 |
| mean (cd) | Lab result number- Triglyceride level | 2,479 | 2,463 | | 313 | 286 | | 2,792 | 2,749 | |
| | (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| Missing n N | mean (sd) | 143.65 (99.39) | 142.29 (96.50) | 0.01 | 157.67 (107.86) | 191.88 (288.25) | -0.16 | 152.92 (105.07) | 175.08 (241.03) | -0.12 |
| Maining n (%) Sale (17,0%) Sal | median [IQR] | 122.00 [86.50, | 121.50 [87.00, | 0.01 | 133.00 [89.00, | 144.50 [102.00, | -0.05 | 129.27 (105.07) | 136.71 (241.03) | -0.04 |
| Lab result number - Hemoglobin mean (only 20 included) 13.51 (1.64) 13.38 (1.69) 0.08 698.10 (10,564.86) 1,097.55 0.04 466.17 (8590.85) 730.24 (9806.31) 0.03 0.05 0.05 | | 174.00] | 174.00] | | 197.00] | 210.25] | | | | |
| [only 30 included]mean [std] | Missing; n (%) | 8,319 (77.0%) | 8,335 (77.2%) | 0.00 | 20,761 (98.5%) | 20,788 (98.6%) | -0.01 | 29,080 (91.2%) | 29,123 (91.4%) | -0.01 |
| 13.51 (1.64) 13.38 (1.69) 0.08 698.10 (10.564.86) 1.097.55 -0.04 466.17 (8590.85) 730.24 (8806.31) -0.03 | Lab result number- Hemoglobin mean | 2,149 | 2,271 | | 238 | 248 | | 2,387 | 2,519 | |
| median [IOR] 13.60 [12.50, 14.60] 13.40 [12.30, 14.50] 0.12 13.40 [12.34, 13.40 [12.30, 0.00 13.47 (8590.85) 13.40 (9806.31) 0.00 14.52 14.52] 14. | (only >0 included) | | | | | | | | | |
| Missing, n (%) Lab result number-Serum sodium mean (only > 50 and < 190 included)mean (st)mean (st | mean (sd) | 13.51 (1.64) | 13.38 (1.69) | 80.0 | 698.10 (10,564.86) | | -0.04 | 466.17 (8590.85) | 730.24 (9806.31) | -0.03 |
| Lab result number- Serum sodium mean (only >0 and <190 included)median [IQR]median [IQ | median [IQR] | 13.60 [12.50, 14.60] | 13.40 [12.30, 14.50] | 0.12 | | | 0.00 | 13.47 (8590.85) | 13.40 (9806.31) | 0.00 |
| (only >90 and <190 included)mean (sd) 140.20 [139.00, 140.50 [139.00, 0.01 139.96 (2.35) 139.62 (2.36) 0.14 140.06 [2.47) 139.82 (2.54) -0.10median [IQR] 140.20 [139.00, 140.50 [139.00, 0.01 141.50] 141.50] 141.50]mean (sd) 140.20 [139.00, 142.00] 142.00] 142.00 1 141.50] 141.50]mean (sd) 140.20 [139.00, 140.00 [138.00, 0.00 140.07 (2.47) 140.17 (2.54) -0.04 142.00] 142.00]mean (sd) 140.20 [139.00, 140.00 [138.00, 0.00 140.07 (2.47) 140.17 (2.54) -0.04 142.00] 142.00] 142.00] 142.00]mean (sd) 140.20 [139.00, 140.00 [138.00, 0.00 140.07 (2.47) 140.17 (2.54) -0.04 142.00] 142.00] 142.00] 0.00 142.00] 142.00] 0.00 142.00] 142.00] 0.00 142.00] 0.00 142.00] 0.00 142.00] 0.00 140.07 (2.47) 140.17 (2.54) -0.04 140.00 [138.00, 0.00 140.00] 28,663 (89.94) 28,598 (89.7%) 0.01 28,663 (89.94) 28,598 (89.7%) 0.0 | Missing; n (%) | 8,649 (80.1%) | 8,527 (79.0%) | 0.03 | 20,836 (98.9%) | 20,826 (98.8%) | 0.01 | 29,485 (92.5%) | 29,353 (92.1%) | 0.02 |
| mean (sd) | Lab result number-Serum sodium mean | 2,899 | 2,971 | | 310 | 303 | | 3,209 | 3,274 | |
| median [IQR] 140.20 [139.00, 140.50 [139.00, 141.50] 140.00 [139.00, 140.00 [138.00, 0.00] 140.07 (2.47) 140.17 (2.54) -0.04 142.00] 142.00] 142.50] 142 | (only > 90 and < 190 included) | | | | | | | | | |
| 142.00 142.00 141.50 141.00 141.00 | mean (sd) | 140.25 (2.70) | 140.22 (2.86) | 0.01 | 139.96 (2.35) | 139.62 (2.36) | 0.14 | 140.06 (2.47) | 139.82 (2.54) | 0.10 |
| Lab result number-Albumin mean (only >0 and <=10 included)mean (sd) | median [IQR] | | • | -0.11 | • | • | 0.00 | 140.07 (2.47) | 140.17 (2.54) | -0.04 |
| and <10 included)mean (sd) | Missing; n (%) | 7,899 (73.2%) | 7,827 (72.5%) | 0.02 | 20,764 (98.5%) | 20,771 (98.6%) | -0.01 | 28,663 (89.9%) | 28,598 (89.7%) | 0.01 |
| mean (sd) | Lab result number- Albumin mean (only >0 | 2,731 | 2,785 | | 293 | 288 | | 3,024 | 3,073 | |
| median [IQR] | and <=10 included) | | | | | | | | | |
| Missing; n (%) Lab result number-Glucose (fasting or random) mean (only 10-1000 included)median [IQR]median [IQR]mesh (sd)median [IQR]mesh (sd)mesh | mean (sd) | 4.22 (0.34) | 4.21 (0.34) | 0.03 | 4.16 (0.62) | 4.12 (0.70) | 0.06 | 4.18 (0.54) | 4.15 (0.60) | 0.05 |
| Lab result number-Glucose (fasting or random) mean (only 10-1000 included)mean (sd) | median [IQR] | 4.25 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.15 | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.22 (0.54) | 4.20 (0.60) | 0.04 |
| random) mean (only 10-1000 included)mean (sd)median [IQR] 126.20 (54.75) 122.77 (52.41) 0.06 140.15 (65.72) 138.06 (59.88) 0.03 135.42 (62.22) 132.88 (57.46) 0.04median [IQR] 107.00 [93.00, 106.00 [93.00, 120.00 [100.00, | Missing; n (%) | 8,067 (74.7%) | 8,013 (74.2%) | 0.01 | 20,781 (98.6%) | 20,786 (98.6%) | 0.00 | 28,848 (90.5%) | 28,799 (90.4%) | 0.00 |
| mean (sd)median [IQR] median [IQR] mean (sd) | Lab result number- Glucose (fasting or | 2,878 | 2,947 | | 303 | 302 | | 3,181 | 3,249 | |
| median [IQR] 107.00 [93.00, 106.00 [93.00, 0.02 121.00 [100.00, 120.00 [100.00, 0.02 116.26 [62.22] 115.26 [57.46] 0.02 139.50] 134.00] 157.00] 157.25] 7,920 (73.3%) 7,851 (72.7%) 0.01 20,771 (98.6%) 20,772 (98.6%) 0.00 28,691 (90.0%) 28,623 (89.8%) 0.01 24 1.71 included) 3333 328 3,274 3,333 3,274 3,333 3,274 3 | random) mean (only 10-1000 included) | | | | | | | | | |
| 139.50] 134.00] 157.00] 157.25] Missing, n (%) 7,920 (73.3%) 7,851 (72.7%) 0.01 20,771 (98.6%) 20,772 (98.6%) 0.00 28,691 (90.0%) 28,623 (89.8%) 0.01 Lab result number- Potassium mean (only 1-7 included) mean (sd) 4.43 (0.43) 4.39 (0.44) 0.09 4.35 (0.41) 4.33 (0.43) 0.05 4.38 (0.42) 4.35 (0.43) 0.07 median [IQR] 4.40 [4.15, 4.70] 4.40 [4.10, 4.70] 0.00 4.35 [4.10, 4.60] 4.30 [4.10, 4.60] 0.12 4.37 (0.42) 4.33 (0.43) 0.09 Missing, n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 Comorbidity Scores CCI (180 days)- ICD9 and ICD10 mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01 median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days, mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.10 (0.05) 0.00 | mean (sd) | 126.20 (54.75) | 122.77 (52.41) | 0.06 | 140.15 (65.72) | 138.06 (59.88) | 0.03 | 135.42 (62.22) | 132.88 (57.46) | 0.04 |
| Missing, n (%) Lab result number- Potassium mean (only 1-7 included)mean (sd)mean (sd)median [IQR]Missing, n (%) Comorbidity Scores CCI (180 days)- ICD9 and ICD10mean (sd)mean (sd)m | median [IQR] | 107.00 [93.00, | 106.00 [93.00, | 0.02 | 121.00 [100.00, | 120.00 [100.00, | 0.02 | 116.26 (62.22) | 115.26 (57.46) | 0.02 |
| Lab result number- Potassium mean (only 1-7 included)mean (sd) 4.43 (0.43) 4.39 (0.44) 0.09 4.35 (0.41) 4.33 (0.43) 0.05 4.38 (0.42) 4.35 (0.43) 0.07median [IQR] 4.40 [4.15, 4.70] 4.40 [4.10, 4.70] 0.00 4.35 [4.10, 4.60] 4.30 [4.10, 4.60] 0.12 4.37 (0.42) 4.33 (0.43) 0.09Missing, n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 Comorbidity Scores CCI (180 days)- ICD9 and ICD10mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | 139.50] | 134.00] | | 157.00] | 157.25] | | | | |
| 1-7 included)mean (sd)mean (sd)median [IQR]meidian [IQR]median [IQR]median [IQR]median [IQR]mesing; n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 Comorbidity Scores CCI (180 days)- ICD9 and ICD10mean (sd)mean (sd)median [IQR] 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.17 (0.06) 0.17 (0.06) 0.00 0.18 (0.05) 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 | Missing; n (%) | 7,920 (73.3%) | 7,851 (72.7%) | 0.01 | 20,771 (98.6%) | 20,772 (98.6%) | 0.00 | 28,691 (90.0%) | 28,623 (89.8%) | 0.01 |
| mean (sd) 4.43 (0.43) 4.39 (0.44) 0.09 4.35 (0.41) 4.33 (0.43) 0.05 4.38 (0.42) 4.35 (0.43) 0.07median [IQR] 4.40 [4.15, 4.70] 4.40 [4.10, 4.70] 0.00 4.35 [4.10, 4.60] 4.30 [4.10, 4.60] 0.12 4.37 (0.42) 4.33 (0.43) 0.09Missing, n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 Comorbidity Scores CCI (180 days)- ICD9 and ICD10mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | 2,941 | 3,005 | | 333 | 328 | | 3,274 | 3,333 | |
| median [IQR] 4.40 [4.15, 4.70] 4.40 [4.10, 4.70] 0.00 4.35 [4.10, 4.60] 4.30 [4.10, 4.60] 0.12 4.37 (0.42) 4.33 (0.43) 0.09Missing, n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 CCI (180 days)-ICD9 and ICD10mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | 1-7 included) | | | | | | | | | |
| Missing, n (%) 7,857 (72.8%) 7,793 (72.2%) 0.01 20,741 (98.4%) 20,746 (98.4%) 0.00 28,598 (89.7%) 28,539 (89.5%) 0.01 Comorbidity Scores CCI (180 days)-ICD9 and ICD10mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01 median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | . , | | | | | | | | | |
| Comorbidity Scores CCI (180 days)-ICD9 and ICD10mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01 1.96 (1.69) 1.95 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.10 (0.05) | | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10mean (sd) | | 7,857 (72.8%) | 7,793 (72.2%) | 0.01 | 20,741 (98.4%) | 20,746 (98.4%) | 0.00 | 28,598 (89.7%) | 28,539 (89.5%) | 0.01 |
| mean (sd) 2.46 (1.91) 2.44 (1.87) 0.01 1.71 (1.57) 1.70 (1.52) 0.01 1.96 (1.69) 1.95 (1.65) 0.01 median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days, mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | - | | | | | | | | | |
| median [IQR] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 0.00 1.00 [1.00, 2.00] 0.00 1.34 (1.69) 1.34 (1.65) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | | | | | | | | | |
| Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | | | | | | | | | |
| days,mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | | 2.00 [1.00, 3.00] | 0.00 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 1.34 (1.69) | 1.34 (1.65) | 0.00 |
| mean (sd) 0.17 (0.06) 0.17 (0.06) 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) 0.00 | | | | | | | | | | |
| median [IQR] 0.16 [0.14, 0.20] 0.16 [0.14, 0.20] 0.00 0.15 [0.13, 0.18] 0.15 [0.13, 0.18] 0.00 0.15 (0.05) 0.15 (0.05) | | | | | | | | | | |
| | median [IQR] | 0.16 [0.14, 0.20] | 0.16 [0.14, 0.20] | 0.00 | 0.15 [0.13, 0.18] | 0.15 [0.13, 0.18] | 0.00 | 0.15 (0.05) | 0.15 (0.05) | 0.00 |

Table 1: Telmisartan vs Ramipril

| Healthcare Utilization | I | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization; n (%) | 1,039 (9.6%) | 1,047 (9.7%) | 0.00 | 2,526 (12.0%) | 2,508 (11.9%) | 0.00 | 3,565 (11.2%) | 3,555 (11.2%) | 0.00 |
| Any hospitalization during prior 31-180 | 796 (7.4%) | 817 (7.6%) | -0.01 | 1,965 (9.3%) | 1,935 (9.2%) | 0.00 | 2,761 (8.7%) | 2,752 (8.6%) | 0.00 |
| days; n (%) | , | (* :-:-) | | _,, | 2,222 (0.2.0) | | _,, (,_, | _,, (_,,,,, | |
| Endocrinologist Visit; n (%) | 775 (7.2%) | 760 (7.0%) | 0.01 | 1,210 (5.7%) | 1,226 (5.8%) | 0.00 | 1,985 (6.2%) | 1,986 (6.2%) | 0.00 |
| Endocrinologist Visit (30 days prior); n (%) | 285 (2.6%) | 279 (2.6%) | 0.00 | 462 (2.2%) | 468 (2.2%) | 0.00 | 0,747 (2.3%) | 0,747 (2.3%) | 0.00 |
| | ` ' | . , | | . , | ` ' | | , , , | , , , | |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 668 (6.2%) | 659 (6.1%) | 0.00 | 1,050 (5.0%) | 1,072 (5.1%) | 0.00 | 1,718 (5.4%) | 1,731 (5.4%) | 0.00 |
| Internal medicine/family medicine visits; n<br>(%) | 8,235 (76.3%) | 8,214 (76.1%) | 0.00 | 16,197 (76.9%) | 16,428 (78.0%) | -0.03 | 24,432 (76.7%) | 24,642 (77.3%) | -0.01 |
| Internal medicine/family medicine visits<br>(30 days prior); n (%) | 5,405 (50.1%) | 5,194 (48.1%) | 0.04 | 10,493 (49.8%) | 10,094 (47.9%) | 0.04 | 15,898 (49.9%) | 15,288 (48.0%) | 0.04 |
| Internal medicine/family medicine visits | 7,225 (66.9%) | 7,227 (66.9%) | 0.00 | 14,210 (67.4%) | 14,711 (69.8%) | -0.05 | 21,435 (67.3%) | 21,938 (68.8%) | -0.03 |
| (31 to 180 days prior); n (%) | | | | | | | | | |
| Cardiologist visit; n (%) | 4,248 (39.3%) | 4,215 (39.0%) | 0.01 | 6,932 (32.9%) | 6,906 (32.8%) | 0.00 | 11,180 (35.1%) | 11,121 (34.9%) | 0.00 |
| Number of Cardiologist visits (30 days | 1,865 (17.3%) | 1,875 (17.4%) | 0.00 | 3,056 (14.5%) | 3,045 (14.4%) | 0.00 | 4,921 (15.4%) | 4,920 (15.4%) | 0.00 |
| prior); n (%) | | | | | | | | | |
| Number of Cardiologist visits (31 to 180 | 3,390 (31.4%) | 3,420 (31.7%) | -0.01 | 5,653 (26.8%) | 5,635 (26.7%) | 0.00 | 9,043 (28.4%) | 9,055 (28.4%) | 0.00 |
| days prior); n (%) | | | | | | | | | |
| Electrocardiogram ; n (%) | 4,169 (38.6%) | 4,291 (39.7%) | -0.02 | 8,178 (38.8%) | 8,113 (38.5%) | 0.01 | 12,347 (38.7%) | 12,404 (38.9%) | 0.00 |
| Use of glucose test strips; n (%) | 296 (2.7%) | 275 (2.5%) | 0.01 | 336 (1.6%) | 353 (1.7%) | -0.01 | 0,632 (2.0%) | 0,628 (2.0%) | 0.00 |
| Dialysis; n (%) | 35 (0.3%) | 33 (0.3%) | 0.00 | 64 (0.3%) | 43 (0.2%) | 0.02 | 99 (0.3%) | 76 (0.2%) | 0.02 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 8.42 (4.74) | 8.35 (4.89) | 0.01 | 8.79 (5.01) | 8.75 (4.98) | 0.01 | 8.66 (4.92) | 8.61 (4.95) | 0.01 |
| median [IQR] | 8.00 [5.00, 11.00] | 8.00 [5.00, 11.00] | 0.00 | 8.00 [5.00, 11.00] | 8.00 [5.00, 11.00] | 0.00 | 8.00 (4.92) | 8.00 (4.95) | 0.00 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.11 (0.37) | 0.12 (0.39) | -0.03 | 0.13 (0.39) | 0.13 (0.39) | 0.00 | 0.12 (0.38) | 0.13 (0.39) | -0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.38) | 0.00 (0.39) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 0.61 (2.77) | 0.64 (3.07) | -0.01 | 0.72 (2.86) | 0.70 (3.05) | 0.01 | 0.68 (2.83) | 0.68 (3.06) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (2.83) | 0.00 (3.06) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.43 (1.17) | 0.45 (1.15) | -0.02 | 0.12 (0.90) | 0.12 (1.01) | 0.00 | 0.23 (1.00) | 0.23 (1.06) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.00) | 0.00 (1.06) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 5.51 (4.70) | 5.46 (4.45) | 0.01 | 5.62 (4.90) | 5.60 (4.62) | 0.00 | 5.58 (4.83) | 5.55 (4.56) | 0.01 |
| median [IQR] | 4.00 [2.00, 7.00] | 4.00 [2.00, 7.00] | 0.00 | 4.00 [2.00, 8.00] | 5.00 [2.00, 8.00] | -0.21 | 4.00 (4.83) | 4.66 (4.56) | -0.14 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.33 (1.76) | 0.34 (1.95) | -0.01 | 0.27 (1.70) | 0.27 (1.74) | 0.00 | 0.32 (1.54) | 0.33 (1.57) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.54) | 0.00 (1.57) | 0.00 |
| Number of internal medicine/family | | | | | | | | | |
| medicine visits | | | | | | | | | |
| mean (sd) | 7.93 (12.42) | 8.01 (12.57) | -0.01 | 6.43 (10.52) | 6.42 (9.97) | 0.00 | 6.94 (11.20) | 6.96 (10.92) | 0.00 |
| median [IQR] | 4.00 [1.00, 10.00] | 4.00 [1.00, 10.00] | 0.00 | 3.00 [1.00, 8.00] | 4.00 [1.00, 8.00] | -0.10 | 3.34 (11.20) | 4.00 (10.92) | -0.06 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 2.26 (5.11) | 2.19 (4.76) | 0.01 | 1.74 (4.37) | 1.77 (4.23) | -0.01 | 1.92 (4.63) | 1.91 (4.42) | 0.00 |
| - | - | | | | | | | | |

Table 1: Telmisartan vs Ramipril

| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (4.63) | 0.00 (4.42) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Number electrocardiograms received | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (4.03) | 0.00 (4.42) | 0.00 |
| mean (sd) | 0.77 (1.52) | 0.79 (1.47) | -0.01 | 0.67 (1.21) | 0.67 (1.18) | 0.00 | 0.70 (1.32) | 0.71 (1.29) | -0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.32) | 0.00 (1.29) | 0.00 |
| Number of HbA1c tests ordered | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (2.52) | 0.00 (2.25) | 0.00 |
| mean (sd) | 0.62 (0.87) | 0.62 (0.85) | 0.00 | 0.33 (0.67) | 0.32 (0.67) | 0.01 | 0.43 (0.74) | 0.42 (0.74) | 0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.74) | 0.00 (0.74) | 0.00 |
| Number of glucose tests ordered | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (0.1.1) | 0.00 (0.7.1) | 5.55 |
| mean (sd) | 0.32 (1.98) | 0.30 (1.24) | 0.01 | 0.19 (2.25) | 0.18 (0.74) | 0.01 | 0.23 (2.16) | 0.22 (0.94) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (2.16) | 0.00 (0.94) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.81 (0.97) | 0.82 (0.96) | -0.01 | 0.47 (0.99) | 0.47 (0.92) | 0.00 | 0.59 (0.98) | 0.59 (0.93) | 0.00 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.34 (0.98) | 0.34 (0.93) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.08 (0.46) | 0.08 (0.44) | 0.00 | 0.06 (0.35) | 0.06 (0.34) | 0.00 | 0.07 (0.39) | 0.07 (0.38) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.39) | 0.00 (0.38) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.06 (0.53) | 0.06 (0.49) | 0.00 | 0.04 (0.36) | 0.04 (0.36) | 0.00 | 0.05 (0.43) | 0.05 (0.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.43) | 0.00 (0.41) | 0.00 |
| Number of tests for microal buminuria | | | | | | | | | |
| mean (sd) | 0.39 (0.92) | 0.39 (0.93) | 0.00 | 0.17 (0.61) | 0.18 (0.62) | -0.02 | 0.24 (0.73) | 0.25 (0.74) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.73) | 0.00 (0.74) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at | | | | | | | | | |
| the 3rd digit level<br>mean (sd) | 4.68 (7.40) | 4.67 (7.41) | 0.00 | 1.33 (3.41) | 1.34 (3.40) | 0.00 | 2.46 (5.12) | 2.47 (5.12) | 0.00 |
| median [IQR] | 1.00 [0.00, 7.00] | 1.00 [0.00, 7.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.34 (5.12) | 0.34 (5.12) | 0.00 |
| For PS | 1.00 [0.00, 7.00] | 1.00 [0.00, 7.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.34 (3.12) | 0.34 (3.12) | 0.00 |
| Hemorrhagic stroke+Other | 415 (3.8%) | 390 (3.6%) | 0.01 | 600 (2.8%) | 563 (2.7%) | 0.01 | 1015 (3.2%) | 953 (3.0%) | 0.01 |
| cerebrovascular disease+Cerebrovascular | | () | | (2.2.0) | () | | () | () | |
| procedure (for PS); n (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for | 608 (5.6%) | 592 (5.5%) | 0.00 | 874 (4.1%) | 832 (3.9%) | 0.01 | 1,482 (4.6%) | 1,424 (4.5%) | 0.00 |
| PS); n (%) | | | | | | | | | |
| Occurrence of BUN tests ordered (for PS); n | 391 (3.6%) | 382 (3.5%) | 0.01 | 613 (2.9%) | 590 (2.8%) | 0.01 | 1,004 (3.2%) | 0,972 (3.0%) | 0.01 |
| (%) | | | | | | | | | |
| Occurrence of chronic renal insufficiency | 620 (5.7%) | 575 (5.3%) | 0.02 | 555 (2.6%) | 547 (2.6%) | 0.00 | 1,175 (3.7%) | 1,122 (3.5%) | 0.01 |
| w/o CKD (for PS) ; n (%) | 004 (0.70) | 002 (0.70) | | 222 (4.484) | 225 (4.424) | | F07 (4 70/) | 540 (4.50) | 0.04 |
| Chronic kidney disease Stage 1-2 (for PS); n<br>(%) | 294 (2.7%) | 293 (2.7%) | 0.00 | 233 (1.1%) | 225 (1.1%) | 0.00 | 527 (1.7%) | 518 (1.6%) | 0.01 |
| (70) Chronic kidney disease Stage 3-6 (for PS); n | 1,058 (9.8%) | 1,009 (9.3%) | 0.02 | 945 (4.5%) | 939 (4.5%) | 0.00 | 2,003 (6.3%) | 1,948 (6.1%) | 0.01 |
| (%) | 1,056 (5.6%) | 1,005 (5.5%) | 0.02 | 343 (4.370) | 333 (4.3%) | 0.00 | 2,003 (6.3%) | 1,546 (6.170) | 0.01 |
| Bladder stones+Kidney stones (for PS); n | 236 (2.2%) | 226 (2.1%) | 0.01 | 353 (1.7%) | 360 (1.7%) | 0.00 | 0,589 (1.8%) | 0,586 (1.8%) | 0.00 |
| (%) | | () | | ( /-) | (2/2) | | -, (2.0.0) | -, (2.074) | |
| Diabetes with peripheral circulatory | 485 (4.5%) | 484 (4.5%) | 0.00 | 450 (2.1%) | 448 (2.1%) | 0.00 | 0,935 (2.9%) | 0,932 (2.9%) | 0.00 |
| disorders+Gangrene+Osteomyelitis(for PS) | | • | | | • | | | | |
| with ICD10; n (%) | | | | | | | | | |
| Alcohol abuse or dependence+Drug abuse | 184 (1.7%) | 181 (1.7%) | 0.00 | 147 (0.7%) | 146 (0.7%) | 0.00 | 331 (1.0%) | 327 (1.0%) | 0.00 |
| or dependence (for PS); n (%) | | | | | | | | | |

Table 1: Telmisartan vs Ramipril

| Diabetes with other ophthalmic<br>manifestations+Retinal detachment,<br>vitreous hemorrhage, vitrectomy+Retinal | 171 (1.6%) | 178 (1.6%) | 0.00 | 777 (3.7%) | 745 (3.5%) | 0.01 | 0,948 (3.0%) | 0,923 (2.9%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| laser coagulation therapy (for PS); n (%) Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS); n (%) | 1,890 (17.5%) | 1,940 (18.0%) | -0.01 | 3,122 (14.8%) | 3,069 (14.6%) | 0.01 | 5,012 (15.7%) | 5,009 (15.7%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA (for PS) | 819 (7.6%) | 827 (7.7%) | 0.00 | 696 (3.3%) | 720 (3.4%) | -0.01 | 1,515 (4.8%) | 1,547 (4.9%) | 0.00 |
| ; n (%) Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 2,036 (18.9%) | 2,026 (18.8%) | 0.00 | 2,345 (11.1%) | 2,302 (10.9%) | 0.01 | 4,381 (13.7%) | 4,328 (13.6%) | 0.00 |
| Delirium + Psychosis (for PS); n (%) | 205 (1.9%) | 188 (1.7%) | 0.02 | 246 (1.2%) | 264 (1.3%) | -0.01 | 451 (1.4%) | 452 (1.4%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | 69 (0.6%) | 70 (0.6%) | 0.00 | 229 (1.1%) | 236 (1.1%) | 0.00 | 298 (0.9%) | 306 (1.0%) | -0.01 |
| Any use of AGIs (for PS); n (%) | 13 (0.1%) | 14 (0.1%) | 0.00 | 3,122 (14.8%) | 3,069 (14.6%) | 0.01 | 5,012 (15.7%) | 5,009 (15.7%) | 0.00 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 1,062 (9.8%) | 1,017 (9.4%) | 0.00 | 966 (4.6%) | 942 (4.5%) | 0.00 | 2,028 (6.4%) | 1,959 (6.1%) | 0.00 |
| Use of thiazide; n (%) | 1,217 (11.3%) | 1,206 (11.2%) | 0.00 | 2,245 (10.7%) | 2,192 (10.4%) | 0.01 | 12,766 (40.1%) | 12,770 (40.1%) | 0.00 |
| Use of beta blockers; n (%) | 4,323 (40.0%) | 4,313 (39.9%) | 0.00 | 8,443 (40.1%) | 8,457 (40.1%) | 0.00 | 9,032 (28.3%) | 8,944 (28.1%) | 0.00 |
| Use of calcium channel blockers; n (%) | 3,057 (28.3%) | 3,052 (28.3%) | 0.00 | 5,975 (28.4%) | 5,892 (28.0%) | 0.01 | 9,980 (31.3%) | 9,933 (31.2%) | 0.00 |
| All antidiabetic medications except<br>Insulin; n (%) | 3,614 (33.5%) | 3,591 (33.3%) | 0.00 | 6,366 (30.2%) | 6,342 (30.1%) | 0.00 | 3,462 (10.9%) | 3,398 (10.7%) | 0.01 |
| DM Medications - Insulin ; n (%) | 1,311 (12.1%) | 1,288 (11.9%) | 0.01 | 2,346 (11.1%) | 2,279 (10.8%) | 0.01 | 3,657 (11.5%) | 3,567 (11.2%) | 0.01 |
| Use of Low Intensity Statins; n (%) | 2,886 (26.7%) | 2,867 (26.6%) | 0.00 | 5,753 (27.3%) | 5,812 (27.6%) | -0.01 | 8639 (27.1%) | 8,679 (27.2%) | 0.00 |
| Use of High Intensity Statins; n (%) | 2,896 (26.8%) | 2,809 (26.0%) | 0.02 | 4,972 (23.6%) | 4,837 (23.0%) | 0.01 | 7868 (24.7%) | 7,646 (24.0%) | 0.02 |
| Malignant hypertension; n (%) | 314 (2.9%) | 304 (2.8%) | 0.01 | 7,681 (36.4%) | 7,737 (36.7%) | -0.01 | 7995 (25.1%) | 8,041 (25.2%) | 0.00 |
| Cardiovascular stress test; n (%) | 34 (0.3%) | 34 (0.3%) | 0.00 | 79 (0.4%) | 75 (0.4%) | 0.00 | 0,113 (0.4%) | 109 (0.3%) | 0.02 |
| Echocardiogram; n (%) | 1,689 (15.6%) | 1,723 (16.0%) | -0.01 | 3,801 (18.0%) | 3,752 (17.8%) | 0.01 | 5,490 (17.2%) | 5475 (17.2%) | 0.00 |
| Number of BNP tests | | | | | | | | | |
| mean (sd) | 0.05 (0.29) | 0.05 (0.29) | 0.00 | 0.03 (0.20) | 0.03 (0.20) | 0.00 | 0.04 (0.23) | 0.04 (0.23) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.23) | 0.00 |
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.28 (1.16) | 0.29 (1.07) | -0.01 | 0.18 (0.89) | 0.17 (0.94) | 0.01 | 0.21 (0.99) | 0.21 (0.99) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.99) | 0.00 (0.99) | 0.00 |
| Number of Ambulatory Blood pressure | . , . | | | | | | | | |
| monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.05) | 0.00 (0.06) | 0.00 | 0.00 (0.09) | 0.00 (0.07) | 0.00 | 0.00 (0.08) | 0.00 (0.07) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.08) | 0.00 (0.07) | 0.00 |
| N of days on antihypertensive medications | . , , | . , . | | | | | | | |
| during baseline | | | | | | | | | |
| mean (sd) | 84.64 (73.97) | 83.37 (72.98) | 0.02 | 90.02 (73.50) | 89.44 (72.27) | 0.01 | 88.20 (73.66) | 87.38 (72.51) | 0.01 |
| median [IQR] | | 78.00 [1.00, 165.00] | 0.04 | 89.00 [1.00,<br>170.00] | 86.00 [1.00,<br>168.00] | 0.04 | 86.29 (73.66) | 83.29 (72.51) | 0.04 |
| N of days in database anytime prior | | | | | | | | | |
| mean (sd) | 1.658.62 (1.202.43) | 1,646.78 (1,190.83) | 0.01 | 1,693.01 | 1,698.81 | -0.01 | 1681.36 (1159.79) | 1681.18 (1152.93) | 0.00 |
| | -,(-,:15) | -, (2,220.03) | | (1,137.33) | (1,133.02) | | | | |
| median [IQR] | 1,366.00 [726.00,<br>2,255.00] | 1,353.50 [731.00,<br>2,246.00] | 0.01 | 1,441.00 [781.00,<br>2,363.25] | | -0.02 | 1415.59 (1159.79) | 1426.56 (1152.93) | -0.01 |

Table 1: Telmisartan vs Ramipril

| Mean Copay for per prescription cost | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 30.82 (38.30) | 30.67 (37.74) | 0.00 | 23.28 (26.42) | 23.56 (26.22) | -0.01 | 25.83 (30.96) | 25.97 (30.61) | 0.00 |
| median [IQR] | 21.88 [9.56, 38.75] | 21.54 [9.00, 38.59] | 0.01 | 17.14 [6.66, 31.86] | 17.67 [6.64, 32.50] | -0.02 | 18.75 (30.96) | 18.98 (30.61) | -0.01 |
| Missing; n (%) | 692 (6.4%) | 702 (6.5%) | 0.00 | 1,075 (5.1%) | 1,043 (4.9%) | 0.01 | 1,767 (5.5%) | 1745 (5.5%) | 0.00 |
| Colonos; n (%) | 529 (4.9%) | 511 (4.7%) | 0.01 | 1,182 (5.6%) | 1,124 (5.3%) | 0.01 | 1,711 (5.4%) | 1635 (5.1%) | 0.01 |
| Fecal occult blood (FOB) test; n (%) | 560 (5.2%) | 559 (5.2%) | 0.00 | 773 (3.7%) | 775 (3.7%) | 0.00 | 1,333 (4.2%) | 1334 (4.2%) | 0.00 |
| Flu vaccine; n (%) | 1,686 (15.6%) | 1,725 (16.0%) | -0.01 | 2,082 (9.9%) | 2,106 (10.0%) | 0.00 | 3,768 (11.8%) | 3831 (12.0%) | -0.01 |
| Mammogram; n (%) | 1,305 (12.1%) | 1,335 (12.4%) | -0.01 | 2,335 (11.1%) | 2,365 (11.2%) | 0.00 | 3,640 (11.4%) | 3700 (11.6%) | -0.01 |
| Pap smear; n (%) | 465 (4.3%) | 464 (4.3%) | 0.00 | 1,011 (4.8%) | 1,005 (4.8%) | 0.00 | 1,476 (4.6%) | 1469 (4.6%) | 0.00 |
| Pneumonia vaccine; n (%) | 1,049 (9.7%) | 1,038 (9.6%) | 0.00 | 673 (3.2%) | 683 (3.2%) | 0.00 | 1,722 (5.4%) | 1721 (5.4%) | 0.00 |
| PSA test or Prostate exam for DRE; n (%) | 1,615 (15.0%) | 1,643 (15.2%) | -0.01 | 1,947 (9.2%) | 1,950 (9.3%) | 0.00 | 3,562 (11.2%) | 3593 (11.3%) | 0.00 |
| Bone mineral density; n (%) | 459 (4.3%) | 464 (4.3%) | 0.00 | 627 (3.0%) | 648 (3.1%) | -0.01 | 1,086 (3.4%) | 1112 (3.5%) | -0.01 |
| Use of Sympatomimetic agents; n (%) | 137 (1.3%) | 138 (1.3%) | 0.00 | 399 (1.9%) | 427 (2.0%) | -0.01 | 0,536 (1.7%) | 565 (1.8%) | -0.01 |
| Use of CNS stimulants; n (%) | 73 (0.7%) | 66 (0.6%) | 0.01 | 163 (0.8%) | 170 (0.8%) | 0.00 | 0,236 (0.7%) | 236 (0.7%) | 0.00 |
| Use of estrogens, progestins, androgens; n | 567 (5.3%) | 532 (4.9%) | 0.02 | 1,428 (6.8%) | 1,495 (7.1%) | -0.01 | 1,995 (6.3%) | 2027 (6.4%) | 0.00 |
| (%) | | | | | | | | | |
| Use of Angiogenesis inhibitors; n (%) | 6 (0.1%) | 5 (0.0%) | 0.04 | 14 (0.1%) | 12 (0.1%) | 0.00 | 0,020 (0.1%) | 17 (0.1%) | 0.00 |
| Use of Oral Immunosuppressants; n (%) | 35 (0.3%) | 18 (0.2%) | 0.02 | 70 (0.3%) | 54 (0.3%) | 0.00 | 0,105 (0.3%) | 72 (0.2%) | 0.02 |
| Cardiomegaly, LVH, and other cardiopathy | 1,211 (11.2%) | 1,184 (11.0%) | 0.01 | 1,704 (8.1%) | 1,699 (8.1%) | 0.00 | 2,915 (9.1%) | 2883 (9.0%) | 0.00 |
| due to hypertension; n (%) | | | | | | | | | |
| Ultrasound; n (%) | 1,986 (18.4%) | 2,015 (18.7%) | -0.01 | 4,463 (21.2%) | 4,409 (20.9%) | 0.01 | 6,449 (20.2%) | 6424 (20.2%) | 0.00 |
| Symptomatic hypotension; n (%) | 178 (1.6%) | 187 (1.7%) | -0.01 | 265 (1.3%) | 238 (1.1%) | 0.02 | 0,443 (1.4%) | 425 (1.3%) | 0.01 |
| Syncopal episodes; n (%) | 234 (2.2%) | 231 (2.1%) | 0.01 | 321 (1.5%) | 315 (1.5%) | 0.00 | 0,555 (1.7%) | 546 (1.7%) | 0.00 |
| N of Generic name drugs only | | | | | | | | | |
| mean (sd) | 11.16 (12.36) | 11.01 (12.23) | 0.01 | 8.52 (8.59) | 8.48 (8.55) | 0.00 | 9.41 (10.03) | 9.34 (9.95) | 0.01 |
| median [IQR] | 8.00 [3.00, 15.00] | 7.00 [3.00, 15.00] | 0.08 | 6.00 [2.00, 12.00] | 6.00 [2.00, 12.00] | 0.00 | 6.68 (10.03) | 6.34 (9.95) | 0.03 |
| N of Brand name drugs only | ,, | , | | ,, | ,, | | | | |
| mean (sd) | 4.71 (6.40) | 4.64 (6.19) | 0.01 | 5.72 (6.82) | 5.67 (6.39) | 0.01 | 5.38 (6.68) | 5.32 (6.32) | 0.01 |
| median [IQR] | 2.00 [0.00, 7.00] | 2.00 [0.00, 6.00] | 0.00 | 4.00 [1.00, 8.00] | 4.00 [1.00, 8.00] | 0.00 | 3.32 (6.68) | 3.32 (6.32) | 0.00 |
| Number of distinct antihypertensive | | | | | | | | (/ | |
| generic medications (180-1 days before | | | | | | | | | |
| index) | | | | | | | | | |
| mean (sd) | 1.07 (1.21) | 1.07 (1.20) | 0.00 | 1.09 (1.21) | 1.08 (1.20) | 0.01 | 1.08 (1.21) | 1.08 (1.20) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 (1.21) | 1.00 (1.20) | 0.00 |
| Number of distinct antihypertensive | | | | | [] | | | | |
| generic medications on CED | | | | | | | | | |
| mean (sd) | 1.26 (0.57) | 1.26 (0.61) | 0.00 | 1.26 (0.58) | 1.26 (0.60) | 0.00 | 1.26 (0.58) | 1.26 (0.60) | 0.00 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.58) | 1.00 (0.60) | 0.00 |
| Hypertensive retinopathy; n (%) | 95 (0.9%) | 104 (1.0%) | -0.01 | 119 (0.6%) | 117 (0.6%) | 0.00 | 0 | 0 | #VALUE! |
| Commercial vs Medicare Advantage- | () | | | () | () | | _ | _ | |
| Business Type Code - CORRECT ONE -<br>TRUVEN | | | | | | | | | |
| Commercial; n (%) | 4,759 (44.1%) | 4,766 (44.1%) | 0.00 | 12,068 (57.3%) | 11,960 (56.8%) | 0.01 | 16,827 (52.8%) | 16726 (52.5%) | 0.01 |
| Medicare Advantage; n (%) | 6,039 (55.9%) | 6,032 (55.9%) | 0.00 | 9,006 (42.7%) | 9,114 (43.2%) | -0.01 | 15,045 (47.2%) | 15146 (47.5%) | -0.01 |
| Commercial vs Medicare Advantage- | -, () | -, | | -,( | -,, | | | | |
| Business Type Code | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 4,759 (44.1%) | 4,766 (44.1%) | 0.00 | | | #VALUE! | 4,759 (44.1%) | 4,766 (44.1%) | 0.00 |

Table 1: Telmisartan vs Ramipril

| MCR = MEDICARE; n (%) | 6,039 (55.9%) | 6,032 (55.9%) | 0.00 | - | - | #VALUE! | 6,039 (55.9%) | 6,032 (55.9%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage-Data<br>Type | - | - | #VALUE! | 0 | 0 | #VALUE! | 0 | 0 | #VALUE! |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 8,196 (38.9%) | 8,292 (39.3%) | -0.01 | 8,196 (38.9%) | 8,292 (39.3%) | -0.01 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 810 (3.8%) | 822 (3.9%) | -0.01 | 810 (3.8%) | 822 (3.9%) | -0.01 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 11,407 (54.1%) | 11,287 (53.6%) | 0.01 | 11,407 (54.1%) | 11,287 (53.6%) | 0.01 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 661 (3.1%) | 673 (3.2%) | -0.01 | 661 (3.1%) | 673 (3.2%) | -0.01 |
| Metropolitan Statistical Area - Urban (any<br>MSA) vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 15,898 (75.4%) | 15,898 (75.4%) | 0.00 | 15,898 (75.4%) | 15,898 (75.4%) | 0.00 |
| Rural; n (%) | - | - | #VALUE! | 220 (1.0%) | 199 (0.9%) | 0.01 | 220 (1.0%) | 199 (0.9%) | 0.01 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 4,956 (23.5%) | 4,977 (23.6%) | 0.00 | 4,956 (23.5%) | 4,977 (23.6%) | 0.00 |